Title: A Phase IIa, Double-Blind, Randomized, Placebo-Controlled, Exploratory Study to Evaluate the Safety, Biological Activity and Pharmacokinetics of GBR 830 in Adult Patients With Moderate-to-Severe Atopic Dermatitis

NCT02683928

Document Date: 12-Apr-2018

## STATISTICAL ANALYSIS PLAN

## Version 6.0: Addendum to Version 5.0 DATE OF PLAN:

12-Apr-2018

#### **BASED ON:**

Statistical Analysis Plan (SAP) Version 5.0, 06-Jul-2017 Protocol Amendment 3.0 Protocol Version 4.0, 16-Feb-2017 Case Report Form (CRF) Version 5.0, 03-June 2016

#### **STUDY DRUG:**

GBR 830

#### **PROTOCOL NUMBER:**

GBR 830-201

#### **STUDY TITLE:**

A Phase IIa, Double-Blind, Randomized, Placebo-controlled, Exploratory Study to Evaluate the Safety, Biological Activity and Pharmacokinetics of GBR 830 in Adult Subjects with Moderate to Severe Atopic Dermatitis

#### **SPONSOR:**

Glenmark Pharmaceuticals SA, Chemin de la Combeta 5, 2300 La Chaux-de-Fonds, Switzerland

This study was conducted in compliance with Good Clinical Practice, including the archiving of essential documents.

#### **SIGNATURE PAGE**

This document has been reviewed and approved by:

Hui Fang

Project Statistician

Glenmark Pharmaceuticals

Signature

10 p 1. 1-, 20

Date

Gerhard Wolff

Vice President Clinical Sciences

Glenmark Pharmaceuticals

Signature

Date

## TABLE OF CONTENTS

| SIGNATURE PAGE | 2 |
|---|---|
| 1. REVISION HISTORY AND SUMMARY OF CHANGES | 4 |
| 2. PURPOSE OF ADDENDUM | 5 |
| APPENDIX 1. TABLE OF CONTENTS FOR DATA DISPLAY SPECIFICATIONS – ALL TABLES, LISTINGS AND FIGURES | 7 |
| APPENDIX 2. DATA DISPLAY SPECIFICATIONS – NEW TABLE 14.2.4.6, NEW LISTINGS 16.2.6.17 AND 16.2.6.18 | 8 |

## 1. REVISION HISTORY AND SUMMARY OF CHANGES

## **REVISION HISTORY**

Statistical Analysis Plan (SAP) version 6.0, an SAP addendum, and SAP version 5.0 supersede the previous versions of the SAP.

| Version | Description | <b>Document Date</b> |
|---------|-------------------------|----------------------|
| 1.0 | Draft, not signed-off | 06-Sep-2016 |
| 2.0 | Draft, not signed-off | 18-Jan-2017 |
| 3.0 | Draft, not signed-off | 14-Mar-2017 |
| 4.0 | Signed-off | 04-Apr-2017 |
| 5.0 | Signed-off | 06-Jul-2017 |
| 6.0 | Addendum to version 5.0 | 26-Mar-2018 |

## **SUMMARY OF CHANGES IN ADDENDUM V6.0**

The following table and listings that were pre-specified in the protocol are being added to the SAP in addendum v6.0.

| Table or Listing<br>Number | Title | Analysis Set |
|---|---|---|
| Table 14.2.4.6 | Percent Change from Baseline in Body Surface Area<br>Involved for Atopic Dermatitis at Each Visit | Full Analysis Set |
| Listing 16.2.6.17 | Body Surface Area Involved for Atopic Dermatitis | Full Analysis Set |
| Listing 16.2.6.18 | Whole Body Photography | Full Analysis Set |

#### 2. PURPOSE OF ADDENDUM

The purpose of this statistical analysis plan (SAP) addendum is to add 1 summary table for body surface area (BSA), 1 listing for BSA, and 1 listing for whole body photography. These data were pre-specified in the protocol and were collected in the case report form (CRF) database prior to database lock.

The SAP version 5.0 dated 06-Jul-2017 was signed-off by Glenmark on 10-Jul-2017 and by Numerus (the Contract Research Organization that performed the statistical analysis) on 11-Jul-2017, before the database lock on 11-Jul-2017. In both study protocol version 4.0 and SAP version 5.0, percent improvement in BSA involved for atopic dermatitis (AD) from baseline at each visit was listed as one of the secondary efficacy endpoints for all subjects, and whole body photography was also to be collected for subjects who gave specific consent for the photography. However, there were no table or listing shell for BSA by visit and no listing shell for the whole body photography included in the SAP version 5.0.

These 3 outputs are needed for the clinical study report. The shells are provided in this statistical addendum. No statistical analyses will be performed for whole body photography.

# APPENDIX 1. TABLE OF CONTENTS FOR DATA DISPLAY SPECIFICATIONS – ALL TABLES, LISTINGS AND FIGURES

| Table, Listing or<br>Figure Number | Title | Analysis Set |
|---|---|---|
| Table 14.2.4.6 | Percent Change from Baseline in Body Surface Area Involved for Atopic Dermatitis at Each Visit | Full Analysis Set |
| Listing 16.2.6.17 | Body Surface Area Involved for Atopic Dermatitis | Full Analysis Set |
| Listing 16.2.6.18 | Whole Body Photography | Full Analysis Set |

## APPENDIX 2. DATA DISPLAY SPECIFICATIONS – NEW TABLE 14.2.4.6, NEW LISTINGS 16.2.6.17 AND 16.2.6.18

Table 14.2.4.6
Percent Change from Baseline in Body Surface Area Involved for Atopic Dermatitis at Each Visit
Full Analysis Set

| Parameter | Statistic | GBR 830<br>(N=xx) | Placebo<br>(N=xx) |
|---|---|---|---|
| Baseline (Day 1) | n | XX | XX |
| | Mean | XX.X | XX.X |
| | SD | XX.XX | XX.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |
| Visit 3 (Day 4) | N | XX | XX |
| (=) | Mean | XX.X | XX.X |
| | SD | XX.XX | XX.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |
| Percent change from Baseline to Visit 3 (Day 4) | n | XX | XX |
| | Mean | XX.X | XX.X |
| | SD | XX.XX | XX.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| etc. | Max. | XX | XX |
| Visit 14 LOCF | n | XX | XX |
| | Mean | XX.X | XX.X |
| | SD | XX.XX | XX.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |
| Percent change from Baseline to Visit 14 | n | XX | XX |
| | Mean | XX.X | XX.X |
| | SD | XX.XX | XX.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | Xx |

Footnote: Visit 12 or Visit 14 last observation carried forward (LOCF) was calculated as the last post baseline measurement prior to or on Visit 12 or Visit 14, respectively.

Listing 16.2.6.17
Body Surface Area Involved for Atopic Dermatitis
Full Analysis Set

| Planned<br>Treatment | Site ID-<br>Subject ID | Visit (Study Day)* | Visit Date | BSA | Measurement Change from Baseline | Percent Change from<br>Baseline |
|---|---|---|---|---|---|---|
| xxxxxxx | xx-xxxxxx | 2 (1)* | DDMMMYYYY | XX | N/A | N/A |
| ΑΛΛΛΛΛΛ | ΛΛ-ΛΛΛΛΛΛ | 3 (4) | DDMMMYYYY | XX | XX | XX |
| | | 4 (8) | DDMMMYYYY | XX | XX | XX |
| | | 5 (15) | DDMMMYYYY | XX | XX | XX |
| | | 6 (22) | DDMMMYYYY | XX | XX | XX |
| | | 7 (29) | DDMMMYYYY | XX | XX | XX |
| | | 8 (32) | DDMMMYYYY | XX | XX | XX |
| | | 9 (36) | DDMMMYYYY | XX | XX | XX |
| | | 10 (43) | DDMMMYYYY | XX | XX | XX |
| | | 11 (50) | DDMMMYYYY | XX | XX | XX |
| | | 12 (57) | DDMMMYYYY | XX | XX | XX |
| | | 13 (71) | DDMMMYYYY | XX | XX | XX |
| | | 14 (85) | DDMMMYYYY | XX | XX | XX |

**Footnote:** \* indicates the baseline record; BSA = body surface area; N/A = not applicable.

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Listing 16.2.6.18 Whole Body Photography Full Analysis Set

| Planned<br>Treatment | Site ID-<br>Subject ID | Visit (Study Day)* | Visit Date | Subject<br>Consent? | Photography<br>Taken? | Results |
|---|---|---|---|---|---|---|
| xxxxxxx | xx-xxxxxx | 2 (1)* | DDMMMYYYY | XX | xx | XX |
| | | 3 (4) | DDMMMYYYY | XX | XX | XX |
| | | 4 (8) | DDMMMYYYY | XX | XX | XX |
| | | 5 (15) | DDMMMYYYY | XX | XX | XX |
| | | 6 (22) | DDMMMYYYY | XX | XX | XX |
| | | 7 (29) | DDMMMYYYY | XX | XX | XX |
| | | 8 (32) | DDMMMYYYY | XX | XX | XX |
| | | 9 (36) | DDMMMYYYY | XX | XX | XX |
| | | 10 (43) | DDMMMYYYY | XX | XX | XX |
| | | 11 (50) | DDMMMYYYY | XX | XX | XX |
| | | 12 (57) | DDMMMYYYY | XX | XX | XX |
| | | 13 (71) | DDMMMYYYY | XX | XX | XX |
| | | 14 (85) | DDMMMYYYY | XX | XX | XX |

Footnote: \* indicates the baseline record.

 $SOURCE: X: \Numerus \Studies \XXX \XXYYY \Analysis \Prod \Progs \XXXXXX.sas \\Date/time of run: DDMMYYYY HH:MM; Date of data extraction: DDMMYYYY$ 

## STATISTICAL ANALYSIS PLAN PHASE IIA

VERSION: 5.0 DATE OF PLAN:

6-JUL-17

#### **BASED ON:**

Protocol Amendment 3.0 Protocol Version 4.0 16-Feb-2017 CRF Version 5.0 3-June 2016

#### **STUDY DRUG:**

GBR 830

#### **PROTOCOL NUMBER:**

GBR 830-201

#### **STUDY TITLE:**

A Phase IIa, Double-Blind, Randomized, Placebo-controlled, Exploratory Study to Evaluate the Safety, Biological Activity and Pharmacokinetics of GBR 830 in Adult Subjects with Moderate-to-Severe Atopic Dermatitis

#### **SPONSOR:**

Glenmark Pharmaceuticals SA
Chemin de la Combeta 5,
2300 La Chaux-de-Fonds,
Switzerland

This study is being conducted in compliance with good clinical practice, including the archiving of essential documents.

## SIGNATURE PAGE

This document has been prepared and/or reviewed by:

| Miche | lic | Light |
|-------|-----|-------|
|-------|-----|-------|

Senior Statistician Numerus Ltd

Jonathan Alsop

Director Numerus Ltd Signature

11Jul 2017

This document has been reviewed and accepted by:

Hui Fang

Project Statistician Glenmark Pharmaceuticals SA

Tul. 10, 2017

Vinu C A

**Principal Scientist** Glenmark Pharmacouticals SA

Gerhard Wolff

Vice President Clinical Sciences Glenmark Pharmaceuticals SA

7th July 2017

07/10/2017

## **TECHNICAL SUMMARY REPORT (TSR)**

| Name of Sponsor/Company<br>Glenmark Pharmaceuticals SA | Individual Study Table Referring to Part of the Dossier: Volume: | (For National Authority Use Only): |
|---|---|---|
| Name of Finished Product:<br>GBR 830 | Page: | |
| Name of Active Ingredient: | | |
| GBR 830 | | |
| Title Of Study: | · | |
| A Phase IIa, Double-Blind, Randor | nized, Placebo-controlled, Exploratory Stu | dy to Evaluate the Safety, Biological |

## Investigators:

Study Center(s):

Approximately 16 sites in regions that include USA and Canada.

| Studied period (years): | Phase of development: |
|-------------------------|-----------------------|
| approx. 2 years | Phase IIa |

Activity and Pharmacokinetics of GBR 830 in Adult Subjects With Moderate-to-Severe Atopic Dermatitis

#### **Objectives:**

Primary:

- Safety and tolerability of repeated doses of GBR 830 in adult subjects with atopic dermatitis (AD).
- Effect of repeat doses of GBR 830 on biomarkers of disease activity in adult subjects with AD.

#### Secondary:

- Effect of GBR 830 on additional efficacy parameters in adult subjects with AD.
- Pharmacokinetics (PK) of repeated doses of GBR 830 in adult subjects with AD.
- Immunogenicity of GBR 830 in adult subjects with AD.

#### Exploratory:

• Additional exploratory objectives to understand the mechanism of GBR 830 including effect on cellular infiltrates and immune pathways.

#### Methodology:

The study is a phase IIa, double-blind, randomized, placebo-controlled, repeated dose study to evaluate safety, biological activity and PK of GBR 830 in adult subjects with AD. The study will be conducted in approximately 16 centers in US/Canada. The study will be conducted in three phases: screening phase, treatment phase and follow-up phase.

During the screening phase, after providing informed consent all subjects will be screened for eligibility prior to inclusion in the study and sufficient numbers of subjects will be screened to ensure at least 40 subjects meeting the eligibility criteria will be enrolled. At screening, subjects will be assessed on Eczema Area and Severity Index (EASI), Investigator's Global Assessment (IGA), Severity Scoring of Atopic Dermatitis (SCORAD) and Body Surface Area (BSA) rating scales for AD. Subjects will be withdrawn from use of other medication being used to control their AD as mentioned in prior and concomitant medication section. On Day 1, prior to dosing, subjects will be reassessed on EASI, IGA, SCORAD and BSA rating scales for AD to ensure that they qualify for the study. A sufficient number of patients will be randomized such that approximately 40 evaluable patients complete at least the Day 29 visit. Approximately 60 to 80 patients are planned to be randomized in a ratio of 3:1 to receive GBR 830 (10 mg/kg) or placebo, in a two-arm, parallel design study. Subjects who meet eligibility criteria will undergo Day 1/baseline assessments, randomization, and then receive the first intravenous (IV) infusion of GBR 830 or placebo. Each subject will receive two doses of GBR 830 or placebo administered 4 weeks apart on Day 1 and Day 29. Subjects will be closely monitored at the study site for 6 hours after the first infusion (Day 1/baseline) and for 3 hours after the next dose (Day 29). Subjects will return for follow-up visits as mentioned in Appendix 1 - schedule of events. The study site will contact subjects by telephone approximately 24 hours after each infusion (Days 2 and 30) for concomitant medication and procedures, and a general adverse event (AE) query.

Figure 1: Study Design Schematic



Apart from the dosing visits, subjects will be seen in the clinic on Days 4, 8, 15, 22, 29, 32, 36, 43, 50, 57, 71 and the end of study visit occurs on Day 85 (week 12) for study assessments and PK sample collection.



\* Visits and assessments done in relation to the second infusion will be calculated from the actual day/start time of the second infusion. This applies to V8 to V11, inclusively. For V12, V13, and V14, the time points for assessment will be 672hr, 1008hr, and 1344hr, respectively, from the start time of the second infusion.

#### Number of Subjects (planned and analyzed):

Approximately 60 to 80 adult subjects with AD are planned to be randomized using a ratio of 3 active: 1 placebo, to receive either GBR 830 (10mg/kg) or placebo.

A sufficient number of patients will be randomized such that approximately 40 evaluable patients complete at least the Day 29 visit.

#### Diagnosis and main criteria for inclusion (see protocol section 9):

The target study population is adult males and females with chronic moderate-to-severe AD as defined by EASI score of  $\geq$  12; SCORAD of  $\geq$  20; IGA score of  $\geq$  3 at baseline and with history of inadequate response to topical therapies.

#### Inclusion criteria:

Subjects eligible for enrolment in the study must meet all of the following criteria:

- 1. Male or female subjects, age  $\geq$  18 years at the time of informed consent with physician diagnosis of AD for > 1 year, diagnosis of AD as defined by the Hanifin and Rajka (Hanifin et al., 1980) criteria for AD.
- 2. AD involvement of  $\geq 10\%$  body surface area (BSA) prior to randomization
- 3. EASI score of ≥ 12 prior to randomization; SCORAD of ≥ 20 prior to randomization; baseline IGA score of ≥ 3 prior to randomization; and history of inadequate response to a stable (> 1 month) regimen of class 3 or higher strength topical corticosteroids (TCS), or calcineurin inhibitors or for whom topical treatments are otherwise inadvisable (e.g., because of important side effects or safety risks).
- 4. Subject's body mass index (BMI) should be within the range 18.5-35 kg/m² (inclusive); weight must be ≥ 50 kg.
- 5. Subjects deemed fit to receive the study medication, as determined by medical history, vital signs, physical examinations, Electrocardiogram (ECG), laboratory studies, and other tests performed within 30 days prior to drug administration, as judged by the Investigator.
- 6. Subjects must agree to the following requirements during the study:
  - a) Women of child-bearing potential and men with partners of child-bearing potential must ensure that two effective means of contraception are used, by them and/or their partners for the period between signing of informed consent and a minimum of 180 days after the last dose of study drug.

Acceptable forms of effective contraception include:

- Established use of oral, injected, or implanted hormonal methods of contraception.
- Tubal ligation.
- Placement of an intrauterine device (IUD) or intrauterine system (IUS).
- Barrier methods only when used consistently with spermicidal foam/gel/film/cream or suppository. Acceptable barrier methods include the following:
  - i. Male or female condom.
  - ii. Occlusive cap (diaphragm or cervical/vault caps).
- Male sterilization (with post-vasectomy documentation of the absence of sperm in the ejaculate) (For female patients on the study, the vasectomized male partner should be the sole partner for that patient). If a subject cannot provide written documentation of male sterilization, a verbal statement from the subject will suffice.
- Maintenance of abstinence when this is in line with the preferred and usual lifestyle of the patient (i.e., not periodic abstinence, such as during ovulation) judged reliable by the Investigator.

Patients in relation with a same-sex partner do not need to use contraception, if he/she is the sole partner for that patient)

Of the acceptable forms of effective contraception, at least one method needs to be a barrier method.

- b) Male patents should agree not to donate sperm until 180 days after administration of the last dose of the study medication. Female subjects should not donate eggs for 180 days following investigational product administration.
- c) All female subjects must be non-pregnant and non-lactating and test negative for pregnancy at the time of screening and prior to randomization.
- 7. Female subjects of non-child-bearing-potential (i.e. are postmenopausal or permanently sterilized [bilateral oophorectomy, hysterectomy, bilateral salpingectomy]). Such subjects will not be required to use contraception. Postmenopausal is defined as at least 1 year post cessation of menses (without an alternative medical cause) with follicle stimulating hormone (FSH) ≥ 40.0 mIU/mL.
- 8. Provide written informed consent.
- 9. Willing and able to comply with all aspects of the protocol including willingness to undergo 4 on study skin biopsies.

#### Exclusion criteria:

Subjects meeting any of the following criteria must not be enrolled in the study:

- 1. Subjects with a history of drug or other allergy considered clinically significant in the opinion of the Investigator, which contraindicates participation or a previous history of hypersensitivity to murine proteins.
- 2. Subjects who have had a live vaccination within 12 weeks before randomization, or intend to have a live vaccination during the course of the study, or have participated in a vaccine clinical trial within 12 weeks prior to randomization.
- 3. History of a serious local infection, systemic infection, or gastrointestinal infection within 12 weeks of baseline, infections requiring systemic antibiotic/ anti-viral /anti-parasitic/ anti-fungals within 4 weeks of baseline; evidence of clinically significant active infection, or fever ≥38.0°C (100.4°F) within one week of randomization.
- 4. Subjects who have evidence of active or latent tuberculosis as documented medical history, or test positive for QuantiFERON Gold Blood TB Test.
- 5. Subjects with evidence of skin conditions at screening that would interfere with evaluations of the study drug.
- 6. Treatment with systemic corticosteroids within 4 weeks before randomization, and topical steroids/tacrolimus and/or pimecrolimus within 1 week before the randomization (except emollients, and mild steroids (class 6 or 7)
- 7. Treatment with systemic therapy for AD (such as psoralen and ultraviolet A light therapy, cyclosporine, methotrexate, mycophenolate mofetil, thioguanine, hydroxyurea, sirolimus, azathioprine), or phototherapy (including ultraviolet B or self-treatment with tanning beds or therapeutic sunbathing) within the 4 weeks before randomization or other drugs with potential for immunosuppression such as cytotoxic agents or cyclophosphamide taken within 4 weeks prior to randomization.

- 8. Any cell-depleting agents including but not limited to rituximab: within 6 months prior to the baseline visit, or until lymphocyte and CD 19+ lymphocyte counts return to normal, whichever is longer. Other biologics: within 5 half-lives or 8 weeks prior to the baseline visit, whichever is longer. Allergen immunotherapy within 6 months before the baseline visit.
- 9. Subjects who are immunocompromised, have had a recent (within 3 months before randomization) or current serious systemic or local infection (including infectious mononucleosis-like illness or herpes zoster) suggestive of immunocompromise.
- 10. Subjects who have current or a history of lymphoproliferative disease or history of malignant disease; or signs or symptoms suggestive of possible lymphoproliferative disease, including lymphadenopathy or splenomegaly; or active primary or recurrent malignant disease.
- 11. Subjects with history or presence of other inflammatory or auto-immune disease or rheumatological or joint diseases other than AD.
- 12. History of parasitic infections within 1 year before randomization.
- 13. History of alcohol or drug abuse or dependence within 2 years of the screening visit.
- 14. Subjects with a positive result from the drug and alcohol screen.
- 15. Subjects who test positive for disease markers of Human immunodeficiency virus (HIV), Hepatitis B or Hepatitis C.
- **16.** Subjects with an abnormal ECG (including a QTc >450 msec for men, >460 msec for women) considered clinically significant in the opinion of the Investigator at screening and/prior to randomization (QTc calculated based on Fridericia's formula).
- 17. Subjects with lab values, which are significantly different from normal references ranges and/or judged clinical significant by the Investigator, including but not limited to:
  - a) Subjects with estimated glomerular filtration rate (eGFR) <60 mL/min/1.73m<sup>2</sup> as determined by the modification of diet in renal diseases (MDRD) method.
  - b) Alanine amino transferase (ALT) or Aspartate amino transferase (AST)  $\geq$  2.5 times upper limit of normal (ULN), and/or serum total bilirubin  $\geq$  1.5 times ULN, at screening.
  - c) Hemoglobin (Hb) value less than 9 g/dL at screening.
  - d) Absolute neutrophil count  $\leq 1,500/\mu L$  or absolute lymphocyte count  $\leq 800/\mu L$  or platelet count  $\leq 150,000/\mu L$  or any abnormal evaluations judged clinically significant by the Investigator at screening and prior to randomization.
- 18. Subjects with any evidence of organ dysfunction or any clinically significant medical history or findings in physical examinations or investigations or has a clinical condition or receiving therapy that, in the opinion of the Investigator, would make the subjects unsuitable for study.
- 19. Subjects with a history of current or previous psychiatric illnesses or previous psychiatric events that would either put the subject at undue risk or interfere with study procedures according to the investigator.
- 20. Treatment with an investigational drug within 8 weeks or within 5 half-lives, if known (whichever is longer), before the baseline visit.

#### Test product, dose and mode of administration:

GBR 830 (10 mg/kg) will be diluted in normal saline and administered as IV infusion over 60 minutes. Two doses will be administered at an interval of once every 4 weeks.

#### **Duration of treatment:**

Screening phase (4 weeks), study duration including treatment phase and follow-up (12 weeks), total study duration for each subject (16 weeks).

Screening phase occurs on days -30 to -1.

Treatment phase occurs on day 1 and 29.

Follow-up occurs on days 4, 8, 15, 22, 32, 36, 43, 50, 57, 71, and 85.

#### Reference therapy, dose and mode of administration:

Placebo (formulation buffer) will be diluted in normal saline and administered as IV infusion over 60 minutes. Two doses will be administered at an interval of once every 4 weeks.

#### **Criteria for evaluation (see protocol section 8):**

#### Primary Endpoints:

- All treatment emergent adverse events (TEAEs) occurring in the study, in terms of nature, onset, duration, severity, relationship and outcome of adverse events (AEs) and serious AEs (SAEs), in adult subjects with moderate-to-severe AD.
- Effect of GBR 830 in adult subjects with AD in terms of change from baseline in the active AD mRNA expression signature and the pathologic epidermal phenotype measures obtained from skin biopsies.

#### Secondary Endpoints:

- Proportion of subjects who achieve an IGA score of 0 or 1 at each study visit.
- Proportion of subjects who achieve an EASI 50 and 75 response at each study visit.
- Percent improvement in clinical scores EASI, SCORAD, IGA, BSA (Body surface area), Pruritus numeric rating scale (NRS) and Dermatology Life Quality Index (DLQI) from baseline to each visit.
- Changes from baseline AD activity as determined by changes in Transepidermal water loss (TEWL).
- PK of GBR 830 in adult subjects with moderate to severe AD in terms of  $C_{max}$ ,  $AUC_{0-tau}$ ,  $AUC_{0-\infty}$ , and  $AUC_{0-t_{1}}$ ,  $t_{1/2}$ , volume of distribution, clearance and other parameters assessed as relevant after the first and last doses.
- Anti-drug antibodies (ADA) to GBR 830 to evaluate immunogenicity.

#### Exploratory Endpoints (change from baseline in levels of):

- Cytokines and chemokines in serum: Interleukin (IL)-22, IL-13, chemokine ligand (CCL)-17 (TARC = thymus and activation-regulated chemokine), Eotaxin (CCL11), TSLP, CXCL10 (IP-10), CCL2 (MCP-1), CCL20 (MIP3A), CCL22 (MDC), CCL3 (MIP-1α), CCL4 (MIP-1β), CCL13 (MCP-4), CXCL11 (IP-9; I-TAC) and CXCL9 (MIG).
- Leukocyte sub-population cell counts (Total T, T helper, Cytotoxic T, T<sub>regs</sub> Memory T cells).
- Cellular infiltrates (T-cells, Dendritic cells) as assessed by CD3, FcEpsilon RI, and OX40L, OX40, and MBP.
- $\bullet$  Serum total Immunoglobulin E (IgE), serum soluble OX40 (sOX40), serum soluble OX40 ligand (sOX40L), and circulating eosinophil counts.

#### Safety:

• Safety and tolerability assessments of GBR 830 will include AEs, SAEs, vital signs, laboratory parameters, ECGs, and physical examinations.

#### Statistical methods:

Determination of Sample Size

No formal sample size calculation will be performed for this study. The sample size chosen is based on experience from previous studies of similar nature. Subjects, who are permanently discontinued from study drug due to reasons other than an AE and before the first post baseline skin biopsies or before receiving two doses of study drug, will not be considered evaluable for the Biological Analysis Set. The sample size of 60 to 80 adult patients with AD randomized in ratio of 3:1 (GBR 830 vs placebo), with approximately 40 evaluable patients, is considered to be sufficient to provide descriptive information on the PK, safety, tolerability and potential efficacy of GBR 830

A patient will be considered evaluable if he/she completes the Day 29 visit and has at least one post-baseline skin biopsy (Visit 7) and received two doses of study drug (Visit 7).

Efficacy Analyses

Analysis of Primary Efficacy Endpoint(s)

The primary endpoint will be absolute change from baseline in the active AD mRNA expression signature.

Analysis of Secondary Efficacy Endpoint(s)

The statistical methods, including methods for the handling of missing data, for analyzing the secondary endpoints will be fully described in the sections below.

Pharmacokinetic, Pharmacodynamic, Pharmacogenomic, and Other Biomarker Analyses

Pharmacokinetic Analyses

PK parameters will be summarized in tabular and graphic form. Results of exploratory analyses will be summarized.

Pharmacodynamic, Pharmacogenomic, and Other Biomarker Analyses

PD parameters will be summarized in tabular and graphic form. Results of exploratory analyses will be summarized.

Safety Analyses

Adverse events will be summarized by system organ class, preferred term and treatment group. Subjects will be counted only once for each preferred term, system organ class, and by the highest severity of an event. Vitals, physical examinations and ECG evaluations will be summarized with descriptive statistics. Laboratory evaluations will be summarized with descriptive statistics at each visit, and change from baseline summarized for each post baseline visit. Laboratory measurements will also be summarized based on the number and percentage of subjects above or below a pre-specified threshold for each test.

## **TABLE OF CONTENTS**

| 1. | LIST OF ABBREVIATIONS | 19 |
|---|---|---|
| 2. | INTRODUCTION | 22 |
| 3. | STUDY OBJECTIVES AND ENDPOINTS | 23 |
| 3.1. | Study Objectives | 23 |
| 3.1.1. | Primary Objective | 23 |
| 3.1.2. | Secondary Objective | 23 |
| 3.1.3. | Exploratory Objective | 23 |
| 3.2. | Study Endpoints | 23 |
| 3.2.1. | Primary Endpoints | 23 |
| 3.2.2. | Secondary Endpoints | 24 |
| 3.2.3. | Exploratory endpoints | 24 |
| 4. | STUDY DESIGN | 25 |
| 4.1. | Summary of Study Design | 25 |
| 4.2. | Definition of Study Drugs | 26 |
| 4.3. | Sample Size Considerations | 27 |
| 4.3.1. | Sample Size Justifications | 27 |
| 4.3.2. | Sample Size Re-estimation | 27 |
| 4.4. | Randomization | 27 |
| 4.5. | Clinical Assessments | 28 |
| 4.5.1. | Efficacy Assessments | 28 |
| 4.5.2. | Pharmacokinetic, Pharmacodynamic and Biomarker Assessments | 29 |
| 4.5.3. | Safety Assessments | 31 |
| 4.5.4. | Schedule of Assessments | 31 |
| 5. | PLANNED ANALYSES | 35 |
| 5.1. | Interim Analyses | 35 |
| 5.2. | Final Analyses | 35 |
| 6. | GENERAL CONSIDERATIONS FOR DATA ANALYSES AND HANDLING | 36 |
| 6.1. | General Summary Table and Individual Subject Data Listing Considerations | 36 |
| 6.2. | General Post Text Summary Table and Individual Subject Data Listing Format Considerations | |

| 6.3. | Data Management | 37 |
|---|---|---|
| 6.4. | Data Presentation Conventions | 38 |
| 6.5. | Analysis Populations | 39 |
| 6.5.1. | Screen Failures | 39 |
| 6.5.2. | Full Analysis Set (FAS) Population | 39 |
| 6.5.3. | Biological Activity Set (BAS) Population | 39 |
| 6.5.4. | Safety Analysis Set (SAF) Population | 39 |
| 6.5.5. | Pharmacokinetic Analysis Set (PKAS) Population | 40 |
| 6.6. | Baseline Definition | 40 |
| 6.7. | Derived and Transformed Data | 40 |
| 6.7.1. | Baseline Age | 40 |
| 6.7.2. | Age at AD diagnosis | 40 |
| 6.7.3. | Study Day | 40 |
| 6.7.4. | Change from Baseline | 41 |
| 6.7.5. | Visit 12 and Visit 14 LOCF Visits | 41 |
| 6.7.6. | End of Study Visit | 41 |
| 6.7.8. | Multiple Assessments | 41 |
| 6.7.9. | Missing Efficacy Endpoints. | 41 |
| 6.7.10. | Missing Start and Stop Dates for Prior and Concomitant Medication | 42 |
| 6.7.11. | Missing Start and Stop Dates for Adverse Events | 42 |
| 7. | STUDY POPULATION | 43 |
| 7.1. | Subjects Disposition | 43 |
| 7.2. | Screen Failures | 44 |
| 7.3. | Protocol Deviations | 44 |
| 7.4. | Demographic and Baseline Characteristics | 45 |
| 7.5. | Listing of Subject Inclusion and Exclusion Criteria | 46 |
| 7.6. | Medical History and Medical Conditions Present at Entry | 46 |
| 7.7. | Prior Medication History | 48 |
| 7.7.1. | Diagnosis Related Medication History | 49 |
| 7.7.2. | Non-Diagnosis Related Medication History | 49 |
| 7.8. | Baseline Physical Examination | 49 |
| 7.9. | Baseline Vital Signs | 50 |

| 7.10. | Baseline Laboratory Data | 51 |
|---|---|---|
| 7.11. | Baseline ECG | 51 |
| 7.12. | Baseline Clinical Scores | 52 |
| 7.13. | Baseline Skin Biopsy (Non-lesion only) | 52 |
| 8. | EFFICACY | 53 |
| 8.1. | General Considerations | 53 |
| 8.2. | Testing Statistical Assumptions Including Comparability at Baseline | 53 |
| 8.3. | Statement of the Null and Alternate Hypotheses | 53 |
| 8.4. | Subgroup Analyses | 53 |
| 8.5. | Multiple Comparisons and Multiplicity | 53 |
| 8.6. | Analysis of the Primary Efficacy Endpoint | 54 |
| 8.6.1. | Primary Efficacy Analysis | 54 |
| 8.6.2. | Sensitivity Analyses of the Primary Efficacy Endpoint | 55 |
| 8.7. | Analysis of the Secondary Endpoints | 55 |
| 8.7.1. | Proportion of subjects who achieve an IGA score of 0 or 1 at each study visit | 55 |
| 8.7.2. | Proportion of subjects who achieve an EASI 50 and 75 responses at each study visit | 55 |
| 8.7.3. | Analysis of covariance EASI scores | 56 |
| 8.7.4. | Percent improvement in clinical scores EASI, SCORAD, IGA, Pruritus NRS and DLQI from baseline to each visit | 56 |
| 8.7.5. | Changes from baseline AD activity as determined by changes in Transepidermal water loss (TEWL) | 56 |
| 8.7.6. | Anti-drug antibodies (ADA) to GBR 830 to evaluate immunogenicity | 57 |
| 8.8. | Analysis of the Exploratory Endpoints | 57 |
| 8.8.1. | Change from Baseline in Cytokines in serum | 57 |
| 8.8.2. | . Change from Baseline in Leukocyte sub-population cell counts (Total T, T helper, Cytotoxic T, T <sub>regs</sub> , Memory T cells) | |
| 8.8.3. | Change from Baseline in Cellular infiltrates (T-cells, dendritic cells) as assessed by CD3, FcEpsilon RI, OX40L, OX40 and MBP | |
| 8.8.4. | Change from Baseline in Serum total Immunoglobulin E (IgE), serum soluble OX40 (sOX40), serum soluble OX40 ligand (sOX40L) and circulating eosinophil counts. | 58 |
| 8.9. | Summary of Reasons for Efficacy Non-Evaluability/Exclusion from Efficacy Analyses | 58 |

| 9. | SAFETY AND TOLERABILITY | |
|---|---|---|
| 9.1. | Treatment Emergent Adverse Event Preferred Term and Body/Organ System Summary Tables | |
| 9.1.1. | 1. Summaries of Adverse Event Incidence Rates for All Subjects | |
| 9.1.2. | Summaries of Adverse Incidence Rates for Serious Adverse Events (SAE),<br>Adverse Event Dropouts, and Death | 60 |
| 9.2. | Total Duration of Therapy, Average Daily Dose, Maximum Daily Dose, Final Daily Dose of Study Medication, and Compliance | 61 |
| 9.3. | Concomitant Medications and Non-Drug Treatments | 61 |
| 9.4. | Routine Laboratory Data | 61 |
| 9.4.1. | Laboratory tests | 62 |
| 9.5. | Vital Signs | 64 |
| 9.6. | Physical Examination | 65 |
| 9.7. | ECG | 65 |
| 9.8. | Rescue Medication | 66 |
| 9.9. | Study Termination Status | 67 |
| 10. | CLINICAL PHARMACOLOGY DATA ANALYSES | 68 |
| 10.1. | Pharmacokinetic/ Pharmacodynamic Analyses | 68 |
| 10.1.1. | Dosing intervals | 68 |
| 10.1.2. | Analysis of Parameters | 68 |
| 10.1.3. | Handling of values below the limit of quantification | 71 |
| 10.1.1. | Treatment of outliers | 72 |
| 11. | CHANGES FROM THE PLANNED PROTOCOL ANALYSIS | 73 |
| 11.1. | Shift Tables | 73 |
| 11.2. | Exploratory Cytokines Analysis | 73 |
| APPENDI | IX 1. SCHEDULE OF EVENTS | 74 |
| APPEND | IX 2. TABLE OF CONTENTS FOR DATA DISPLAY SPECIFICATIONS | 78 |
| APPEND | IX 3. DATA DISPLAY SPECIFICATIONS | 86 |
| 12. | REFERENCES | 181 |

| Glenmark Pharmaceutical SA |
|--------------------------------------------------|
| Statistical Analysis Plan – Protocol GBR 830-201 |

## LIST OF TABLES

| Table 1: | List of Abbreviations | 19 |
|----------|-----------------------|----|
| Table 3: | PK Parameters | 68 |

| Glenmark Pharmaceutical SA |
|--------------------------------------------------|
| Statistical Analysis Plan – Protocol GBR 830-201 |

## LIST OF FIGURES

| Figure 1: | Study Design Schematic | 26 |
|-----------|------------------------|----|
| Figure 2: | Study Flow Chart | 26 |

## 1. LIST OF ABBREVIATIONS

**Table 1:** List of Abbreviations

| Abbreviation | Term |
|----------------------|-----------------------------------------|
| AD | Atopic dermatitis |
| ADA | Anti-drug antibodies |
| AE | Adverse event |
| ALT | Alanine aminotransferase |
| ANCOVA | Analysis of covariance |
| ANOVA | Analysis of variance |
| AST | Aspartate amino transferase |
| AUC <sub>0-t</sub> | Area under the curve (0 to t) |
| AUC <sub>0-tau</sub> | Area under the curve (0 to tau) |
| $AUC_{0-\infty}$ | Area under the curve (0 to infinity) |
| CCL | Chemokine ligand |
| СМН | Cochran Mantel-Haenszel |
| CV | Coefficient of variation |
| BLQ | Below the lower limit of quantification |
| BMI | Body mass index |
| BSA | Body surface area |
| $C_{\text{max}}$ | Maximum observed serum concentration |
| CRO | Contract research organization |
| CSR | Clinical study report |
| DOB | Date of birth |
| DLQI | Dermatology Life Quality Index |
| DP | Drug product |
| EASI | Eczema Area and Severity Index |
| ECG | Electrocardiogram |
| eGFR | Estimated glomerular filtration rate |
| ELISA | Enzyme-linked immunosorbent assay |
| FSH | Follicle stimulating hormone |
| GCP | Good clinical practices |

| GGT | Gamma-glutamyl transferase |
|---|---|
| Hb | Hemoglobin |
| HIV | Human immunodeficiency virus |
| ICD-9 | International Classification of Diseases – 9 <sup>th</sup> Edition |
| IEC | Independent Ethics Committee |
| IGA | Investigator's Global Assessment |
| IgE | Immunoglobulin E |
| IHC | Immunohistochemistry |
| IL | Interleukin |
| IRB | Institutional review board |
| IV | Intravenous |
| LOCF | Last observation carried forward |
| LS | Lesion skin |
| MAR | Missing at random |
| MedDRA | Medical Dictionary for Regulatory Activities Terminology |
| MDRD | Modification of diet in renal disease |
| MMRM | Mixed model repeated measures |
| NLS | Non-lesion skin |
| PK | Pharmacokinetic |
| RO | Receptor occupancy |
| s.d. | Standard deviation |
| s.e. | Standard error |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| SCORAD | Severity Scoring of Atopic Dermatitis |
| t <sub>1/2</sub> | Elimination half life |
| TARC | Thymus and activation-regulated chemokine |
| TCS | Topical corticosteroids |
| TEAE | Treatment emergent adverse event |
| TEWL | Trans epidermal water loss |
| $T_{regs}$ | Regulatory T cells |
| TS | Transdermal Delivery System-Placebo |

| ULN | Upper limit of normal |
|---|---|
| V | Visit |
| VAS | Visual Analogue Scale |
| WBC | White blood cell count |
| WHO (DDE) World Health Organization (Drug Dictionary Enhanced) | |

## 2. INTRODUCTION

The purpose of this statistical analysis plan (SAP) is to describe the planned analyses and data displays to be included in the Clinical Study Report (CSR) for Protocol GBR 830-201.

| Protocol Revision Chronology: | | |
|---|---|---|
| Protocol | 12-OCT-2015 | Original. |
| Amendment 1 | 19-MAY-2016 | Amendment No. 01: The changes of this amendment were non-substantial. |
| Amendment 2 | 07-NOV-2016 | Amendment No. 02: The changes of this amendment were substantial and are detailed in the protocol version 3.0. |
| Amendment 3 | 16-FEB-2017 | Amendment No. 03: The changes of this amendment were substantial and non-substantial and are detailed in the protocol version 4.0. |

This SAP was developed in accordance with ICH E9 guidelines. All decisions regarding final analysis, as defined in this SAP document, will be made prior to database freeze (unblinding) of the study data (unless otherwise stated).

#### 3. STUDY OBJECTIVES AND ENDPOINTS

## 3.1. Study Objectives

#### 3.1.1. Primary Objective

The primary study objectives are as follows:

- Safety and tolerability of repeated doses of GBR 830 in adult subjects with atopic dermatitis (AD).
- Effect of repeated doses of GBR 830 on biomarkers of disease activity in adult subjects with AD.

#### 3.1.2. Secondary Objective

The secondary study objectives are as follows:

- Effect of GBR 830 on clinical efficacy parameters in adult subjects with AD.
- Pharmacokinetics (PK) of repeated doses of GBR 830 in adult subjects with AD.
- Immunogenicity of GBR 830 in adult subjects with AD.

#### 3.1.3. Exploratory Objective

The exploratory study objective is as follows:

• Additional exploratory objectives to understand the mechanism of GBR 830 including effect on cellular infiltrates and immune pathways.

## 3.2. Study Endpoints

#### 3.2.1. Primary Endpoints

The primary endpoints of the study are as follows:

- All treatment emergent adverse events (TEAEs) occurring in the study, in terms of nature, onset, duration, severity, relationship and outcome of adverse events (AEs) and serious AEs (SAEs), in adult subjects with moderate-to-severe AD.
- Effect of GBR 830 in adult subjects with AD in terms of change from baseline in the active AD mRNA expression signature and the pathologic epidermal phenotype measures obtained from skin biopsies.

#### 3.2.2. Secondary Endpoints

The secondary endpoints of the study are as follows:

- Proportion of subjects who achieve an Investigator's Global Assessment (IGA) score of 0 or 1 at each study visit.
- Proportion of subjects who achieve an Eczema Area and Severity Index (EASI) 50 and 75 response at each study visit.
- Percent improvement in clinical scores EASI, Severity Scoring of Atopic Dermatitis (SCORAD), IGA, Body surface area (BSA), Pruritus numerical rating score (NRS) and Dermatology Life Quality Index (DLQI) from baseline to each visit.
- Changes from baseline AD activity as determined by changes in Transepidermal water loss (TEWL).
- PK of GBR 830 in adult subjects with moderate to severe AD in terms of C<sub>max</sub>, AUC<sub>0-tau</sub>, AUC<sub>0-∞</sub>, and AUC<sub>0-t</sub>, t<sub>√2</sub>, volume of distribution, clearance and other parameters assessed as relevant after the first and last doses.
- Anti-drug antibodies (ADA) to GBR 830 to evaluate immunogenicity.

### 3.2.3. Exploratory endpoints

The exploratory endpoints of the study are as follows:

- Cytokines in serum: IL-22, IL-13, CCL17 (TARC = Thymus and activation-regulated chemokine), Eotaxin (CCL11), TSLP, CXCL10 (IP-10), CCL2 (MCP-1), CCL20 (MIP3A), CCL22 (MDC), CCL3 (MIP-1α), CCL4 (MIP-1β), CCL13 (MCP-4), CXCL11 (IP-9; I-TAC), and CXCL9 (MIG)
- Leukocyte sub-population cell counts (Total T, T helper, Cytotoxic T, T<sub>regs</sub>, Memory T cells,).
- Cellular infiltrates (T-cells, Dendritic cells) as assessed by CD3, FcEpsilon RI, OX40, MB, and OX40L.
- Serum total Immunoglobulin E (IgE), serum soluble OX40 (sOX40), serum soluble OX40 ligand (sOX40L), and circulating eosinophil counts.

#### 4. STUDY DESIGN

### 4.1. Summary of Study Design

The study is a phase IIa, double-blind, randomized, placebo-controlled, repeated dose study to evaluate safety, biological activity and PK of GBR 830 in adult subjects with AD. The study will be conducted in approximately 16 centers in US/Canada. The study will be conducted in three phases: screening phase, treatment phase and follow-up phase.

During the screening phase, after providing informed consent, all subjects will be screened for eligibility prior to inclusion in the study and sufficient number of subjects will be screened to ensure at least 40 subjects meeting the eligibility criteria will be enrolled. At screening, subjects will be assessed on EASI, IGA, SCORAD and BSA rating scales for AD. Subjects will be withdrawn from use of other medication being used to control their AD. On Day 1, prior to dosing, subjects will be reassessed on EASI, IGA, SCORAD and BSA rating scales for AD to ensure that they qualify for the study.

A sufficient number of subjects will be randomized such that approximately 40 evaluable subjects complete at least the Day 29 visit. Approximately 60 to 80 subjects are planned to be randomized in a ratio of 3:1 to receive GBR 830 (10 mg/kg) or placebo, in a two-arm, parallel design study.

Subjects who meet eligibility criteria will undergo Day 1/baseline assessments, randomization, and then receive the first intravenous (IV) infusion of GBR 830 or placebo. Each subject will receive two doses of GBR 830 or placebo administered 4 weeks apart on Day 1 and Day 29. Subjects will be closely monitored at the study site for 6 hours after the first infusion (Day 1/baseline) and for 3 hours after the next dose (Day 29). Subjects will return for follow-up visit is as mentioned in Appendix 1 – schedule of events. The study site will contact subjects by telephone approximately 24 hours after each infusion (Days 2 and 30) for concomitant medications and procedures, and a general AE query.

Apart from the dosing visits, subjects will be seen in the clinic on Day 4, 8, 15, 22, 29, 32, 36, 43, 50, 57, 71 and the end of study visit occurs on Day 85 (week 12) for study assessments and PK sample collection.

Skin punch biopsy samples for biomarker analysis will be collected at Day 1/baseline, Day 29 and Day 71. Analyses will be performed where samples are available. A gene/mRNA expression profiling will be performed to evaluate the effects of OX40 blockade on both lesional and non-lesional skin from subjects with AD. Changes in gene expression in the AD transcriptome of lesional skin in comparison to a non-lesional molecular phenotype will be used to evaluate treatment-associated effects. In addition any correlation with improvements in disease activity and clinical outcomes will also be evaluated.

The end of the study will be the date of the last study visit for the last subject in the study.

An overview of the study design is shown in Figure 1.
Figure 1: Study Design Schematic



Figure 2: Study Flow Chart



\*The timing of the visits and assessments done in relation to the second infusion will be calculated from the actual day/start time of the second infusion. This applies to V8 to V11, inclusively. For V12, V13, and V14, the time points for assessment will be 672hr, 1008hr, and 1344hr, respectively, from the start time of the second infusion.

# 4.2. Definition of Study Drugs

Investigational products:

Test drug: GBR 830 (10mg/kg) drug product (DP), diluted in normal saline and administered as IV infusion over 60 minutes. Two doses administered at an interval of once every 4 weeks.

Placebo: Formulation buffer, diluted in normal saline and administered as IV infusion over 60 minutes. Two doses administered at an interval of once every 4 weeks.

### 4.3. Sample Size Considerations

#### **4.3.1.** Sample Size Justifications

No formal sample size calculations were performed for this study. The sample size chosen is based on experience from previous studies of similar nature. Subjects, who are permanently discontinued from study drug due to reasons other than an AE and before the first post baseline skin biopsies (Visit 7) or before receiving two doses of study drug (Visit 7), will be replaced. The sample size of 40 adult subjects with AD randomized in ratio of 3:1 (GBR 830 versus placebo) is considered to be sufficient to provide description information on the PK, safety, tolerability and potential efficacy of GBR 830.

#### 4.3.2. Sample Size Re-estimation

The sample size for this study has not been formally re-estimated. However, at the time of SAP writing the number of subjects randomized has been increased to 60 to 80 subjects, in order to allow for high levels of subject withdrawal and provide approximately 40 evaluable subjects.

#### 4.4. Randomization

Following confirmation of eligibility, subjects were assigned a randomization number through interactive voice response system (IVRS)/interactive web response system (IWRS) central randomization. The randomization scheme and identification for each subject will be included in the final CSR for this study. The randomization list was generated using Statistical Analysis System (SAS) Version 9.1.3 or higher. All eligible subjects entering the study were randomized to one of the two treatment arms. If a subject discontinues from the study, the subject number will not be re-used and the subjects will not be allowed to re-enter the study.

Subjects are randomly assigned to receive either GBR 830 or placebo in a 3:1 ratio. A randomization number that uniquely identified each subject and the subject's treatment is assigned on Day 1. Randomization numbers are allocated from the schedule in strict chronological order.

A sufficient number of subjects (approximately 60 to 80) will be randomized such that approximately 40 evaluable subjects complete at least the Day 29 visit.

• For subjects randomized prior to protocol version 3 (amendment 2) who do not complete at least the Day 29 visit: A replacement patient will be given the patient number corresponding to the person he/she is replacing plus 100. For example, at site 01, if randomized patient 011001 is to be replaced, the subject number for the replacement randomized patient would be 011101. Randomized replacement patient 011101 will receive the same treatment assignment (via IWRS) as the original randomized patient 011001 had received.

• For subjects randomized after protocol version 3 (amendment 2 who do not complete at least the Day 29 visit: Replacement of subjects (to receive the same treatment assignment as the original subject he/she is replacing) will no longer be performed.

Randomization will be done using IVRS/IWRS software.

#### 4.5. Clinical Assessments

#### 4.5.1. Efficacy Assessments

#### 4.5.1.1. EASI

The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. Four AD disease characteristics will be assessed for severity by the investigator or designee on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement will be assessed as a percentage by body area of head, trunk, arms, and legs and converted to a score of 0 to 6 (Hanifin et al., 2001).

#### 4.5.1.2. SCORAD

The SCORAD is a validated tool used in clinical research and clinical practice that was developed to standardize the evaluation of the extent and severity of AD (Dermatology, 1993). The extent of AD is assessed as a percentage of each defined body area and reported as the sum of all areas, with a maximum score of 100% (assigned as "A" in the overall SCORAD calculation). The severity of 6 specific symptoms of AD is assessed using the following scale: none (0), mild (1), moderate (2), or severe (3) (for a maximum of 18 total points, assigned as "B" in the overall SCORAD calculation). Subjective assessment of itch and sleeplessness is recorded for each symptom by the subject or relative on a visual analogue scale (VAS), where 0 is no itch (or sleeplessness) and 10 is the worst imaginable itch (or sleeplessness), with a maximum possible score of 20. This parameter is assigned as "C" in the overall SCORAD calculation. The SCORAD is calculated as: A/5 + 7B/2 + C (Kunz et al, 1997).

#### 4.5.1.3. IGA

The IGA is an assessment scale used in clinical studies to determine severity of AD and clinical response to treatment based on a 5-point scale ranging from 0 (clear) to 4 (severe/very severe). The proportion of subjects who achieve an IGA 0 or 1 score is another key secondary endpoint which will be included in the primary analysis.

#### 4.5.1.4. NRS

Pruritus Numerical Rating Scale (NRS): Subjects will record once daily and respond to the following question, "On a scale of 0 - 10, with 0 being no itch and 10 being the worst itch

imaginable, how would you rate your worst degree of itch during the previous 24 hours?" Subject compliance on the pruritus NRS will be followed at each clinic visit.

#### 4.5.1.5. **DLQI**

The Dermatological Life Quality Index (DLQI) is a simple, subject-administered, 10-question, validated, quality-of-life questionnaire that covers 6 domains including symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. Response categories include "a little", "a lot" and "very much" with corresponding scores of 1, 2, and 3 respectively and "nor at all", "not relevant" responses score as "0". Totals range from 0 to 30 (less to more impairment) and a 5-point change from baseline is considered clinically relevant (Basra et al, 2008, Finlay et al, 1994).

#### 4.5.2. Pharmacokinetic, Pharmacodynamic and Biomarker Assessments

#### 4.5.2.1. Pharmacokinetic Assessments

Blood samples will be collected as per routine phlebotomy procedures and at time points specified in the Schedule of Events (Appendix 1). Briefly, blood samples (1 x 3.5 mL each) will be collected during the course of the study through indwelling cannula placed in forearm veins or alternatively, by a fresh clean venipuncture using a disposable sterilized syringe and a needle. The cannulae will be maintained patent as per local practice.

The minute of collection of each blood sample will be recorded. Actual time points will be used for PK calculations.

The details of sample collection, processing and storage are outlined in the laboratory manual. The sample will be shipped to the specified bioanalytical laboratory. Serum concentration of GBR 830 will be quantified using a validated Enzyme-linked immunosorbent assay (ELISA) method.

#### 4.5.2.2. Immunogenicity Assessments

Blood samples will be collected at appropriate time points defined in Appendix 1, to evaluate ADA to GBR 830, as per procedures similar to collection of PK samples. Antibodies of GBR 830 will be detected and confirmed using a validated ELISA method. The details of sample collection, processing and storage are outlined in the lab manual. The samples will be shipped to the specified bioanalytical lab.

#### 4.5.2.3. Biomarker Assessments

#### 4.5.2.3.1. Flow cytometry/ Leukocyte sub-population cell counts

Blood samples will be collected at appropriate time points defined in Appendix 1. The details of sample collection, processing and storage are outlined in the lab manual.

#### 4.5.2.3.2. Cytokine and Chemokines

Blood samples will be collected at appropriate time points defined in Appendix 1. The details of sample collection, processing and storage are outlined in the lab manual.

#### 4.5.2.3.3. Total IgE

Subjects with AD often have elevated IgE. Total IgE levels have been found to modestly correlate with AD severity and may be involved in the pathogenesis of the disease. Changes in total IgE reflects not only on AD, but atopy in general. Baseline IgE levels will be assessed for potential predictive value for treatment response. Post-treatment samples will be evaluated for effects of GBR 830 on total IgE. Detailed instructions for blood sample collection are outlined in the lab manual. Blood samples will be collected at appropriate time points defined in Appendix 1.

#### 4.5.2.3.4. Transepidermal Water Loss

Transepidermal Water Loss (TEWL) is a skin barrier function test that measures perspiration or water loss through the skin. This procedure involves the non-invasive application of a probe on the surface of the skin on the arm or leg. Affected and non-affected areas of skin will be tested. This procedure will only be performed at specified study centers. The detailed procedure for TEWL is provided in the Study Reference Manual.

#### 4.5.2.3.5. Immunohistochemistry (IHC)

Skin biopsy samples will be collected at appropriate time points defined in Appendix 1. Two punch biopsies (1 from lesion skin (LS) and 1 from non-lesion skin (NLS)) will be collected at baseline visit and one punch biopsy (from LS) at the subsequent time point. For LS, biopsy should be taken from a target lesion initially and always taken from the same lesion or location thereafter. Scar tissue from previous biopsies should be avoided. A 4.5 mm punch biopsy should be taken from the most involved chronic active erythematous, scaly lesions. For NLS, a 4.5 mm sample should be collected from the most normal appearing skin in a relative proximity to the LS biopsy site, at least 5 cm away from the lesion (at least 1 cm away, if 5 cm is not possible). Full details of sample collection, processing and storage are outlined in the lab manual.

#### 4.5.2.3.6. RT-PCR

Skin biopsy samples, as collected and mentioned previously will also be used for RT-PCR. The detailed methodology will be outlined in the lab manual.

### 4.5.2.3.7. Serum Soluable OX40 Ligand and Serum Soluable OX40

The PK samples will be used for the estimation of soluble OX40L and sOX40 in serum at the time points specified in the schedule of events in Appendix 1. The samples will be shipped to the specified bioanalytical lab. Serum concentrations of soluble OX40L and OX40 will be quantified using a qualified commercial ELISA kit.

#### 4.5.3. Safety Assessments

Safety assessments will consist of monitoring and recording all AEs and SAEs; regular monitoring of hematology, blood chemistry, and urinary laboratory values; periodic measurement of vital signs and ECGs; and performance of physical examinations as detailed in the Schedule of Events (Appendix 1). At the end of the study another clinical assessment consisting of a physical examination and all laboratory tests performed at the time of screening (except viral serology, and FSH) will be performed. Dosing will be based on evaluations performed by physicians/Investigator. Additional assessments can be integrated into the protocol further to investigator judgment.

#### 4.5.4. Schedule of Assessments

Study procedures and assessments are summarized across all study visits within the Schedule of Events (Appendix 1). The visit windows are mentioned below.

#### 4.5.4.1. Visit Identification (ID)

The visits are defined at the following study days:

- Visit ID 1 (V1) [Baseline visit]: Study day -30 to -1
- V2: Study day 1
- V3: Study day  $4 \pm 1$
- V4: Study day  $8 \pm 1$
- V5: Study day  $15 \pm 1$

- V6: Study day  $22 \pm 2$
- V7 (Dosing visit)\*: Study day  $29 \pm 1$
- V8: Study day  $32 \pm 1$
- V9: Study day  $36 \pm 1$
- V10: Study day  $43 \pm 1$
- V11: Study day  $50 \pm 2$
- V12: Study day  $57 \pm 2$
- V13: Study day  $71 \pm 2$
- V14: Study day  $85 \pm 2$

#### 4.5.4.2. Visit windows

The visit windows for assessments are defined as follows:

#### Window for collection of samples for GBR-830 PK analysis:

- V2 and V7:
  - Pre-dose: within 15 minutes before administration of each dose
  - Post-dose:
    - Immediately at the end of each infusion  $\pm$  10 mins;
    - 1.5 hrs  $\pm$  10 mins estimated from the start time of infusion
    - 2 hrs  $\pm$  10 mins estimated from the start time of infusion
    - 4 hrs  $\pm$  10 mins estimated from the start time of infusion
- V3 and V8: 72 hrs  $\pm$  24 hrs estimated from the start time of infusion
- V4 and V9: 168 hrs  $\pm$  24 hrs estimated from the start time of infusion
- V5 and V10: 336 hrs  $\pm$  24 hrs estimated from the start time of infusion
- V6 and V11: 504 hrs  $\pm$  48 hrs estimated from the start time of infusion
- V12, V13, V14: 1344 hrs (Day 57) ± 48 hrs, 1680 hrs (Day 71) ± 48 hrs, and 2016 hrs (Day 85) ± 48 hrs estimated from the start time of first infusion. Visits and assessments done in relation to the second infusion will be calculated from the actual day/start time of the second infusion. This applies to V8 to V11, inclusively. For V12,

<sup>\*</sup>If the second dosing visit is altered, then the time-points for visits V12, V13 and V14 will be calculated from the second infusion.

V13, and V14, the time points for assessment will be 672hr, 1008hr, and 1344hr, respectively, from the start time of the second infusion.

#### Window for vital signs:

- V2 and V7:
  - Pre-dose: within 30 minutes before administration of each dose
  - Post-dose:
    - Every half hour during infusion  $\pm$  10 mins;
    - 0.5 hrs  $\pm$  10 mins estimated from the end time of infusion
    - 1 hr  $\pm$  10 mins estimated from the end time of infusion
    - 2 hrs  $\pm$  10 mins estimated from the end time of infusion
    - 6 hrs  $\pm$  10 mins (in V2 only) estimated from the end time of infusion
    - 3 hrs  $\pm$  10 mins (in V7 only) estimated from the end time of infusion
- V3 and V8: 72 hrs  $\pm$  24 hrs estimated from the start time of infusion
- V4 and V9: 168 hrs  $\pm$  24 hrs estimated from the start time of infusion
- V5 and V10: 336 hrs  $\pm$  24 hrs estimated from the start time of infusion
- V6 and V11: 504 hrs  $\pm$  48 hrs estimated from the start time of infusion

V12, V13, V14: 1344 hrs (Day 57)  $\pm$  48 hrs, 1680 hrs (Day 71)  $\pm$  48 hrs, and 2016 hrs (Day 85)  $\pm$  48 hrs estimated from the start time of first infusion. Visits and assessments done in relation to the second infusion will be calculated from the actual day/start time of the second infusion. This applies to V8 to V11, inclusively. For V12, V13, and V14, the time points for assessment will be 672hr, 1008hr, and 1344hr, respectively, from the start time of the second infusion.

•

### **Window for ECG recording:**

- V2:
  - Pre-dose: before administration of each dose
  - Post-dose: 2 hrs  $\pm$  30 mins and 6 hrs  $\pm$  30 mins estimated from the end time of infusion
- V3 and V8: 72 hrs  $\pm$  24 hrs estimated from the start time of infusion
- V4 and V9: 168 hrs  $\pm$  24 hrs estimated from the start time of infusion
- V7:
  - Pre-dose: before administration of each dose

- Post-dose: 2 hrs  $\pm$  15 mins and 3 hrs  $\pm$  15 mins estimated from the end time of infusion

V12, V13, V14: 1344 hrs (Day 57)  $\pm$  48 hrs, 1680 hrs (Day 71)  $\pm$  48 hrs, and 2016 hrs (Day 85)  $\pm$  48 hrs estimated from the start time of first infusion. Visits and assessments done in relation to the second infusion will be calculated from the actual day/start time of the second infusion. This applies to V8 to V11, inclusively. For V12, V13, and V14, the time points for assessment will be 672hr, 1008hr, and 1344hr, respectively, from the start time of the second infusion.

#### For all other safety and pharmacodynamics/biomarker/immunogenicity assessments:

- V2: before administration of each dose
- V3 and V8: 72 hrs  $\pm$  24 hrs estimated from the start time of infusion
- V4 and V9: 168 hrs  $\pm$  24 hrs estimated from the start time of infusion
- V5 and V10: 336 hrs  $\pm$  24 hrs estimated from the start time of infusion
- V6 and V11: 504 hrs  $\pm$  48 hrs estimated from the start time of infusion
- V7: before administration of each dose

V12, V13, V14: 1344 hrs (Day 57)  $\pm$  48 hrs, 1680 hrs (Day 71)  $\pm$  48 hrs, and 2016 hrs (Day 85)  $\pm$  48 hrs estimated from the start time of first infusion. Visits and assessments done in relation to the second infusion will be calculated from the actual day/start time of the second infusion. This applies to V8 to V11, inclusively. For V12, V13, and V14, the time points for assessment will be 672hr, 1008hr, and 1344hr, respectively, from the start time of the second infusion.

In the event that assessments are planned for the same scheme time, the order of assessments should be arranged in such a way that PK blood sampling will be performed first, followed by ECG and vital signs, with blood sampling exactly on time. Samples collected outside the window period will be reported as protocol deviations and the actual time point of sample will be recorded.

### 5. PLANNED ANALYSES

# 5.1. Interim Analyses

There is no interim analysis planned.

# 5.2. Final Analyses

The final analysis top line results will be performed two weeks after the receipt of post-database lock data. All other analysis will be performed four weeks after the receipt of post-database lock data.

# 6. GENERAL CONSIDERATIONS FOR DATA ANALYSES AND HANDLING

# 6.1. General Summary Table and Individual Subject Data Listing Considerations

Summary tables and listings will include a "footer" providing explanatory notes that indicate:

- Date of data extraction (this is to link the output to the archived database that is locked to ensure the replication of the results.)
- Date of output generation.
- SAS program name, including the path that generates the output.
- Other output specific details such as abbreviation and acronym definitions, relevant methodological detail.

Tables will include reference(s) to the subject data listing(s) that supports the summary data.

The tables will be organized with respect to treatment group (GBR 830 then placebo) and a column will be included to summarize all treated subjects. Row entries in tables will only appear if data exists for at least one subject (e.g., a row with all zeros will not appear). The exception to this rule applies to tables that summarize the study termination status of subjects (e.g., reasons for not completing the study). In this case, zeros will appear for study termination reasons that no subject satisfied. The summary tables clearly indicate the number of subjects to which the data apply and unknown or not performed are distinguished from missing data.

Summary tables for medications and medical conditions are coded according to the WHO DDE September 2015 dictionary. Adverse event preferred terms and body/organ systems are coded using MedDRA 19.0 March 2016 dictionary. The MedDRA dictionary will also be used in the coding of signs and symptoms, medical history, physical examination abnormalities, and clinical diagnoses.

Supportive subject data listings will be sorted and presented by treatment group (group). Listings also include subject number, visit number, visit date, and days relative to the initiation of double-blind treatment.

No imputations are imposed for missing clinical data apart from for the primary and secondary endpoints analysis. Imputed or derived data will be flagged in the subject listings. Imputed data are not incorporated into any raw or primary datasets. These data are retained in derived analysis datasets.

# 6.2. General Post Text Summary Table and Individual Subject Data Listing Format Considerations

The tables and listings will be numbered using a decimal system to reflect main levels of unique tables and listings and sub-levels of replicate tables and listings with two digits per level (e.g., Table XX.YY.ZZ).

The first level number will be consistent with the corresponding CSR appendix in which the tables or listings will appear. For example, the post text tables usually occupy Appendix 14 and the individual subject data listings are put in Appendix 16. All post text tables will have a main number level 14 and listings 16. The subject accounting and disposition table are usually first in the first section of the report therefore will be numbered Table 14.1. The supportive subject data listing would be Listing 16.1.

The title will be complete, accurate, and concise. The last line of the title will provide the analysis group being summarized (e.g., Full Analysis Set, Safety Analysis Set, Biological Activity Set or Pharmacokinetic Analysis Set). If possible, the units of measurement for data contained in the table can appear in parentheses to conserve space in the body of the table. For example, the summary of vital signs title could read "Summary of Sitting and Standing Blood Pressure (mmHg) and Heart Rate (bpm)." Whether in the title or body of a table or listing, units must always be specified for all appropriate data.

If possible, variables being summarized and statistics reported should appear in the left most column of a table. The next columns for treatment groups should report the data from left to right for GBR 830, placebo and (optional) overall subjects, respectively.

In general, the listings will be sorted and presented by treatment assignment, and subject number. From left to right, the treatment assignment, subject number, visit number, visit date, and relative day should appear. All tables and listings will have explanatory notes that give, data extraction date, output generation date, and complete program name and path where it is stored. The definition of all derived variables and decodes for coded data will appear in the notes. Due to space limitations, tables and listings may require a page of notes as a one-time preface to the output.

# **6.3.** Data Management

Data from the study will be managed by Glenmark Pharmaceutics Ltd or their representative.

All data will be recorded on Electronic Case Report Forms (eCRFs). The Investigator will allow representatives of the Sponsor, regulatory agencies, and their designees to inspect all study documents (including, but not limited to, consent forms, investigational product accountability forms, Institutional Review Board [IRB]/Independent Ethics Committee [IEC] approvals) and pertinent hospital or clinical records for confirmation of data throughout and after completion of the study. Monitoring visits will be conducted as needed during the course of the study. A complete review of source documentation of key efficacy and safety data will be conducted at each monitoring visit for verification that all information recorded in the CRF accurately reflects the data recorded in the subject's source documents.

All data verification, using hospital or clinic records, will be performed respecting subject confidentiality and will be carried out in accordance with Standard Operating Procedures (SOPs). An electronic copy of the study eCRF will be provided to the investigational site upon final query resolution and Database closure.

All subject data generated during the study will be recorded and transcribed in the eCRF. The Principal Investigator must approve the eCRF to confirm eligibility. The final authorization of the CRF data is the Investigator Signature form. This form must be approved by the Principal Investigator to signify that he/she has reviewed the eCRF, including all laboratory and safety assessments, and that all of the data there is complete and accurate.

The data will be reviewed to ensure that the forms were completed properly and that all data has the correct subject identification number throughout.

Derived datasets are created using (SAS®) software. Data analyses and summary tables are generated using SAS version 9.4 or above.

#### **6.4.** Data Presentation Conventions

Continuous variables (e.g. age) will be summarized using descriptive statistics (the number of subjects with available data, the mean, standard deviation (SD), median and minimum and maximum). Categorical variables (e.g. race) will be summarized using counts and percentages. Percentages are calculated using the total subjects per treatment group.

The following conventions are applied to all data presentations and summaries.

For continuous variables, all mean and median values are formatted to one more decimal place than the measured value. Standard deviation values are formatted to two more decimal places than the measured value. Minimum and maximum values are presented with the same number of decimal places as the measured value.

For categorical variables, the number and percentage of responses are presented in the form "XX (XXX)" where the percentage is in the parentheses.

Date variables are formatted as DDMMMYYYY for presentation. Time is formatted in military time as HH:MM for presentation.

Wherever possible, data will be decimal aligned.

P-values will be presented to 3 decimal places. If the p-value is less than 0.001 then it will be presented as <0.001. If the rounded result is a value of 1.000, it will be displayed as >0.999.

Unless otherwise stated, any statistical tests performed will use 2-sided tests at the 5% significance level.

All tables and listings will use Times New Roman font of size 9. Page layout will be landscape and page size A4 unless otherwise specified in the shells.

The table and listing shells and table of contents as part of this SAP provide the expected layout and titles of the tables, listings and figures. Any changes to format, layout, titles, numbering, or any other minor deviation will not necessitate a revision to the SAP nor will it be considered a

deviation from planned analyses. Only true differences in the analysis methods or data handling will necessitate such documentation. The appropriate listings supporting the tables will be included and are not specified in the individual sections throughout the document.

### 6.5. Analysis Populations

Prior to hard database lock, a final blinded data review meeting to verify the data that will be used for analysis set classification. The Pharmacokinetic Analysis Set will be assessed and finalized once data has been unblinded post database lock.

#### 6.5.1. Screen Failures

Subjects who give informed written consent but are not dispensed study treatment are considered screen failures. No attempt will be made to further characterize the reason for screen failures (e.g., lost-to-follow-up, did not meet entry criteria, administrative) in summary tables due to the paucity of information usually gathered however the verbatim reason for screen failure will be included in the supportive listing.

#### 6.5.2. Full Analysis Set (FAS) Population

The Full Analysis Set (FAS) will consist of all subjects who are randomized and have received at least one partial or full dose of study treatment. FAS population will be used for the analysis of the efficacy data not obtained from skin biopsy. Subjects will be analyzed according to the treatment by which they were randomized to.

### 6.5.3. Biological Activity Set (BAS) Population

The Biological Activity Set (BAS) will consist of all FAS subjects who have at least one post-baseline skin biopsy (Visit 7, Visit 13), and received two doses of study drug. The primary analyses on biomarkers of disease activity obtained from biopsy will be based on the BAS. Subjects will be analyzed according to the treatment by which they were randomized to.

#### 6.5.4. Safety Analysis Set (SAF) Population

The Safety Analysis Set (SAF) consists of all subjects who took at least one full or partial dose of study treatment and will be used in the assessment and reporting of safety data. Subjects will be analyzed according to the treatment which they received rather than the treatment which they were randomized to. If a subject receives both treatments over the course of the study, they will be assigned to the active drug.

#### 6.5.5. Pharmacokinetic Analysis Set (PKAS) Population

The Pharmacokinetic Analysis Set (PKAS) consists of the subset of the Safety Analysis Set population for which sufficient serum concentration data is available to:

- 1. facilitate derivation of at least one PK parameter, and
- 2. the time (HH:MM) of dosing on the day of sampling is known

for at least one of the dosing visits. Additional subjects may be excluded from the PKAS at the discretion of the pharmacokineticist. The PKAS will include only subjects treated with GBR830. The exclusion of subjects or time-points from the PKAS are defined as:

- Subjects will be excluded from the analysis if the pre-dose concentration level before  $1^{st}$  dosing event is greater than 5% of the individual subject  $C_{max}$  after  $1^{st}$  dose.
- Subjects will be excluded if all of their post-dose values are less than lower limit of concentration.
- Subjects will be excluded if there is a major protocol deviation likely to affect the validity of the concentration levels.

#### 6.6. Baseline Definition

#### 6.7. Derived and Transformed Data

#### 6.7.1. Baseline Age

Subject's age in years will be calculated based on date of informed consent date using the following formula:

Age (years) = FLOOR((date of informed consent - date of birth)/365.25) where FLOOR() function returns the integer part of the result.

#### 6.7.2. Age at AD diagnosis

Subject's age in years at AD diagnosis will be calculated based on date of AD diagnosis using the following formula:

Age at AD diagnosis (years) = FLOOR((date of AD diagnosis - date of birth)/365.25)

Where FLOOR() function returns the integer part of the result.

### **6.7.3. Study Day**

If the date of interest occurs on or after the first infusion/randomization date then study day will be calculated as (date of interest – date of first infusion/randomization) + 1 day. If the date of interest occurs prior to the first infusion/randomization date then study day will be calculated as (date of interest – date of first infusion/randomization). There is no study day 0.

### 6.7.4. Change from Baseline

Baseline is defined as study day 1 unless stated otherwise.

Change from baseline is calculated as (post-baseline result – baseline result).

Percent change from baseline is calculated as [(change from baseline/baseline result) x 100].

If either the baseline or the post-baseline result is missing, the change from baseline and percentage change from baseline is set to missing as well unless imputation rules are applied for efficacy endpoints.

#### 6.7.5. Visit 12 and Visit 14 LOCF Visits

The Visit 12 and 14 LOCF derived visits are defined on a Last Observation Carried Forward basis as the last measurement available for each subject up to or on Visit 12 and 14. These visits will be used for the analysis of secondary endpoints (EASI, IGA, SCORAD, DLQI, TEWL).

For subjects who discontinue the study early and have completed the Visit 14/EOS assessment their Visit 12 and 14 LOCF will be derived using the re-mapped visit specified in 6.7.6

#### 6.7.6. End of Study Visit

Unless otherwise specified, the end of study visit will include those subjects who complete Visit 14 or who complete the early withdrawal visit. It will be abbreviated to Visit 14/EOS.

For the analysis of secondary efficacy variables (EASI, IGA, SCORAD, DLQI, TEWL), for patients who withdraw prematurely from the study and complete the Early Termination Visit, their Visit 14/EOS visit will be re-categorized as the visit immediately following their last scheduled visit.

#### 6.7.7. Multiple Assessments

Where multiple assessments occur within the same visit, the visit closest to the scheduled visit day described in the protocol will be used. If the values are equidistant to the scheduled visit day, the mean of these values is used for the summaries over time (by visit) in the case of continuous data, and the maximum of these values in the case of ordered categorical data. If the data is categorical, e.g. normal/abnormal not clinically significant/abnormal clinically significant then the assessment with the worst case scenario will be selected.

#### 6.7.8. Missing Efficacy Endpoints

Data will be assumed to be missing at random (MAR). Subjects that dropout are assumed will behave similarly to other subjects in the same treatment group, and with similar covariate values, had they not dropped out.

Missing data will be imputed where necessary and details can be found in Section 8.

#### 6.7.9. Missing Start and Stop Dates for Prior and Concomitant Medication

Incomplete concomitant medication start and/or stop dates will be imputed as follows:

- If either the start of medication date is completely missing or the month and/or year of the start date is missing, the start date will be set to the treatment start date. If imputed start date is after the stop date, then change the imputed start date to stop date minus 1 day.
- If only the day is missing, the day will be set to the first day of the month except if the start month is the same as the treatment start month. If the latter is true, the start day will be set to the treatment start day. If imputed start date is after the stop date, then change the imputed start date to stop date minus 1 day.
- No imputations will be applied to the stop date.

Imputed dates will be flagged in the subject data listings.

#### 6.7.10. Missing Start and Stop Dates for Adverse Events

Completely missing or partially missing AE start dates will be imputed as follows:

- If the AE start date is completely missing or the month and/or year are missing, the AE start date will be set to the treatment start date. If imputed start date is after the stop date, then change the imputed start date to stop date minus 1 day.
- If only the day is missing, and month and year are the same as treatment start date then start date will be set to the treatment start date. Otherwise the first day of the month will be assumed. If imputed start date is after the stop date, then change the imputed start date to stop date minus 1 day.
- No imputations will be applied to the stop date.

Imputed dates will be flagged in the subject data listings.

#### 7. STUDY POPULATION

The study population will be analyzed using the Full Analysis Set unless otherwise specified.

### 7.1. Subjects Disposition

Subject disposition will be summarized using counts and percentages. Percentages will be based on the number of randomized subjects. All subjects screened and randomized will be summarized and listed.

The count and percentage of subjects included in each analysis set (as described in Section 6.5) will be presented. Percentages will be based on the number of randomized subjects.

The count and percentage of subjects who completed or discontinued from the clinical study will be summarized in a table and listed by treatment arm and overall. Percentages will be based on the number of randomized subjects. This will include a summary of the reasons for early termination or withdrawal from the study.

The following categories for early termination and withdrawal from the study will be presented:

- Withdrawal of consent
- Adverse event
- Investigator's discretion
- Non compliance with study procedures/protocol deviation
- Pregnancy
- Subjects requiring rescue medications or interventions/treatment with another therapeutic agent
- Disease progression/exacerbation
- Subjects randomized in the study who withdrawal their consent for the first post-baseline skin biopsies
- Lost to follow-up
- Death
- Other

For subjects who are non-completers a listing will be provided containing further details on the reasons for early termination/withdrawal and the Study Day of early termination/withdrawal see section 6.7.3 for Study Day calculation.

Descriptive statistics will be provided for the subject's time on study and will be analyzed using the Full Analysis Set. Time on study (days) will be calculated as:

End of Study Date – Randomization Date + 1 day

A subject listing will be provided containing, for each subject, the date of first and last use of study treatment and the date of withdrawal from study.

#### 7.2. Screen Failures

Screen failures are subjects who are screened but not randomized. The number of subjects who are screening failures will be summarized.

A subject listing will be provided on all screen failures including the reason for screening failure. Screen failure subjects will neither contribute to other data presentations, nor participate in formal analyses.

#### 7.3. Protocol Deviations

A subject listing will be provided containing detail of the protocol deviation as captured in the CRF, including the protocol deviation number, date reported, deviation coding, protocol deviation reportable to ethics (yes or no) and also any further detail; for example a description of the actions taken (if any).

The protocol deviation coded terms are defined as follows:

- Subject non-compliance with study procedures
- Missed dose(s)
- Extra dose(s)
- Fasting period not respected
- Randomization error
- Study visit not done
- Visit performed out of window
- Procedure(s) done but not required by the protocol
- Prohibited Medication
- Study procedure(s) not done
- Time window / order of events for study procedures not respected
- Washout period not respected
- Other

### 7.4. Demographic and Baseline Characteristics

Descriptive statistics will be used to summarize baseline demographics and characteristics separately for subjects in each analysis set (FAS, BAS and PKAS).

Descriptive statistics will be provided for the following continuous variables:

- Age (years) at entry into the study
- Age (years) at AD diagnosis
- Weight (kg)
- Height (cm)
- BMI (kg/m²) [This will be calculated in the clinical database from baseline height and weight.]
- Body Surface Area (m<sup>2</sup>) [This will be calculated using BSA = 0.007184 x weight (kg)<sup>0.425</sup> x height(cm)<sup>0.725</sup> (Du Bois D, Du Bois EF, 1916).]

The following categorical demographics will be summarized using count and percentages of subjects by treatment group and overall. Percentages will be based on the appropriate analysis set:

- Age group at study entry
  - < 65 years
  - >= 65 years
- Sex
  - Male
  - Female
- Ethnicity
  - Hispanic or Latino
  - Not Hispanic or Latino
- Race
  - American Indian or Alaska Native
  - Asian
  - Black
  - Native Hawaiian or Other Pacific Islander
  - White
  - Other

- Country
  - USA
  - Canada
- Child bearing potential (female only)
  - Yes
  - No
    - Post menopausal
    - Permanently sterilized
    - Duration of non child bearing potential ( $\leq 1$  year, > 1 year)

Child bearing potential will be summarized for females only and percentages will be calculated using female subjects only. All demographics will be presented in a subject listing.

# 7.5. Listing of Subject Inclusion and Exclusion Criteria

A listing will be provided for all screened subjects which states for each subject whether the inclusion and exclusion criteria were met and, if not met, the applicable failed inclusion/exclusion criteria reason as captured in the CRF. The enrollment status (randomized or screen failure) and if randomized, the treatment allocated will also be listed.

# 7.6. Medical History and Medical Conditions Present at Entry

Medical history at baseline will be summarized in three separate tables for the Full Analysis Set by treatment group and overall:

- AD history
- Medical/surgical history
- Smoking, alcohol and drug abuse history

For AD history the following continuous variables will be summarized using descriptive statistics:

• Time since AD diagnosis (years)

The following categorical variables will be summarized using counts and percentages. Percentages will be based on the analysis set:

• Time since AD diagnosis category

- < 2 years
- -2-5 years
- >= 5 years
- Type of AD: Intrinsic; Extrinsic
- Any history of allergy: Yes; No
- Was patch test performed: Yes; No
- Any other concomitant atopic illness? Yes; No
  - Type of Concomitant atopic illness: Asthma; Allergic rhinitis, Skin conditions;
    Other
- Was Skin biopsy performed in past? Yes; No
  - Result of skin biopsy: Eosinophilic; Non-eosinophilic; Other
- Any treatment administered for AD or associated conditions? Yes; No

A subject listing will also be provided for AD history data.

Medical/surgical history will be considered as they are captured in the CRF.

Each preferred term within a body system will be summarized using counts and percentage. Percentages will be based on the analysis set. Subjects will be counted only once at the system organ class level and will be counted once for each applicable preferred term. Data will be sorted by descending frequency of system organ class, then descending frequency of preferred term within organ class for the overall group. The following body systems will be considered:

- HEENT
- Cardiovascular System
- Respiratory System
- Musculoskeletal System
- Dermatological System
- Skin and its appendages
- Lymphatic System
- Gastrointestinal System
- Genitourinary System
- Nervous System
- Endocrine System
- Immunological System

- Allergic Conditions
- Other

A subject listing of all medical/surgical history data will be provided including body system, preferred term, start and end dates, ongoing status and severity grade (mild; moderate; severe; not known).

Smoking, alcohol and drug abuse history will be summarized.

The following continuous variables will be summarized using descriptive statistics, for current users only (subjects with zero will be considered missing):

- Alcohol consumption, ml/week
- Number of cigarettes per day

The following categorical variables will be summarized using counts and percentages. Percentages will be based on the analysis set:

- Former/current alcohol user: Former; Current; N/A
  - History of alcohol abuse: Yes; No
- Former/current drug user: Former; Current; N/A
  - Does the subject meet DSM-V criteria for addiction or abuse: Yes; No
- Former/current smoker: Former; Current; N/A
- Former/current smokeless tobacco user: Former; Current; N/A

Missing data will also be summarized where appropriate.

A subject listing of smoking, alcohol and drug abuse history will also be provided. In addition to the above, it will include specified forms of drug and tobacco as well as stop dates for former users.

# 7.7. Prior Medication History

Medications with a start date before the date of the first dose of study treatment will be classified as a prior medication.

All prior medications will be coded by anatomic-therapeutic-class (ATC) coding system, WHO DDE (September 2015) and the data will be summarized by each ATC level and preferred term (generic name).

The Full Analysis Set will be used.

#### 7.7.1. Diagnosis Related Medication History

Medications administered for AD and related conditions will be summarized using counts and percentages by preferred term for each treatment group and overall. Data will be sorted by descending frequency within the overall group.

A subject listing will be provided including medication start and stop dates, whether the medication is ongoing, dose, frequency of administration, route of administration, trade name (if known) and indication for use.

### 7.7.2. Non-Diagnosis Related Medication History

Those medications which are not considered in Section 7.7.1 will be summarized using counts and percentages by preferred term for each treatment group and overall. Data will be sorted by descending frequency within the overall group.

A subject listing will be provided including medication start and stop dates, whether the medication is ongoing, dose, frequency of administration, route of administration, trade name (if known) and indication for use.

## 7.8. Baseline Physical Examination

The results of the baseline physical examination will be listed by treatment group and subject. The following body systems will be listed:

- General appearance
- Neck
- HEENT
- Cardiovascular system
- Respiratory system
- Musculoskeletal system
- Skin
- Gastrointestinal System

- Genitourinary System
- Neurological System
- Other

Each body system will be categorized into one of the following: normal; abnormal, not clinically significant; abnormal, clinically significant.

The count and percentage of subjects whose physical examination is performed/not performed will be summarized.

### 7.9. Baseline Vital Signs

Baseline vital signs are defined as the vital signs measured at the visit immediately prior to the first dose of study drug.

Descriptive statistics will be used to summarize baseline vital signs by treatment group, for Safety Analysis Set subjects.

Descriptive statistics will be provided for the following vital signs:

- Systolic blood pressure (mmHg)\*
- Diastolic blood pressure (mmHg)\*
- Body temperature (°C)
- Pulse rate (beats per minute [bpm])\*
- Weight (kg)
- BMI  $(kg/m^2)$
- Body Surface Area (m<sup>2</sup>)

Blood pressure, body temperature and pulse rate will be categorized as normal; abnormal, not clinically significant; abnormal, clinically significant and the count and percentage of subjects by treatment group will be summarized.

All baseline vital signs data will be displayed in subject listings and clinically significant findings will be flagged.

<sup>\*</sup>Blood pressure and pulse rate are tested in supine position.

#### 7.10. Baseline Laboratory Data

Baseline laboratory results are defined as the last assessment prior to the first dose of study treatment regardless of whether it was scheduled, retest or unscheduled. Since laboratory retests can occur for individual parameters, it is necessary to define the baseline individually for each parameter.

All laboratory tables will be analyzed using the Safety Analysis Set.

Summary tables will be presented for each category of data (Haematology, Serum Biochemistry, Liver Function Tests, Renal Function Tests, Lipid Profile, Urinalysis, Serology, Other [for full list of laboratory parameters see Section 9.4]) by treatment group and overall. Descriptive statistics will be used to summarize the data:

- Quantitative laboratory test result will include mean, median, standard deviation, minimum and maximum.
- Qualitative tests (e.g. some urinalysis assessments and serum Beta-HCG pregnancy test) will be categorized accordingly.

The results of the serum pregnancy test will be reported as positive or negative for the female subjects and not applicable (NA) for male subjects in the summary of hematology results. The set of laboratory parameters included in each table will correspond to those requested in the study protocol. Units will be as found in the data.

All baseline laboratory data will be listed and will include the type of visit (e.g. scheduled test, retest, or unscheduled), age, sex, laboratory test, test units, laboratory test result, and the laboratory standard normal ranges adjusted as appropriate for age and sex, if available.

#### 7.11. Baseline ECG

Baseline ECG results are defined as the ECG results measured at the visit immediately prior to the first dose of study drug.

Descriptive statistics will be used to summarize baseline ECG results by treatment group and overall for Safety Analysis Set subjects.

Descriptive statistics will be provided for the following ECG results:

- Heart Rate (bpm)
- PR Interval (ms)
- RR Interval (ms)
- QRS Interval (ms)

- QT Interval (ms)
- QTcF Interval (ms)

The result of the ECG assessment will be categorized as normal; abnormal, not clinically significant; abnormal, clinically significant and the count and percentage of subjects by treatment group and overall will be summarized. Percentages will be based on the analysis set.

All ECG data will be displayed in a subject listing and clinically significant findings will be flagged. Triplicate ECG performed at baseline will be listed only.

#### 7.12. Baseline Clinical Scores

Baseline clinical scores are defined as the clinical scores recorded at the visit immediately prior to the first dose of study drug. Descriptive statistics will be used to summarize baseline clinical scores by treatment group and overall.

Descriptive statistics will be provided for the following clinical scores:

- EASI
- SCORAD
- Pruritus NRS
- DLQI

The result of the IGA assessment will be categorized as not done; clear; almost clear; mild; moderate; severe/very severe and the count and percentage of subjects by treatment group and overall will be summarized. Percentages will be based on the Full Analysis Set.

# 7.13. Baseline Skin Biopsy (Non-lesion only)

The non-lesion samples will be collected at baseline only. The mRNA expressions and pathologic epidermal phenotype markers (referred to here after as biomarkers) will be log transformed and summarized for the Biological Activity Set. Descriptive statistics will be used to summarize the biomarkers by treatment group and overall.

19 biomarkers from RT-PCR Panels (normalized to hARP) and the Immunohistochemistry (IHC) and will be summarized. A selection of these markers is found in Section 8.6.1

#### 8. EFFICACY

#### 8.1. General Considerations

Categorical data will be summarized using counts and percentages.

Continuous data will be summarized using counts, mean, s.d., s.e., median, minimum, maximum and 25<sup>th</sup> and 75<sup>th</sup> percentile where appropriate.

Formal statistical tests will be two-sided using a significance level of 5%, unless stated otherwise.

The Full Analysis Set will be used for the analysis of efficacy data, except the biopsy data which will be analyzed using the Biological Activity Set.

# 8.2. Testing Statistical Assumptions Including Comparability at Baseline

There will be no tests performed on the baseline data.

# 8.3. Statement of the Null and Alternate Hypotheses

The primary objective of this study is safety therefore there are no null or alternative hypotheses stated in the protocol.

# 8.4. Subgroup Analyses

There are no planned subgroup analyses.

## **8.5.** Multiple Comparisons and Multiplicity

There will be no adjustment for multiplicity in this study.

### **8.6.** Analysis of the Primary Efficacy Endpoint

#### 8.6.1. Primary Efficacy Analysis

The primary analysis will examine the effect of GBR 830 in adult subjects with AD in terms of change from baseline in selected biomarkers obtained from skin biopsies. Only the lesion samples will be analyzed for the primary efficacy analysis.

19 mRNA biomarkers (K16, IL13, IL17A, IL22, INFg, IL-23p19, IL-23p40, OX40L, MMP12, S100A12, IL-5, CCL17, CCL18, CCL11, CCL26, S100A9, CXCL10, FOXP3, TSLPR) from the RT-PCR Panels will be assessed for the primary endpoint analysis.

The 19 biomarkers will be normalized to housekeeping gene hARP and log transformed for analysis. Measurements under the limit of detections will be imputed as 20% of the minimum value observed for that biomarker normalized to hARP prior to the log transformation.

For each of the mRNA normalized to hARP, a mixed model repeated measure (MMRM) approach of the repeated measures data will be implemented. The outcome for each MMRM will be the changes from baseline in the log transformed biomarkers.

The model will include the following:

- Categorical fixed effects: planned study treatment, planned visit
- Continuous fixed effects: baseline (log transformed) biomarker
- Random effects: planned visits within subjects

An unstructured covariance structure will be used to model the within-subject variability. If this analysis fails to converge, no other structures will be fitted and only summary statistics will be provided for that biomarker.

From the model the geometric mean change (with 95% CIs) from baseline at Visit 13 will be obtained for each treatment group. The overall least squares mean treatment difference (with 95% CIs) and the p-value between GBR 830 and placebo will also be presented.

As there are no adjustments for multiplicity, no inferences will be drawn from the p-values of the mixed model.

The mRNA normalized to hARP will be summarized at baseline, each study visit (Visit 7, Visit 13) and for change from baseline by treatment group using descriptive statistics. The geometric mean (with 95% CI) and CV (%) will also be reported. If non-lesion samples are available these will also be summarized

Box plots by treatment will also be produced for each of the biomarkers.

Pathologic epidermal phenotype measures for H&E thickness, K16.IHC and Histological response will be summarized by visits at both baseline and post-baseline. In addition, CD3, Ki67, FcEpsilonRI, OX40, OX40L, MBP will also be summarized by visit for epidermis and dermis measures. If non-lesion samples are available these will also be summarized

#### 8.6.2. Sensitivity Analyses of the Primary Efficacy Endpoint

Not required.

### 8.7. Analysis of the Secondary Endpoints

#### 8.7.1. Proportion of subjects who achieve an IGA score of 0 or 1 at each study visit

IGA scores will be categorized as follows:

- 0 (clear) or 1 (almost clear)
- 2+ (mild, moderate, severe/very severe)

The proportion of subjects, who achieved the IGA scores above at each study visit (Visit 3 to Visit 14) and the Visit 12/14 LOCF visits, will be summarized by treatment group and overall.

For subjects who use prohibited medication, any IGA score on or after the date of first use of prohibited medication will be set to missing.

A Cochran-Mantel-Haenszel (CMH) test will be performed to compare the IGA categories above for GBR 830 treatment and placebo at both the Visit 12 LOCF and Visit 14 LOCF visits. The CMH test will be stratified by categorical baseline IGA score (less or equal to 3, greater or equal to 4).

# 8.7.2. Proportion of subjects who achieve an EASI 50 and 75 responses at each study visit

The proportion of subjects who achieve an EASI 50 (and 75) response each study visit (Visit 3 to Visit 14), the Visit 12/14 LOCF visits, will be summarized by treatment group and overall.

- An EASI 50 responder is defined as a subject with at least a 50% reduction in EASI score compared to baseline.
- An EASI 75 responder is defined as a subject with at least a 75% reduction in EASI score compared to baseline.

For subjects who use prohibited medication, any EASI score on or after the date of first use of prohibited medication will be set to missing.

A line plot will be produced of the EASI 50 rate over time by treatment group. Mean and SE  $(\pm 1)$  will be presented.

#### 8.7.3. Analysis of covariance EASI scores

For the Visit 12 LOCF change from baseline will be analyzed using an analysis of covariance (ANCOVA) model with treatment and baseline EASI score as linear covariates.

The LS-means at Visit 12 LOCF for each treatment group will be provided as well as the treatment difference at Visit 12 LOCF, with the corresponding standard errors, associated 95% confidence intervals and p-value. If the assumptions of the ANCOVA are not met (e.g. not meeting any of the following: normality, homogeneity of variance, random independent samples or a linear relationship between the dependent variable and the covariates) then a non-parametric rank-based ANCOVA method will be used instead, where the ranked values are the change from baseline in EASI scores.

# 8.7.4. Percent improvement in clinical scores EASI, SCORAD, IGA, Pruritus NRS and DLOI from baseline to each visit

The percent change from baseline in the following clinical scores will be summarized by each treatment group at each study visit (Visit 3 to Visit 14), and for the Visit 12/14 LOCF visits

- EASI
- SCORAD
- IGA
- Pruritus NRS
- DLQI

For subjects who use prohibited medication, any clinical score on or after the date of first use of prohibited medication will be set to missing.

Line plots will be produced of the percentage change over time for Pruritus NRS and EASI score by treatment group. Mean and SE  $(\pm 1)$  will be presented.

# 8.7.5. Changes from baseline AD activity as determined by changes in Transepidermal water loss (TEWL)

Lesion and non-lesion areas average transepidermal water loss (TEWL) reading values and change from baseline will be summarized separately at each planned study visit and the Visit 12/14 LOCF visits, as well as the change from baseline at each time point by treatment group and overall using descriptive statistics.

For subjects who use prohibited medication, the TEWL average reading on or after the date of first use of prohibited medication will be set to missing.

#### 8.7.6. Anti-drug antibodies (ADA) to GBR 830 to evaluate immunogenicity.

Anti-drug antibodies (ADA) will be summarized using counts and percentages by treatment group at each planned study visit and overall (including the overall number of subjects and percentage of subjects with positive and negative ADA at any post baseline visit), for the following categories:

- Positive
- Negative
- Not done

The individual subject ADA results will be listed.

The impact of ADA on the PK will be evaluated graphically by scatter plot with individual subject concentration levels vs ADA status, stratified by treatment.

#### 8.8. Analysis of the Exploratory Endpoints

All exploratory endpoints will be summarized using descriptive statistics as well as the geometric mean (with 95% CI) and CV (%).

The endpoints below will be analyzed as described below, however these analyses, and biomarkers, could be subject to change when the final exploratory biomarkers are known.

#### 8.8.1. Change from Baseline in Cytokines in serum

The exploratory cytokines analysis will be determined after database lock of the study, therefore no statistical analysis of those parameters will be included in this SAP.

# 8.8.2. Change from Baseline in Leukocyte sub-population cell counts (Total T, T helper, Cytotoxic T, T<sub>regs</sub>, Memory T cells)

Descriptive statistics will be summarized for each Leukocyte sub-population cell counts (Total T, T helper, Cytotoxic T,  $T_{regs}$ , Memory T cells) by treatment group, separately for baseline and each visit (Visit 7, Visit 13).

The actual and percentage change from baseline will also summarized by treatment group.

# 8.8.3. Change from Baseline in Cellular infiltrates (T-cells, dendritic cells) as assessed by CD3, FcEpsilon RI, OX40L, OX40 and MBP

Descriptive statistics will be summarized for Cellular infiltrates (T-cells, Dendritic cells) as assessed by CD3, FcEpsilon RI, OX40L, OX40 and MBP by treatment group and overall for baseline and each visit (Visit 7, Visit 13).

The actual and percentage change from baseline will also summarized by treatment group.

# 8.8.4. Change from Baseline in Serum total Immunoglobulin E (IgE), serum soluble OX40 (sOX40), serum soluble OX40 ligand (sOX40L) and circulating eosinophil counts.

Descriptive statistics will be summarized for total IgE, serum soluble OX40 (sOX40), serum soluble OX40 ligand (sOX40L), and circulating eosinophil counts by treatment group and overall for baseline and each visit (Visit 7, Visit 13).

The actual and percentage change from baseline will also summarized by treatment group.

# 8.9. Summary of Reasons for Efficacy Non-Evaluability/Exclusion from Efficacy Analyses

If subjects use prohibited medication, and the deviation is classified as a major deviation by the medical monitor at the blinded review meeting, any clinical endpoint data (i.e. IGA, EASI, SCORAD, Pruritus NRS, DLQI, TEWL) collected on or after the recorded deviation will be considered as non-evaluable and set to missing.

The date of prohibited medications which will be used is the earliest reported date of a major deviation for each subject from the protocol deviations page of the CRF. Note that this date may be on or after the actual start date of the prohibited medication(s).

Descriptive statistics will be used to summarize the major deviations by study visit on which the first major deviation of prohibited medication occurs. Counts and percentages will be used to summarize the visits which have been excluded due to use of prohibited medication.

The assessment of major or minor deviation for prohibited medications be provided as a SAS dataset and incorporated into the analysis.

#### 9. SAFETY AND TOLERABILITY

All safety analysis will be based on the Safety Analysis Set.

# 9.1. Treatment Emergent Adverse Event Preferred Term and Body/Organ System Summary Tables

All treatment emergent adverse events (TEAEs) occurring in the study, in terms of nature, onset, duration, severity, relationship and outcome of adverse events (AEs) and serious adverse events (SAEs), in adult subjects with moderate-to-severe AD will be assessed.

Adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) version 19.0 (March 2016).

Rules for missing AE dates are found in Section 6.7.10.

The analysis described below will be summarized for events considered to be treatment emergent. For an event to be treatment emergent it must have an onset date or worsening on or after the first dose of study drug. All AEs will be listed.

#### 9.1.1. Summaries of Adverse Event Incidence Rates for All Subjects

The count and percentage of subjects with each of the following will be summarised by system organ class, preferred term and treatment group:

- AEs
- SAEs
- AEs leading to permanent withdrawal of study treatment
- AEs leading to withdrawal from study
- AEs related to investigational product
- AEs leading to death

Subjects will be counted only once at the system organ class level and once for each applicable preferred term; regardless of how many of those events they have had. Data will be sorted by descending frequency of system organ class, then descending frequency of preferred term within each system organ class for the GBR 830 group.

The count and percentage of AEs by severity will also be summarized. If severity is missing, AEs will be considered to be severe. If there are multiple severities for the same preferred term, the most severe will be used

All AEs will be displayed in a two-part subject listing sorted by treatment group and including the following information:

#### • Part 1:

- AE onset date/time and relative study day
- AE end date/ time and relative study day
- Duration of AE (days) [derived as: AE end date AE start date +1 day]
- Treatment emergent flag
- SAE (Yes; No)
- MedDRA body system
- MedDRA preferred term
- Investigator included term (verbatim)
- Subject's age at baseline and sex
- Time on treatment at the onset of the event [derived as: treatment start date AE start date +1 day]

#### • Part 2:

- Event severity: Mild; Moderate; Severe
- Relationship to study treatment: Related; Not related
- Action taken with study treatment: None; Permanently withdrawn, Temporary interrupted; Dose increased; Dose reduced
- Other action taken: None; Concomitant Medication given; Withdrawn; Other
- Outcome: Completely resolved; Resolved with sequelae; Improved; Ongoing;
  Worsened; Death; Unknown

# 9.1.2. Summaries of Adverse Incidence Rates for Serious Adverse Events (SAE), Adverse Event Dropouts, and Death

All SAEs will be listed as above by treatment group (refer to Section 9.1.1).

The following criteria for the SAE will be included in this listing. The criteria are as follows:

- Fatal
- Life threatening
- Required inpatient hospitalization
- Hospitalization prolonged
- Persistent or significant disability or incapacity

- Congenital anomaly/birth defect
- Other medically significant event

# 9.2. Total Duration of Therapy, Average Daily Dose, Maximum Daily Dose, Final Daily Dose of Study Medication, and Compliance

On Visit 2 and Visit 7, the count and percentage of subjects who received any infusion of study treatment will be summarized by treatment group and overall. Descriptive statistics for the percentage compliance will be summarized at each visit and overall by treatment group and overall.

The daily percentage compliance for each subject will be derived as:

(actual volume administered / planned volume to be administered) x 100.

The total percentage compliance for each subject will also be calculated as:

(Visit 2 actual volume administered + Visit 7 actual volume administered) / (Visit 2 planned volume to be administered + Visit 7 planned volume to be administered) x 100.

For total percentage compliance, if a subject discontinues the study before their Visit 7, the actual and planned volume for Visit 7 will be both zero.

A subject listing will also be provided containing IV infusion data and compliance calculations.

## 9.3. Concomitant Medications and Non-Drug Treatments

Concomitant medications that subjects took after the baseline visit will be summarized by treatment group and overall. Concomitant medications will be coded using WHO DDE (September 2015).

A supportive subject listing will be provided including trade and generic drug names, start and stop dates, days relative to the start of treatment [derived as: Concomitant start date – treatment start date + 1 day], dose, frequency, route, and indication(s).

Concomitant non-drug treatment will also be summarized by treatment group and overall in a separate table and listing.

Rescue medications and treatments will be summarized in a separate table and listing to concomitant medications and concomitant non-drug treatment (see Section 9.8 for further details).

# 9.4. Routine Laboratory Data

Summary tables will be presented for each parameter [for a full list of laboratory parameters see below] by treatment group of the following of laboratory categories: Haematology, Serum
Biochemistry, Liver function tests, Renal function tests, Lipid Profile, Urinalysis, Serology, Other. Descriptive statistics will be used to summarize the data:

- Quantitative laboratory test result will include count, mean, s.d., median, minimum and maximum.
- Qualitative tests (e.g. some urinalysis assessments) will be categorized accordingly.

Analyses of the laboratory data will focus on the changes from baseline to each planned visit. For each laboratory test, there will be three sets of descriptive statistics that summarize the results at baseline, result at each visit, and the change from baseline to each visit. The final assessment available will also be summarized.

Shift tables will be included that summarize the count and percentage by laboratory parameter of the following categories:

- Abnormal, low
- Normal
- Abnormal, high
- Missing

Changes from baseline to the worst post-baseline values for each subject will be displayed. Unscheduled visits will be considered for the worst post baseline result. The following categories will also be presented if there is both an abnormal, low and abnormal, high shift post baseline.

• Abnormal, (low and high)

The supportive listings for hematology, serum chemistry, and urinalysis will include the sample collection date, time of collection, and relative day; type of visit; subject age at baseline and sex; and laboratory test, lab test units, and lab test result; and the lower and upper limits of normal.

#### 9.4.1. Laboratory tests

The following laboratory tests will be summarized:

Haematology

- Haemoglobin (g/L)
- Hematocrit (V/V)
- White blood cell count (x10E9/L)
- Differential white cell count (%)
- Red blood cell count with mean cell volume, mean cell hemoglobin and mean cell hemoglobin concentration (x10E12/L)

• Platelets (x10E9/L)

## Serum Biochemistry

- Electrolytes (TBC)
- Sodium (mmol/L)
- Potassium (mmol/L)
- Calcium (mmol/L)
- Chloride (mmol/L)
- Bicarbonate (mmol/L)

#### Liver function tests

- Total and direct bilirubin (umol/L)
- Total protein (g/L)
- Globulin (g/L)
- Albumin (g/L)
- AST (U/L)
- ALT (U/L)
- GGT (U/L)
- ALP (Alkaline phosphatase) (IU/L)
- Lactate dehydrogenase (U/L)

## Renal function tests

- Creatinine (umol/L)
- Blood urea nitrogen (BUN) (mmol/L)

## Other

- Fasting blood sugar (TBC)
- Serum FSH (female, only at screening) (IU/L)
- Serum and urine Beta-HCG (for females only) (N/A)
- Serum Immunoglobulins (TBC)

# Lipid Profile

- Total cholesterol (mmol/L)
- Triglycerides (mmol/L)
- HDL (mmol/L)
- LDL (mmol/L)
- VLDL (mmol/L)

## Urinalysis

- pH (N/A)
- Specific gravity (N/A)

#### Other

- QuantiFERON Gold Blood TB Test (N/A)
- Total IgE (kU/L)
- Circulating eosinophils count (TBC)

# 9.5. Vital Signs

Descriptive statistics will be used to summarize post baseline vital sign results and also changes from baseline by treatment group at each planned visit. Vital signs will be summarized at each visit and at 30 minute time points during infusion visits.

Descriptive statistics will be provided for the following vital sign parameters:

- Systolic blood pressure (mmHg)\*
- Diastolic blood pressure (mmHg)\*
- Body temperature (°C)
- Pulse rate (beats per minute [bpm])\*
- Weight (kg)
- BMI  $(kg/m^2)$

<sup>\*</sup>Blood pressure and pulse rate is to be tested in supine or semi-supine position.

At each planned visit, blood pressure, body temperature and pulse rate will be categorized as normal; abnormal, not clinically significant; abnormal, clinically significant.

Shift tables will present changes from baseline to the worse post-baseline values for the following categories:

- Normal
- Abnormal, not clinically significant
- Abnormal, clinically significant
- Missing

Unscheduled visits will be considered for the worst post baseline result.

All vital signs data will be displayed in a subject listing and clinically significant findings will be flagged.

# 9.6. Physical Examination

The results of the brief physical examination will be summarized by treatment group. Summaries will be presented at baseline and for the worst post-baseline result only. The following body systems will be summarized:

- Thorax/Lungs
- Cardiovascular system
- Neurological examination
- Other

Each body system will be categorized into one of the following: normal; abnormal, not clinically significant; abnormal, clinically significant. The count and percentage of subjects in each category will be summarized by treatment group and overall. The count and percentage of subjects whose brief physical examination is not performed will also be summarized.

The body system data at each visit will be listed and clinically significant values will be flagged.

#### 9.7. ECG

Subjects undergo a 12-lead ECG assessment either singularly or in triplicate at each planned visit. Triplicate ECGs are performed only if clinically significant abnormalities are detected in the subject's single ECG..

The change from baseline will be summarized at each planned visit by treatment group for single ECG. If there are multiple single, then the last available information for that parameter at that

visit will be used for the summary. The following measures will be reported using descriptive statistics:

- Heart rate (bpm)
- PR interval (ms)
- RR interval (ms)
- QRS duration (ms)
- QT interval (ms)
- QTcF interval (ms)

For the overall interpretation of the ECGs at each visit, the count and percentage of subjects for each of the following categories will be reported by treatment group and overall:

- Normal
- Abnormal, non clinically significant
- Abnormal, clinically significant
- Missing

The QTc prolongations below will also be summarized by treatment group and overall:

- QTc interval at any visit > 500ms
- QTc interval increases from baseline > 60ms

For the analysis of the triplicate, the categorization will be derived using worst-case scenario rules such that the following order of precedence will be used: Abnormal, clinically significant; abnormal, non clinically significant; normal.

The ECG will also be listed and clinically significant values will be flagged.

## 9.8. Rescue Medication

Concomitant rescue medications/treatments will be summarized using counts and percentages by treatment group and overall.

Rescue medications/treatments will be coded by WHO DDE (September 2015) and the count and percentage of each preferred term (generic medication) will be summarized by treatment group and overall.

The data for each subject who received rescue medications will also be listed including the preferred term, dose/unit, route and frequency, start study day of rescue medication/treatment, duration of treatment and whether the treatment is ongoing.

# 9.9. Study Termination Status

The end of study status by treatment group is described as part of subject disposition (Section 7.1).

#### 10. CLINICAL PHARMACOLOGY DATA ANALYSES

The Pharmacokinetic (PK) of GBR 830 in adult subjects with moderate to severe AD in terms of  $C_{max}$ ,  $AUC_{0-tau}$ ,  $T_{max}$ ,  $AUC_{0-t}$ ,  $AUC_{0-\infty}$ ,  $t_{1/2}$ , volume of distribution and clearance will be assessed as relevant after the first and last doses.

All PK analysis will be performed on the Pharmacokinetic Analysis Set.

# 10.1. Pharmacokinetic/ Pharmacodynamic Analyses

PK parameters will be calculated from the GBR 830 concentration-time data using SAS v9.4. PK parameters will be estimated from the pre dose time point of each infusion, infusions will take place on Day 1 and 29. Measures will be taken within 15 minutes of administration of each dose (pre dose), immediately at the end of each infusion; then at, 1.5, 2, 4, 72, 168, 336, 504 hours after the start of each infusion; and on Day 57 (1344 hours from the first infusion), 71 (1680 hours), and 85 (2016 hours).

Partial or missing time point information will not be considered in the analysis.

Non-compartmental methods will be used to analyze the PK data. Actual sampling time points will be used for the calculation of PK parameters.

#### **10.1.1.** Dosing intervals

The dosing interval for the first IV infusion will consist of the following time points: pre dose, end of infusion; then at 1.5, 2, 4, 72, 168, 336, 504 hours from the start time of the first infusion, as well as pre dose for the second infusion.

The dosing interval for the second IV infusion will consist of the following time points: pre dose, end of the infusion; then at 1.5, 2, 4, 72, 168, 336, 504 hours from the start time of the second infusion, as well as Day 57. This time duration will be used for the calculation of  $AUC_{0-tau}$ .

In addition, PK samples are collected at day 71 and day 85. These data will be included in calculation of  $AUC_{0-t}$  and  $AUC_{0-\infty}$ .

#### **10.1.2.** Analysis of Parameters

The parameters will be estimated for each dosing intervals as follows:

**Table 2:** PK Parameters

| Parameter name | Description |
|---|---|
| $C_{\text{max}}$ | Maximum observed Concentration after each dosing interval. This will be provided after each dosing event. |

| Parameter name | Description |
|---|---|
| $T_{\text{max}}$ | Time at which $C_{\text{max}}$ was observed. This will be provided after each dosing event. |
| AUC <sub>0-tau</sub> | Trapezoid calculation of area under the serum drug concentration-time curve from time zero (pre dose time point of the infusion) to the end of the dosing interval. This will be provided after each dosing event. |
| AUC <sub>0-t</sub> | Calculation of area under the serum drug concentration-time curve from time zero (pre dose time point of the infusion) to the last time point where quantifiable concentration is observed. This will be provided after each dosing event. |
| AUC <sub>0-∞</sub> | Total AUC computed by combining AUC <sub>0-t</sub> with extrapolated AUC. This will be provided after the second dosing event only. |
| %AUC extrapolated | Percentage extrapolated AUC; This will be provided after the second dosing event only. Only presented if %AUC extrapolated is less than ≤ 20% |
| $\lambda_{\rm z}$ | Terminal elimination rate constant. This will be provided after the second dosing event only. Linear regression of at least three points and an $r^2$ greater than 0.80 are required to retain $\lambda z$ and associated parameters $t_{1/2}$ , $V_d$ , $AUC_{0-\infty}$ . |
| t <sub>1/2</sub> | Half life This will be provided after the second dosing event only. |
| $V_{d}$ | Observed apparent volume of distribution. This will be provided after the second dosing event only. |
| CL | Observed Clearance. This will be provided after the second dosing event only. |
| C <sub>trough</sub> | Trough concentration. Concentration at 672 hours after each infusion (day 29 and day 57) |

# Elimination Rate

Initially to estimate the elimination rate coefficient a linear regression model will be fitted to the individual  $log_{10}$  elimination phase concentration values. The elimination phase is defined between maximum observed concentration and last observed value above the LLOQ. The elimination rate constant is defined as

$$\lambda_z = -2.303 \text{ x slope}$$

Half life (calculated only after second dose)

$$t_{1/2} = \frac{0.693}{\lambda_z}$$

Area under the curve to the last measurable concentration (after each dosing interval)

$$AUC_{0-t} = \sum_{i=0}^{n-1} \frac{t_{i+1} - t_i}{2} (C_i + C_{i+1})$$

Where n is the number of data points.

The area under the concentration curve from time '0' to up to the last time point where quantifiable serum concentrations were observed will be calculated separately for both the dosing occasions. The start time of infusion, for each dosing occasion, would be considered as time '0' for the calculation of AUC<sub>0-t</sub>. The pre dose serum concentration (concentration in the sample collected closest to the start of infusion) would be considered as the concentration at time '0'. The last data point considered for the calculation of AUC<sub>0-t</sub> after the 1<sup>st</sup> dosing event would be the pre dose serum concentrations on day 29 and after 2<sup>nd</sup> dosing event would be the serum concentration on day 85, respectively. If the data point is not available on either of these occasions, the closest time point where the serum concentrations are available would be used for the calculation of AUC<sub>0-t</sub>.

Area under the curve over the dosing interval (after each dosing event)

$$AUC_{0-tau} = \sum_{i=0}^{n-1} \frac{t_{i+1} - t_i}{2} (C_i + C_{i+1})$$

Where n is the number of data points in each interval.

The area under the concentration curve for each dosing interval would be calculated separately after each dosing occasion. The start time of infusion, for each dosing occasion, would be considered as time '0' for the calculation of  $AUC_{0-tau}$ . The pre-dose serum concentration (concentration in the sample collected closest to the start of infusion) would be considered as the concentration at time '0'. The last data point considered for calculation of  $AUC_{0-tau}$  after the 1<sup>st</sup> dosing event would be the pre dose serum concentrations on day 29 and after 2<sup>nd</sup> dosing event would be the serum concentration on day 57, respectively. If the data point is not available on either of these occasions, the closest time point where the serum concentrations are available would be used for the calculation of  $AUC_{0-tau}$ .

Area under the curve extrapolated to infinity (calculated only after second dose)

$$AUC_{\infty} = AUC_{0-t} + \frac{C_n}{\lambda_z}$$

Observed Volume of Distribution at steady state (calculated only after second dose)

$$V_d = \frac{\mathsf{D}}{AUC_{0-tau \times} \lambda_z}$$

(Where D is actual dose received)

Observed Clearance (calculated only after second dose)

$$CL = \frac{D}{AUC_{0-tau}}$$

(Where D is actual dose received)

## 10.1.3. Handling of values below the limit of quantification

When the value that is recorded as below the limit of quantification (BLQ), this will be treated as either zero or missing dependant upon when the BLQ value was observed relative to other non BLO values. Details are below.

- The BLQ value before the beginning of the infusion (Pre dose) will be set to zero.
- All BLQ values observed between the start of infusion and the first observed concentration will be treated as zero
- If a single BLQ value is observed at a time between two non-zero observations it will be treated as missing.
- When two or more BLQ consecutive values are observed these will be treated as zero until the next observed non-zero value.
- All BLQ values after the last measurable observation (C<sub>n</sub>) after each dosing will be treated as zero.

These rules will be applied to the estimation of individual PK parameters detailed above and in the calculation of summary statistics for serum concentration levels and the plot of mean concentration curves. For semi-log plots all BLQ values will be set to missing.

## **10.1.1.** Treatment of outliers

Individual concentration time points or entire individual treatment profiles, if considered anomalous, may be excluded from the analysis at the discretion the pharmacokineticist following a review of the available documentation. Any such exclusion will be clearly outlined in the CSR.

# 11. CHANGES FROM THE PLANNED PROTOCOL ANALYSIS

# 11.1. Shift Tables

All shift tables will now be presented as baseline to worst post baseline visit, rather than on a by visit basis.

# 11.2. Exploratory Cytokines Analysis

Cytokines will now be analyzed post data base lock.

# APPENDIX 1. SCHEDULE OF EVENTS

| Visit' | Screen-<br>ing | Base-<br>line<br>visit | | Follow- | up visits | | Dosing<br>visit | | Follow-up visits | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Day | -30 to -1 | 1 | <b>4</b> 1 | 8 <u>±</u> 1 | 15 <u>±</u> 1 | 22±2 | 29 <u>±</u> 1 | 32 <u>±</u> 1 | 36 <u>±</u> 1 | 43 <u>±</u> 1 | 50±2 | 57±2 | 71 <u>±</u> 2 | 85 <u>±</u> 2 |
| Visit ID | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | п | 12 | 13 | 14 |
| Informed consent | х | | | | | | | | | | | | | |
| Medical history <sup>1</sup> | ж | | | | | | | | | | | | | |
| Demographics (in d. height, weight and BMI) | х | х | | | | | ж | | | | | | | ж |
| Physical examination* | х | х | | | ж | | х | | | ж | | | | ж |
| TB testing <sup>c</sup> | х | | | | | | | | | | | | | |
| Vital signs* | х | х | ж | ж | ж | х | ж | ж | ж | ж | х | ж | ж | ж |
| 12-lead EC G <sup>r</sup> | х | х | ж | ж | | | х | ж | ж | | | х | ж | ж |
| Clinical lab gratory <sup>6</sup> | х | х | х | х | | | х | х | ж | | | х | ж | х |
| Drug and alcohol screen? | х | ж | | | | | х | | | | | | | |
| HBs Ag, Anti-HBc Ag, HCV and HIV tests | х | | | | | | | | | | | | | |
| Serum pregnancy (females only) <sup>10</sup> | х | х | | | | | | | | | | | | х |
| Urine pregnancy (females only) " | | х | | | | | х | | | | | | | |
| EAS I SCORAD, IGA, BSA 13.15 | х | х | ж | ж | ж | ж | ж | ж | ж | ж | ж | ж | ж | ж |
| Whole body photography " | | х | | ж | | | | | | ж | | | | ж |
| DLQĮ NRS | | х | х | ж | х | х | х | ж | ж | ж | х | х | ж | ж |

| Visit! | Screen-<br>ing | Base-<br>line<br>visit | | Follow- | up visits | | Dosing<br>visit | Follow-up visits | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Day | -30 to -1 | 1 | <b>4</b> <u>1</u> 1 | 8 <u>±</u> 1 | 15 <u>±</u> 1 | 22±2 | 29 <u>±</u> 1 | 32 <u>±</u> 1 | 36 <u>±</u> 1 | 43 <u>±</u> 1 | 50±2 | 57±2 | 71 <u>±</u> 2 | 85 <u>±</u> 2 |
| Visit ID | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 |
| Withdraw medication & dispense diary * | х | | | | | | | | | | | | | |
| Inclusion/exclusion criteria | х | х | | | | | | | | | | | | |
| Randomisation 15 | | х | | | | | | | | | | | | |
| Study drug administration <sup>16</sup> | | х | | | | | ж | | | | | | | |
| Previous and concomitant therapies | х | х | ж | х | ж | х | ж | ж | ж | ж | ж | ж | ж | ж |
| PK sampling for GBR 83017 | | ж | ж | х | ж | х | х | ж | ж | ж | ж | ж | ж | ж |
| Leukocyte sub-population cell counts, TEWL,<br>total IgE, eosinophil <sup>15</sup> | | х | | х | х | | х | | х | х | | х | ж | х |
| Cytokines and exploratory analysis 15 | | х | | | | | х | | | | | | ж | |
| Immunogenicity samples" | | ж | | | ж | | х | | | | | ж | | ж |
| Skin hiopsies <sup>10</sup> | | х | | | | | ж | | | | | | ж | |
| Adverse events <sup>11</sup> | х | х | х | х | ж | х | х | ж | ж | ж | ж | ж | ж | х |
| Phone call <sup>11</sup> | | х | | | | | х | | | | | | | |

# Appendix 1– Footnotes

<sup>1.</sup> Visits do not include a Day 0. Visit 1 procedures may be conducted over more than 1 day as long as all tasks are completed within the allowable visit tolerance (at least 3 days should be allowed for receipt of laboratory test results). On visits subjects should fast for at least 4 hours prior to safety sample collection. The last assessments done prior to dosing will be considered as baseline. The last follow-up visit on Day 85 will be considered the end-of study assessments will be done in place of visit procedures, for all subjects receiving the study medication for all early withdrawal and dropouts. Visits and assessments done in relation to the second infusion will be calculated from the actual day/start time of the second infusion. This applies to V8 to V11, inclusively. For V12, V13, and V14, the time points for assessment will be 672hr, 1008hr, and 1344hr, respectively, from the start time of the second infusion.

<sup>2.</sup> Medical history includes recent medical history (any illness occurring within past 4 weeks), previous medical history (only significant medical or surgical illness), smoking, alcohol and intake of drugs of abuse)

- 3. Demographics: includes date of birth, gender, race and ethnicity, height and body weight. BMI will be calculated as weight (kg) / [height (m) x height (m)]. Only body weight will be repeated at subsequent visits. Height measured at screening will be used for calculation of BMI at subsequent visits
- 4. Physical examination: Comprehensive examination at screening and brief examination at all subsequent visits.
- 5. TB testing: Subjects must test negative for a QuantiFERON Gold-TB test done at screening.
- 6. Vital signs: includes supine or semi-supine BP and pulse; and body temperature at screening, within 30 minutes before administration,  $0.5 \pm 10$  mins during infusion,  $1.0 \pm 10$  mins,  $2.0 \pm 10$  mins and 6.0 hours  $\pm 10$  mins estimated from the end time of the first infusion, and within 30 minutes before administration,  $0.5 \pm 10$  mins during infusion,  $1.0 \pm 10$  mins,  $2.0 \pm 10$  mins and 3.0 hours  $\pm 10$  mins estimated from the end time of the second infusion and at each follow-up visit. Vitals have to be monitored every half hour during infusion.
- 7. A single ECG will be taken at screening, at pre-dose,  $2 \pm 30$  mins and 6 hours  $\pm 30$  mins estimated from the end time of the first infusion, at pre-dose,  $2 \pm 15$  mins and 3 hours  $\pm 15$  mins estimated from the end time of the second infusion, and on Day 4, Day 8, Day 32, Day 36, Day 57, Day 71 and on Day 85. A triplicate ECG will be taken if there are any clinically significant abnormalities detected by the physician in single ECG.
- 8. Clinical laboratory tests (labs) include hematology, biochemistry and urinalysis after a 4-hour fast. Detailed panel mentioned in Appendix 2. Labs will be done at screening, Day 1 (pre-dose), Day 4, Day 8, Day 29 (pre-dose), Day 32, Day 36, Day 57, Day 71 and Day 85. Serum FSH and viral serology will be done only at screening.
- 9. Drug and alcohol screen: alcohol or drugs of abuse at screening and before administration of each dose (pre-dose). Drug screen includes amphetamines, BZD, barbiturates, cocaine, opioids, and cannabinoids.
- 10. Serum pregnancy test for women will be done during screening, Day 1 and at the end of study.
- 11. Urine pregnancy test for women will be done before administration of each dose (pre-dose). Results of the pregnancy test should be negative before dispensing of study drug(s)
- 12. Efficacy assessments will be done by a trained, blinded assessor. The same assessor should do the assessments of a particular subject throughout the study. Assessments will be done at screening, at baseline (pre-dose on Day 1), at Days 4, 8, 15, 22, 29 (pre-dose), 32, 36, 43, 50, 57, 71, and 85. If the subject signs for optional consent for photography, whole body photography (from neck down-anterior and posterior), will be taken, at baseline and at Days 8, 43, and 85.
- 13. BSA will be done by the same assessor performing other efficacy assessment, and at similar time points.
- 14. Subject must enter data into the diary every day from start of screening period to end of study visit. Subject will be trained on the use of diary. Subject will be instructed to enter the data every morning at a designated time and how to record them.
- 15. Day of randomization and first dosing are assumed to be same, no waiver allowed. Randomization schedule will be prepared using a centralized computer-based IVRS/IWRS system.
- 16. IP administration: Continuous slow IV infusion for 60 min. The infusion volume must be calculated using the patient's current body weight. The study site will contact subjects by telephone approximately 24 hours after each infusion of IP.
- 17. Serum samples for GBR-830 PK analysis will be obtained 15 minutes before administration of each dose (pre-dose), immediately at the end of each infusion  $\pm$  10 mins; at 1.5  $\pm$  10 mins, 2  $\pm$  10 mins, 4  $\pm$  10 mins hours estimated from the start time of infusion, 72, 168, 336, 504 hours after each infusions; and on Day 57 (1344 hours), 71 (1680 hours), and 85 (2016 hours) estimated from the start time of first infusion. Visits and assessments done in relation to the second infusion will be calculated from the actual day/start time of the

# Glenmark Pharmaceutical SA Statistical Analysis Plan – Protocol GBR 830-201

6-Jul-17

second infusion. This applies to V8 to V11, inclusively. For V12, V13, and V14, the time points for assessment will be 672hr, 1008hr, and 1344hr, respectively, from the start time of the second infusion.

- 18. Leukocyte sub-population cell counts, TEWL, total IgE, eosinophil will be done on Day 1, 8, 15, 29, 36, 43, 57, 71, and 85. Samples for TARC, eotaxin-3, and cytokine panel and additional exploratory analysis will be taken at baseline, at Day 29, and Day 71. TEWL assessment is being performed by sites as per the TEWL manual and a predefined time point as per protocol will not be applicable.
- 19. Samples will be collected for immunogenicity analysis at pre-dose, and at Day 15, (pre-dose) Day 29, Day 57, and Day 85.
- 20. Skin biopsies will be taken at baseline at Day 29, and Day 71.
- 21. Adverse events will be reported as described and classified in the CTCAE version 4.03. At each visit, the Investigator will ask the subject whether he/she has received medical care by another physician since the last visit or is planning to do so in the future.
- 22. The site will contact the subject 24 hours after each infusion by phone.

# APPENDIX 2. TABLE OF CONTENTS FOR DATA DISPLAY SPECIFICATIONS

| | Title | Analysis set | Comments<br>(*subject to<br>request) | New table<br>number* |
|---|---|---|---|---|
| Study Popu | ulation Section | | | |
| Table 14.1.1 | Subject Disposition | Screened<br>Subjects | Unique | Table 14.1.1 |
| Table 14.1.2 | Analysis Sets | Randomized<br>Subjects | Unique | Table 14.1.2 |
| Table 14.1.3 | Study Participation | Full Analysis<br>Set | Unique | Table 14.1.3 |
| Table 14.2.1.1 | Demographic Characteristics | Full Analysis<br>Set | Unique | Table 14.1.4.1.1 |
| Table 14.2.1.2 | Demographic Characteristics | Biological<br>Activity Set | Repeat | Table 14.1.4.1.2 |
| Table 14.2.1.3 | Demographic Characteristics | Pharmacokineti<br>c Analysis Set | Repeat | Table 14.1.4.1.3 |
| Table 14.2.2 | Atopic Dermatitis (AD) History | Full Analysis<br>Set | Unique | Table 14.1.4.2 |
| Table 14.2.3 | Medical/Surgical History | Full Analysis<br>Set | Unique | Table 14.1.4.3 |
| Table 14.2.4 | Smoking, Alcohol and Drug Abuse History | Full Analysis<br>Set | Unique | Table 14.1.4.4 |
| Table 14.2.5.1 | Atopic Dermatitis and Related Conditions<br>Baseline Prior Medications | Full Analysis<br>Set | Unique | Table 14.1.5.1 |
| Table 14.2.5.2 | Other Baseline Prior Medications | Full Analysis<br>Set | Repeat | Table 14.1.5.2 |
| Table 14.2.10 | Baseline Clinical Scores | Full Analysis<br>Set | Unique | Table 14.1.6 |
| Table 14.2.11.1 | Baseline Active AD mRNA Expression<br>Signatures Obtained from Skin Biopsies (Non<br>Lesion Samples) | Biological<br>Activity Set | Repeat | Table 14.1.7.1 |
| Table 14.2.11.2 | Baseline Pathologic Epidermal Phenotype<br>Measures Obtained from Skin Biopsies (Non<br>Lesion Samples) | Biological<br>Activity Set | Repeat | Table 14.1.7.2 |
| Efficacy Se | ection | | | |
| <u>Tables</u> | | | | |

| | Title | Analysis set | Comments<br>(*subject to<br>request) | New table<br>number* |
|---|---|---|---|---|
| 14.3.1.1a | MMRM Analysis Selected Active AD mRNA<br>Expressions (Normalized to hARP) Obtained<br>from Skin Biopsies (Lesion Samples)- Primary<br>Analysis | Biological<br>Activity Set | Unique | Table 14.2.1.1a |
| Table 14.3.1.1b | Change from Baseline in the Selected Active AD mRNA Expression Signatures (Normalized to hARP) Obtained from Skin Biopsies by Lesion Location –Primary Analysis | Biological<br>Activity Set | Unique | Table 14.2.1.1b |
| Table 14.3.1.2 | Change from Baseline in H&E Thickness Obtained from Skin Biopsies by Lesion Location – Primary Analysis | Biological<br>Activity Set | Unique | Table 14.2.1.2 |
| Table 14.3.1.3 | Summary of K16 Obtained from Skin Biopsies by<br>Lesion Location and Visit – Primary Analysis | Biological<br>Activity Set | Unique | Table 14.2.1.3 |
| Table 14.3.1.4 | Summary of Histological Response Obtained<br>from Skin Biopsies by Lesion Location and Visit<br>– Primary Analysis | Biological<br>Activity Set | Unique | Table 14.2.1.4 |
| Table 14.3.1.5 | Summary of IHC Panel from Skin Biopsies by<br>Visit – Primary Analysis | Biological<br>Activity Set | Unique | Table 14.2.1.4 |
| Table 14.2.2 | Proportion of Subjects who Achieved an IGA<br>Score of 0 or 1 by Visit | Biological<br>Activity Set | Unique | Table 14.2.2 |
| Table 14.3.3.1 | Proportion of Subjects who Achieved an EASI 50<br>Response by Visit | Full Analysis<br>Set | Unique | Table 14.2.3.1 |
| Table 14.3.3.2 | Proportion of Subjects who Achieved an EASI 75<br>Response by Visit | Full Analysis<br>Set | Repeat | Table 14.2.3.2 |
| Table 14.3.3.3 | Analysis of Covariance (ANCOVA) of change from baseline in EASI Score to Visit 12 LOCF | Full Analysis<br>Set | Unique | Table 14.2.3.3 |
| Table 14.3.4.1 | Percent Change from Baseline in EASI Clinical<br>Score at Each Visit | Full Analysis<br>Set | Unique | Table 14.2.4.1 |
| Table 14.3.4.2 | Percent change from Baseline in SCORAD<br>Clinical Score at Each Visit | Full Analysis<br>Set | Repeat | Table 14.2.4.2 |
| Table 14.3.4.3 | Percent Change from Baseline in IGA Clinical<br>Score at Each Visit | Full Analysis<br>Set | Repeat | Table 14.2.4.3 |
| Table 14.3.4.4 | Percent change from Baseline in Pruritus NRS<br>Clinical Score at Each Visit | Full Analysis<br>Set | Repeat | Table 14.2.4.4 |
| Table 14.3.4.5 | Percent change from Baseline in DLQI Clinical<br>Score at Each Visit | Full Analysis<br>Set | Repeat | Table 14.2.4.5 |
| Table 14.3.5 | Changes from Baseline in Transepidermal Water<br>Loss (g/m2/h) by Lesion/Non-Lesion Area | Full Analysis<br>Set | Unique | Table 14.2.5 |
| Table 14.3.6 | Anti-Drug Antibodies to GBR 830 by Visit | Full Analysis<br>Set | Unique | Table 14.2.6 |

| | Title | Analysis set | Comments<br>(*subject to<br>request) | New table<br>number* |
|---|---|---|---|---|
| Table 14.3.8 | Changes from Baseline in Leukocytes Sub-<br>Population Cell Counts | Full Analysis<br>Set | Unique* | Table 14.2.7 |
| Table 14.3.9 | Changes from Baseline in Cellular Infiltrates | Full Analysis<br>Set | Repeat* | Table 14.2.8 |
| Table 14.3.10 | Changes from Baseline in Serum Total<br>Immunoglobulin E, Serum Soluble OX40, Serum<br>Soluble OX40 and Circulating Eosinophil Counts | Full Analysis<br>Set | Repeat* | Table 14.2.9 |
| Table 14.3.12 | Prohibited Medications | Full Analysis<br>Set | Unique | Table 14.2.10 |
| Safety Sect | tion | | | |
| <u>Tables</u> | | | | |
| Table 14.4.1 | Overall Treatment Emergent Adverse Events | Safety Analysis<br>Set | Unique | Table 14.3.1.1.1 |
| Table 14.4.2.1 | Treatment Emergent Adverse Events | Safety Analysis<br>Set | Unique | Table 14.3.1.1.2 |
| Table 14.4.2.2 | Serious Treatment Emergent Adverse Events | Safety Analysis<br>Set | Repeat | Table 14.3.1.2 |
| Table 14.4.2.5 | Treatment Emergent Adverse Events Leading to Discontinuation of Study | Safety Analysis<br>Set | Repeat | Table 14.3.1.3 |
| Table 14.4.2.6 | Treatment Emergent Adverse Events Related to the Investigational Product | Safety Analysis<br>Set | Repeat | Table 14.3.1.4 |
| Table 14.4.2.7 | Treatment Emergent Adverse Events Leading to Death | Safety Analysis<br>Set | Repeat | Table 14.3.1.5 |
| Table 14.4.2.8 | Treatment Emergent Adverse Events by Severity | Safety Analysis<br>Set | Unique | Table 14.3.1.6 |
| Table 14.4.3 | Study Drug Treatment Compliance | Safety Analysis<br>Set | Unique | Table 14.3.6.1.1 |
| Table 14.4.4.1 | Concomitant Medications for Atopic Dermatitis and Related Conditions | Safety Analysis<br>Set | Unique | Table 14.3.6.2.1 |
| Table 14.4.4.2 | Concomitant Non-Drug Treatments | Safety Analysis<br>Set | Repeat | Table 14.3.6.2.2 |
| Table 14.4.4.3 | Rescue Medications | Safety Analysis<br>Set | Repeat | Table 14.3.6.2.3 |
| Table 14.4.5.1 | Change from Baseline in Laboratory Results by Category | Safety Analysis<br>Set | Unique | Table 14.3.5.1 |
| Table 14.4.5.2 | Shift Table of Laboratory Results from Baseline to Worst Post Baseline Result by Category and Treatment Group | Safety Analysis<br>Set | Unique | Table 14.3.5.2 |
| Table 14.4.6.1 | Change from Baseline in Vital Signs Results | Safety Analysis<br>Set | Unique | Table 14.3.6.3.1 |

| | Title | Analysis set | Comments<br>(*subject to<br>request) | New table<br>number* |
|---|---|---|---|---|
| Table 14.4.6.2 | Shift Table of Vital Signs from Baseline to Worst<br>Post Baseline Result by Treatment Group | Safety Analysis<br>Set | Unique | Table 14.3.6.3.2 |
| Table 14.4.7 | Physical Examination Results | Safety Analysis<br>Set | Unique | Table 14.3.6.4 |
| Table 14.4.8.1 | Change from Baseline in Electrocardiogram<br>Results | Safety Analysis<br>Set | Unique | Table 14.3.6.5.1 |
| Table 14.4.8.2 | Overall Interpretations of Electrocardiogram | Safety Analysis<br>Set | Unique | Table 14.3.6.5.2 |
| Table 14.4.9 | GBR830 Serum Concentration (ng/mL) Data | Pharmacokineti<br>c Analysis Set | Unique | Table 14.3.6.7 |
| Table 14.4.10 | Pharmacokinetic Parameters of GBR830 | Pharmacokineti<br>c Analysis Set | Unique | Table 14.2.10.1 |
| <u>Figures</u> | | | | |
| Figure 14.3.1.1 | Box plot of biomarker CCL11/hARPby Planned<br>Treatment Group | Biological<br>Activity Set | Unique | Figure 14.2.1 |
| Figure 14.3.3.1 | Line Plot of EASI 50 Responders over Time (days) by Planned Treatment Group | Full Analysis<br>Set | Unique | Figure 14.2.2 |
| Figure 14.3.4.1 | Line Plot of Mean ± SE Percentage Change in EASI Score over Time (days) by Planned Treatment Group | Full Analysis<br>Set | Repeat | Figure 14.2.3 |
| Figure 14.3.4.4 | Line Plot of Mean ± SE Percentage Change in<br>Pruritus NRS over Time (days) by Planned<br>Treatment Group | Full Analysis<br>Set | Repeat | Figure 14.2.4 |
| Figure 14.3.6.1 | Scatter Plot of Serum Concentration (µg/mL) over<br>Anti Drug Antibody Status by Planned Treatment<br>Group | Pharmacokineti<br>c Analysis Set | Unique | Figure 14.2.5 |
| Figure 14.4.11.1 | Mean Serum GBR830 Concentration Data (0 to 2016 hours) Overall | Pharmacokineti<br>c Analysis Set | Unique | Figure 14.2.6.1 |
| Figure 14.4.11.2 | Individual Subject Profiles of Serum GBR830<br>Concentration Data (0 to 2016 hours) | Pharmacokineti<br>c Analysis Set | Unique | Figure 14.2.6.2 |

<sup>\*</sup>New number will be used in final displays

# Listings

| | Title | Population | Comment | New<br>Number* |
|---|---|---|---|---|
| Listing 16.1.1 | Subject Disposition | Randomized Subjects | Unique | Listing 16.2.1.1 |
| Listing 16.1.2 | Analysis Populations | Screened Subjects | Unique | Listing 16.2.3.1 |
| Listing 16.1.3 | Subject Inclusion/Exclusion Criteria | Screened Subjects | Unique | Listing 16.2.1.2 |
| Listing 16.1.4 | Screen Failure Subjects | Screened Subjects | Unique | Listing 16.2.1.3 |
| Listing 16.1.5 | Subject Randomization Information | Randomized Subjects | Unique | Listing 16.1.7 |
| Listing 16.2.1.1.1 | Subject Demographic and Baseline<br>Characteristics – Part 1 | Randomized Subjects | Unique | Listing 16.2.4.1 |
| Listing 16.2.1.1.2 | Subject Demographic and Baseline<br>Characteristics – Part 1 | Screen Failure Subjects | Repeat | Listing 16.2.4.2 |
| Listing 16.2.1.2.1 | Subject Demographic and Baseline<br>Characteristics – Part 2 | Randomized Subjects | Unique | Listing 16.2.4.3 |
| Listing 16.2.1.2.2 | Subject Demographic and Baseline<br>Characteristics – Part 2 | Screen Failure Subjects | Repeat | Listing 16.2.4.4 |
| Listing 16.2.2 | Atopic Dermatitis History | Randomized Subjects | Unique | Listing 16.2.4.5 |
| Listing 16.2.3 | Medical/Surgical History | Randomized Subjects | Unique | Listing 16.2.4.6 |
| Listing 16.2.4.1 | Smoking, Alcohol and Drug Abuse<br>History – Part 1 | Randomized Subjects | Unique | Listing 16.2.4.7 |
| Listing 16.2.4.2 | Smoking, Alcohol and Drug Abuse<br>History – Part 2 | Randomized Subjects | Unique | Listing 16.2.4.8 |
| Listing 16.2.5.1 | Atopic Dermatitis and Related<br>Conditions Baseline Prior<br>Medications | Randomized Subjects | Unique | Listing 16.2.4.9.1 |
| Listing 16.2.5.2 | Other Baseline Prior Medications | Randomized Subjects | Repeat | Listing 16.2.9.4 |
| Listing 16.2.6 | Baseline Physical Examination | Randomized Subjects | Unique | Listing 16.2.9.5 |

| | Title | Population | Comment | New<br>Number* |
|---|---|---|---|---|
| Listing 16.3.1 | Active AD mRNA Expression<br>Signature and Pathologic Epidermal<br>Phenotype Measures | Full Analysis Set | Unique | Listing 16.2.6.1 |
| Listing 16.3.2 | IGA Scores | Full Analysis Set | Unique | Listing 16.2.6.2 |
| Listing 16.3.3 | EASI Scores | Randomized Subjects | Unique | Listing 16.2.6.3 |
| Listing 16.3.4.1 | SCORAD Clinical Scores | Full Analysis Set | Unique | Listing 16.2.6.4 |
| Listing<br>16.3.4.4 | Pruritus NRS Clinical Scores | Full Analysis Set | Repeat | Listing 16.2.6.5 |
| Listing 16.3.4.5 | DLQI Clinical Scores | Full Analysis Set | Repeat | Listing 16.2.6.6 |
| Listing 16.3.5 | Transepidermal Water Loss<br>Readings | Full Analysis Set | Unique | Listing 16.2.6.7 |
| Listing 16.3.6 | Anti-Drug Antibodies (ADA) | Safety Analysis Set | Unique | Listing 16.2.6.8 |
| Listing 16.3.8 | Leukocytes Sub-Population Cell<br>Counts | Full Analysis Set | Unique* | Listing<br>16.2.6.9 |
| Listing 16.3.9 | Cellular Infiltrates | Full Analysis Set | Repeat* | Listing 16.2.6.10 |
| Listing 16.3.10 | Serum Total Immunoglobulin E,<br>Serum Soluble OX40, Serum<br>Soluble OX40 and Circulating<br>Eosinophil Counts | Full Analysis Set | Repeat* | Listing 16.2.6.11 |
| Listing 16.3.12 | Prohibited Medications | Full Analysis Set | Unique | Listing 16.2.2.2 |
| Listing 16.4.1.1.1 | Adverse Events – Part 1 | Safety Analysis Set | Unique | Listing 16.2.7.1 |
| Listing 16.4.1.2.1 | Serious Adverse Events – Part 1 | Safety Analysis Set | Repeat | Listing 16.2.7.3 |
| Listing 16.4.1.5.1 | Adverse Events Leading to<br>Discontinuation of Study – Part 1 | Safety Analysis Set | Repeat | Listing 16.2.7.5 |
| Listing 16.4.1.7.1 | Adverse Events Leading to Death – Part 1 | Safety Analysis Set | Repeat | Listing<br>16.2.7.7 |
| Listing 16.4.1.1.2 | Adverse Events – Part 2 | Safety Analysis Set | Unique | Listing 16.2.7.2 |
| Listing | Serious Adverse Events – Part 2 | Safety Analysis Set | Repeat | Listing |

| | Title | Population | Comment | New<br>Number* |
|---|---|---|---|---|
| 16.4.1.2.2 | | | | 16.2.7.4 |
| Listing 16.4.1.5.2 | Adverse Events Leading to Discontinuation of Study – Part 2 | Safety Analysis Set | Repeat | Listing<br>16.2.76 |
| Listing 16.4.1.7.2 | Adverse Events Leading to Death – Part 2 | Safety Analysis Set | Repeat | Listing 16.2.7.8 |
| Listing 16.4.2 | Study Drug Administration | Safety Analysis Set | Unique | Listing 16.2.5.1 |
| Listing 16.4.3.1 | Concomitant Medications | Safety Analysis Set | Unique | Listing 16.2.5.2 |
| Listing 16.4.3.2 | Concomitant Non-Drug Therapies | Safety Analysis Set | Unique | Listing 16.2.5.3 |
| Listing 16.4.3.3 | Rescue Medications | Safety Analysis Set | Repeat | Listing 16.2.5.4 |
| Listing 16.4.4.1.1 | Heamatology Results | Safety Analysis Set | Unique | Listing 16.2.8.1 |
| Listing 16.4.4.1.2 | Subjects with Abnormal<br>Hematology Results | Safety Analysis Set | Repeat | Listing 16.2.8.2 |
| Listing 16.4.4.2.1 | Serum Biochemistry Results | Safety Analysis Set | Repeat | Listing 16.2.8.3 |
| Listing 16.4.4.2.2 | Subjects with Abnormal Serum<br>Biochemistry Results | Safety Analysis Set | Repeat | Listing 16.2.8.4 |
| Listing 16.4.4.3 | Urinalysis Results | Safety Analysis Set | Repeat | Listing 16.2.8.5 |
| Listing 16.4.4.4 | Serology Results | Safety Analysis Set | Repeat | Listing 16.2.8.6 |
| Listing 16.4.4.5 | Other Laboratory Test Results | Safety Analysis Set | Repeat | Listing 16.2.8.7 |
| Listing 16.4.5 | Vital Signs Results | Safety Analysis Set | Unique | Listing 16.2.9.1 |
| Listing 16.4.6 | Brief Physical Examination | Safety Analysis Set | Unique | Listing 16.2.9.2 |
| Listing 16.4.7 | Electrocardiogram (ECG) Results | Safety Analysis Set | Unique | Listing 16.2.9.3 |
| Listing 16.4.8 | Individual GBR830 Serum<br>Concentration (ng/mL) Data | Pharmacokinetic<br>Analysis Set | Unique | Listing 16.2.6.12 |
| Listing 14.4.9 | Individual Pharmacokinetic<br>Parameters of GBR830 | Pharmacokinetic<br>Analysis Set | Unique | Listing 16.2.6.13 |
| Listing<br>16.4.10 | Time Points used to Calculate the GBR830 Elimination Rate Constant (λz) | Pharmacokinetic<br>Analysis Set | Unique | Listing 16.2.6.14 |

| | Title | Population | Comment | New<br>Number* |
|---|---|---|---|---|
| Listing<br>16.4.11 | Reasons Pharmacokinetic<br>Parameters Could Not be<br>Determined | Pharmacokinetic<br>Analysis Set | Unique | Listing 16.2.6.15 |
| Listing 16.5.2 | Protocol Deviations | Randomized Subjects | Unique | Listing 16.2.2.1 |

<sup>\*</sup>New number is used in final displays

## APPENDIX 3. DATA DISPLAY SPECIFICATIONS

Table 14.1.1 Subject Disposition Screened Subjects

| | Statistic | GBR 830<br>(N=xx) | Placebo<br>(N=xx) | Overall (N=xx) |
|---|---|---|---|---|
| Subjects screened | n | | | X |
| Screen failures | n | | | X |
| Re-screened | n | | | X |
| Subjects randomized | n (%) | x (100) | x (100) | x (100) |
| Subjects replaced | n (%) | x (xxx) | x (xxx) | x (xxx) |
| End of study status | | | | |
| Subject completed study | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Subject withdrawn | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Reason for early termination/withdrawal | | | | |
| Withdrawal of consent | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Adverse event | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Investigator's discretion | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Non compliance with study procedures / protocol deviation | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Pregnancy | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Subjects requiring rescue medications or interventions/treatment with another therapeutic agent | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Disease progression/exacerbation | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Subjects randomized in the study who withdraw their consent for the first post-baseline skin biopsies | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Lost to follow up | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Death | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Other | n (%) | x (xxx) | x (xxx) | x (xxx) |

**Footnote:** Percentages are based on the total number of randomized subjects in each treatment group.

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas

Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY


Table 14.1.2 Analysis Sets Randomized Subjects

| | Statistic | GBR 830 | Placebo | Overall |
|---|---|---|---|---|
| | | (N=xx) | (N=xx) | (N=xx) |
| Full Analysis Set (FAS) | | | | |
| No | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Yes | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Biological Activity Set (BAS) | | | | |
| No | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Yes | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Safety Analysis Set (SAF) | | | | |
| No | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Yes | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Pharmacokinetic Analysis Set (PKAS) | | | | |
| No | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Yes | n (%) | x (xxx) | x (xxx) | x (xxx) |

Footnote: Percentages are based on the total number of randomized subjects in each treatment group.

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Analysis Plan: 06Jul2017 Confidential Page X of Y

Table 14.1.3 Study Participation Full Analysis Set

| | Statistic | GBR 830<br>(N=xx) | Placebo<br>(N=xx) | Overall<br>(N=xx) |
|---|---|---|---|---|
| | | (14-AA) | (11-11) | (11-44) |
| Time on study (days) | N | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX |
| | Median | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |
| Number of subjects with any data at each visit | | | | |
| Visit 2 (day 1) | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Visit 3 (day 4) | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Visit 4 (day 8) | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Visit 5 (day 15) | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Visit 6 (day 22) | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Visit 7 (day 29) | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Visit 8 (day 32) | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Visit 9 (day 36) | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Visit 10 (day 43) | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Visit 11 (day 50) | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Visit 12 (day 57) | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Visit 13 (day 71) | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Visit 14/EOS (day 85/Early Termination) | n (%) | x (xxx) | x (xxx) | x (xxx) |

Footnote: Percentages are based on the total number of Full Analysis Set subjects in each treatment group.

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Analysis Plan: 06Jul2017 Confidential Page X of Y

Table 14.2.1.1
Demographic Characteristics
Full Analysis Set

| Parameter | Statistic | GBR 830 | Placebo | Overall |
|---|---|---|---|---|
| | | (N=xx) | (N=xx) | (N=xx) |
| Age at study entry (years) | n | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX |
| | Median | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |
| Age group at study entry | | | | |
| <65 years | n (%) | x (xxx) | x (xxx) | x (xxx) |
| ≥65 years | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Sex | | | | |
| Female | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Male | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Race | | | | |
| Asian | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Black | n (%) | x (xxx) | x (xxx) | x (xxx) |
| White | n (%) | x (xxx) | x (xxx) | x (xxx) |
| American Indian or Alaska Native | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Native Hawaiian or Other Pacific Islander | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Other | n (%) | x (xxx) | x (xxx) | x (xxx) |

Footnote: Percentages are based on the total number of Full Analysis Set subjects in each treatment group.

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas

Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY


Page X of Y

Table 14.2.1.1
Demographic Characteristics
Full Analysis Set

Cont.

| Parameter | Statistic | GBR 830 | Placebo | Overall |
|--------------------------|-----------|---------|---------|---------|
| | | (N=xx) | (N=xx) | (N=xx) |
| Ethnicity | | | | |
| Hispanic or Latino | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Not Hispanic or Latino | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Not Inspance of Latino | II (70) | X (XXX) | A (AAA) | A (AAA) |
| Weight (kg) | n | XX | XX | XX |
| | Mean | XX.X | XX,X | XX.X |
| | SD | XX.XX | XX,XX | XX.XX |
| | Median | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |
| Height (cm) | n | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X |
| | SD | XX,XX | XX.XX | XX.XX |
| | Median | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |
| BMI (kg/m <sup>2</sup> ) | n | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX |
| | Median | XX.X | XX,X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |

Footnote: Percentages are based on the total number of Full Analysis Set subjects in each treatment group.

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXX.sas
Date/time of run: DDMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Page X of Y

Table 14.2.1.1
Demographic Characteristics
Full Analysis Set

Cont.

| Parameter | Statistic | GBR 830<br>(N=xx) | Placebo (N=xx) | Overall (N=xx) |
|---|---|---|---|---|
| Body surface area (m <sup>2</sup> ) | n | VV | VV | VV |
| Jody Surface area (III ) | n<br>Mean | XX | XX | XX |
| | | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX |
| | Median | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |
| Country | | | | |
| USA | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Canada | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Child bearing potential (female only) | N* | XXX | XXX | XXX |
| No | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Post menopausal | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Duration of non child bearing potential $\leq 1$ year | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Duration of non child bearing potential > 1 year | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Permanently sterilized | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Duration of non child bearing potential $\leq 1$ year | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Duration of non child bearing potential > 1 year | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Yes | n (%) | x (xxx) | x (xxx) | x (xxx) |

Footnote: Percentages are based on the total number of Full Analysis Set subjects in each treatment group.  $N^*$  is the number of female subjects. Percentages of child bearing potential are based on  $N^*$ .

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY
Analysis Plan: 06Jul2017 Confiden

nalysis Plan: 06Jul2017 Confidential Page X of Y

Repeat for:

Table 14.2.1.2

Demographic Characteristics

Biological Activity Set

Table 14.2.1.3
Demographic Characteristics
Pharmacokinetic Analysis Set

Table 14.2.2 Atopic Dermatitis (AD) History Full Analysis Set

| Parameter | Statistic | GBR 830 | Placebo | Overall |
|-----------------------------------|-----------|---------|---------|---------|
| | | (N=xx) | (N=xx) | (N=xx) |
| V AD I' ( ) | | | | |
| Years since AD diagnosis (years) | n | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX |
| | Median | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |
| Years since AD diagnosis category | | | | |
| <2 Years | n (%) | x (xxx) | x (xxx) | x (xxx) |
| 2 – 5 Years | n (%) | x (xxx) | x (xxx) | x (xxx) |
| >5 Years | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Age at AD diagnosis (years) | n | XX | XX | XX |
| 8 | Mean | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX |
| | Median | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |
| Гуре of AD | THUM. | AA | nn. | AA |
| Intrinsic | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Extrinsic | n (%) | x (xxx) | x (xxx) | x (xxx) |
| 2 | 11 (70) | () | () | () |
| Any history of allergy? | | | | |
| Yes | n (%) | x (xxx) | x (xxx) | x (xxx) |
| No | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Was patch test performed? | | | | |
| Yes | n (%) | x (xxx) | x (xxx) | x (xxx) |
| No | n (%) | x (xxx) | x (xxx) | x (xxx) |

Footnote: Percentages are based on the total number of Full Analysis Set subjects in each treatment group.

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Page X of Y

Table 14.2.2 Atopic Dermatitis (AD) History Full Analysis Set

Cont.

| Parameter | Statistic | GBR 830 | Placebo | Overall |
|---|---|---|---|---|
| | | (N=xx) | (N=xx) | (N=xx) |
| Any other concomitant atopic illness? | | | | |
| Yes | n (0/) | v (vvv) | v (vvv) | v (vvv) |
| | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Asthma | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Allergic rhinitis | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Skin conditions | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Other | n (%) | x (xxx) | x (xxx) | x (xxx) |
| No | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Was skin biopsy performed in past? | | | | |
| Yes | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Eosinophilic | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Non-Eosinophilic | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Other | n (%) | x (xxx) | x (xxx) | x (xxx) |
| No | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Any treatment administered for AD or associated condition? | | | | |
| Yes | n (%) | x (xxx) | x (xxx) | x (xxx) |
| No | n (%) | x (xxx) | x (xxx) | x (xxx) |

Footnote: Percentages are based on the total number of Full Analysis Set subjects in each treatment group.

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXX.sas
Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Page X of Y

Table 14.2.3 Medical/Surgical History Full Analysis Set

| Parameter | Statistic | GBR 830<br>(N=xx) | Placebo<br>(N=xx) | Overall (N=xx) |
|---|---|---|---|---|
| HEENT | | | | |
| Preferred term 1 | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Preferred term 2 | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Preferred term 3 | n (%) | x (xxx) | x (xxx) | x (xxx) |

Footnote: Percentages are based on the total number of Full Analysis Set subjects in each treatment group. Preferred terms are sorted in descending order by the overall column.

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas

Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY


Page X of Y

Programming notes: Also include the following body systems Cardiovascular System, Respiratory System, Musculoskeletal System, Dermatological System, Skin and its appendages, Lymphatic System, Gastrointestinal System, Genitourinary System, Nervous System, Endocrine System, Immunological System, Allergic Conditions, Other.

Table 14.2.4 Smoking, Alcohol and Drug Abuse History Full Analysis Set

| Parameter | Statistic | GBR 830 | Placebo | Overall |
|---|---|---|---|---|
| | | (N=xx) | (N=xx) | (N=xx) |
| Former or current alcohol user | | | | |
| N/A | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Former | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Current | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Alcohol consumption (ml/week) | n | XX | XX | xx |
| | Mean | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX |
| | Median | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |
| History or alcohol abuse? | | | | |
| No | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Yes | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Former or current drug user | | | | |
| N/A | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Former | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Current | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Is drug use clinically significant in the opinion of the Investigato meets DSM-V criteria for addiction or abuse? | r or | | | |
| No | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Yes | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Former or current smoker | | | | |
| N/A | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Former | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Current | n (%) | x (xxx) | x (xxx) | x (xxx) |

**Footnote:** Percentages are based on the total number of Full Analysis Set subjects in each treatment group.

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas

Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY


#### Table 14.2.4 Smoking, Alcohol and Drug Abuse History Full Analysis Set

Cont.

| Parameter | Statistic | GBR 830<br>(N=xx) | Placebo<br>(N=xx) | Overall<br>(N=xx) |
|---|---|---|---|---|
| Cigarettes per day | n | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX |
| | Median | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |
| Former or current smokeless tobacco user | | | | |
| N/A | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Former | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Current | n (%) | x (xxx) | x (xxx) | x (xxx) |

**Footnote:** 1.Percentages are based on the total number of Full Analysis Set subjects in each treatment group.

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Analysis Plan: 06Jul2017 Confidential Page X of Y
Table 14.2.5.1
Atopic Dermatitis and Related Conditions Baseline Prior Medications
Full Analysis Set

| ATC Level 1 | Statistic | GBR 830 | Placebo | Overall |
|---|---|---|---|---|
| ATC Level 2 | | (N=xx) | (N=xx) | (N=xx) |
| ATC Level 3 | | | | |
| ATC Level 4 | | | | |
| Preferred Term | | | | |
| ATC Level 1 ATC Level 2 ATC Level 3 ATC Level 4 Preferred term 1 Preferred term 2 Preferred term 3 | n (%)<br>n (%)<br>n (%) | x (xxx)<br>x (xxx)<br>x (xxx) | x (xxx)<br>x (xxx)<br>x (xxx) | x (xxx)<br>x (xxx)<br>x (xxx) |
| Etc | | | | |

Footnote: Percentages are based on the total number of Full Analysis Set subjects in each treatment group. Preferred terms within the ATC Code are sorted in descending order by the overall column.

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Page X of Y

Repeat for:

6-Jul-17

Table 14.2.5.2 Other Baseline Prior Medications Full Analysis Set

Table 14.2.10 Baseline Clinical Scores Full Analysis Set

| Parameter | Statistic | GBR 830 | Placebo | Overall |
|---|---|---|---|---|
| | | (N=xx) | (N=xx) | (N=xx) |
| Engage Anna and Consuits Index (EACI) | | | | |
| Eczema Area and Severity Index (EASI) | n<br>Maar | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX |
| | Median | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |
| Investigator's Global Assessment (IGA) | | | | |
| Severe | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Moderate | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Mild | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Almost clear | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Clear | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Not done | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Scoring of Atopic Dermatitis (SCORAD) | n | XX | XX | xx |
| | Mean | XX.X | XX.X | XX.X |
| | SD | XX,XX | XX.XX | XX.XX |
| | Median | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |
| Dermatology Life Quality Index (DLQI) | n | XX | XX | xx |
| | Mean | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX |
| | Median | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |

Footnote: Percentages are based on the total number of Full Analysis Set subjects in each treatment group.

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas

Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY


#### Table 14.2.10 Baseline Clinical Scores Full Analysis Set

cont.

| Parameter | Statistic | GBR 830<br>(N=xx) | Placebo<br>(N=xx) | Overall (N=xx) |
|---|---|---|---|---|
| Pruritis Numerical Rating Scale (NRS) | n | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX |
| | Median | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |

Footnote: Percentages are based on the total number of Full Analysis Set subjects in each treatment group.

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas Date/time of run: DDMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Analysis Plan: 06Jul2017 Confidential Page X of Y

Repeat for:

#### **Table 14.2.11.1**

# Baseline Active AD mRNA Expression Signatures Obtained from Skin Biopsies (Non Lesion Samples) Biological Activity Set

Programming notes 1) Present baseline visit only, Repeat for all biomarkers

#### **Table 14.2.11.2**

Baseline Pathologic Epidermal Phenotype Measures Obtained from Skin Biopsies (Non Lesion Samples)
Biological Activity Set

Programming notes 1) Present baseline visit only, Repeat for all phenotypes

Table 14.3.1.1.a

MMRM Analysis Selected Active AD mRNA Expressions (Normalized to hARP) Obtained from Skin Biopsies (Lesion Samples)- Primary Analysis
Biological Activity Set

| Biomarke | er: CCL18/hARP | | |
|---|---|---|---|
| Cont. | | | |
| | | GBR 830<br>(N=xx) | Placebo<br>(N=xx) |
| | Geometric LS mean of P/B ratio [2] (95% CI) | xx.x (xx.xx, xx.xx) | xx.x (xx.xx, xx.xx) |
| | Ratio GBR830/placebo [3]: Adjusted LS mean treatment difference (95% CI) | xx.x (xx.xx, xx.xx) | |
| | p-value | X.XXX | |

#### Footnote:

- [1] Geometric mean is exponentially back-transformed from the least squares (LS) mean based on a mixed model. It is presented on the original scale. The same transformation is applied in order to obtain the 95% CI.
- [2] Mixed model with treatment group and planned visit as fixed effects, log transformed baseline value as covariate, and with treatment by visit interaction and unstructured covariance structure. Using log transformed mRNA values.

Ratio: P/B = Post-baseline / Baseline; CI = Confidence interval.

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXXX.sas Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Programming notes: repeat table for all the log transformed biomarkersnormalized to hARP in the SAP text CCL11/hARP, CCL17/hARP, CCL18/hARP, CCL26/hARP, CXCL10/hARP, FOXP3/hARP, IFNg/hARP, IL23p40/hARP, IL13/hARP, IL13/hARP, IL13/hARP, IL22/hARP, IL23p19/hARP, K16/hARP, MMP12/hARP, OX40L/hARP, S100A12/hARP, S100A9/hARP, TSLPR/hARP

Analysis Plan: 06Jul2017 Confidential Page X of Y

Table 14.3.1.1.b

Change from Baseline in the Selected Active AD mRNA Expression Signatures (Normalized to hARP) Obtained from Skin Biopsies by Lesion Location –Primary Analysis

Biological Activity Set

Biomarker: CCL18/hARP

| | Statistic | GBR 830<br>(N=xx) | Placebo<br>(N=xx) |
|---|---|---|---|
| Baseline (day 1) | N | XX | XX |
| Baseline (day 1) | Mean | XX.X | XX.X |
| | SD | XX.XX | XX,XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |
| | Geometric mean (%CV) [1] | xx.x (xx.xx) | xx.x (xx.xx) |
| Visit 7 (day 29) | N | XX | XX |
| · | Mean | XX.X | XX.X |
| | SD | XX.XX | XX.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |
| | Geometric mean (%CV) [1] | xx.x (xx.xx) | xx.x (xx.xx) |
| Change from Baseline to Visit 7 (day 29) | N | XX | xx |
| - | Mean | XX.X | XX.X |
| | SD | XX.XX | XX.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |
| (repeat for Visit 13 (day 71)) | Geometric mean (%CV) [1] | xx.x (xx.xx) | xx.x (xx.xx) |

<sup>[1]</sup> The geometric mean is presented on the original non transformed scale. All other statistics are presented on the log scale unless otherwise stated.

Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Programming notes: the summary (n, mean, SD, median, min, max) will be on the normalize gene without log transformation, repeat table for all mRNA normalized to hARP parameters in the SAP text and produce for lesion and non-lesion samples (if available)

Analysis Plan: 06Jul2017 Confidential Page X of Y

Table 14.3.1.2 Change from Baseline in H&E Thickness Obtained from Skin Biopsies by Lesion Location – Primary Analysis Biological Activity Set

Location: Lesion

| | Statistic | GBR 830<br>(N=xx) | Placebo<br>(N=xx) |
|---|---|---|---|
| | | (1, 1111) | (1, 121) |
| Baseline (day 1) | n | XX | XX |
| | Mean | XX.X | XX.X |
| | SD | XX.XX | XX.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |
| Visit 7 (day 29) | n | XX | XX |
| | Mean | XX.X | XX.X |
| | SD | XX.XX | XX.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |
| Change from Baseline to Visit 7 (day 29) | n | XX | XX |
| | Mean | XX.X | XX.X |
| | SD | XX.XX | XX.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXX.sas

Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY


Page X of Y

Programming notes 1) Repeat for appropriate non lesion.

Table 14.3.1.3
Summary of K16 Obtained from Skin Biopsies by Lesion Location and Visit – Primary Analysis Biological Activity Set

Location: Lesion

| | | Statistic | GBR 830<br>(N=xx) | Placebo<br>(N=xx) |
|---|---|---|---|---|
| Baseline (day 1) | Slight | n (%) | xx | xx |
| | Good | n (%) | xx | xx |
| | Excellent | n (%) | xx | xx |
| Visit 7 (day 29) | Worsening | n (%) | xx | XX |
| | No change | n (%) | xx | XX |
| Visit 13 (day 71) | Worsening | n (%) | xx | XX |
| | No change | n (%) | xx | XX |

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas

Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY


Page X of Y

Programming notes 1) Repeat for appropriate non lesion.

**Table 14.3.1.4** Summary of Histological Response Obtained from Skin Biopsies by Lesion Location and Visit - Primary Analysis **Biological Activity Set** 

Location: Lesion

| | | Statistic | GBR 830<br>(N=xx) | Placebo<br>(N=xx) |
|---|---|---|---|---|
| Baseline (day 1) | Responder | n (%) | XX | XX |
| | Non responder | n (%) | XX | XX |
| Visit 7 (day 29) | Responder | n (%) | XX | XX |
| | Non responder | n (%) | XX | XX |
| √isit 13 (day 71) | Responder | n (%) | xx | xx |
| | Non responder | n (%) | xx | xx |

Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY Analysis Plan: 06Jul2017 Confidential

Programming notes 1) Repeat for appropriate non lesion.

Table 14.2.1.5 Summary of IHC Panel from Skin Biopsies by Visit – Primary Analysis Biological Activity Set

Parameter: CD3 Epidermis # of Cells per 1.2m

| | Statistic | GBR 830<br>(N=xx) | Placebo (N=xx) |
|---|---|---|---|
| Baseline (day 1) | n | XX | XX |
| | Mean | XX.X | XX.X |
| | SD | XX.XX | XX.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |
| | Geometric mean (%CV) [1] | xx.x (xx.xx) | xx.x (xx.xx) |
| Visit 7 (day 29) | n | XX | XX |
| | Mean | XX.X | XX.X |
| | SD | XX.XX | XX.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |
| | Geometric mean (%CV) [1] | xx.x (xx.xx) | xx.x (xx.xx) |
| Change from Pagaline to Vigit 7 (day 20) | _ | | **** |
| Change from Baseline to Visit 7 (day 29) | n<br>Maria | XX | XX |
| | Mean<br>SD | XX.X | XX.X |
| | | XX.XX | XX.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | Xx |
| | Max. | XX | XX |
| | Geometric mean (%CV) [1] | xx.x(xx.xx) | xx.x (xx.xx) |

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas Date/time of run: DDMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Programming notes 1) Repeat for appropriate non lesion.Parameters summarized will include: CD3.EPIDERMIS # of Cells per 1.2mm2, CD3.DERMIS # of Cells per 1.2mm2, Ki67.EPIDERMIS # of Cells per 1.2mm2, Ki67.DERMIS # of Cells per 1.2mm2, FcEpsilonRI.DERMIS # of Cells per 1.2mm2, FcEpsilonRI.EPIDERMIS # of Cells per 1.2mm2, OX40.EPIDERMIS # of Cells per 1.2mm2, OX40L.EPIDERMIS # of Cells per 1.2mm2, OX40L.DERMIS # of Cells per 1.2mm2, MBP.EPIDERMIS # of Cells per 1.2mm2, MBP.DERMIS # of Cells per 1.2mm2

tistical Analysis Plan – Protocol GBR 830-201 6-Jul-17

Analysis Plan: 06Jul2017 Confidential Page X of Y

Table 14.3.2
Proportion of Subjects who Achieved an IGA Score of 0 or 1 by Visit
Full Analysis Set

| Visit | Category | Statistic | GBR 830<br>(N=xx) | Placebo<br>(N=xx) |
|---|---|---|---|---|
| Visit 3 (day 4) | IGA score 0 or 1 | n/N* (%) | x/x (xxx) | x/x (xxx) |
| | IGA score 2+ | n/N* (%) | x/x (xxx) | x/x (xxx) |
| Visit 4 (day 8) | IGA score 0 or 1 | n/N* (%) | x/x (xxx) | x/x (xxx) |
| | IGA score 2+ | n/N* (%) | x/x (xxx) | x/x (xxx) |
| etc. | IGA score 0 or 1 | n/N* (%) | x/x (xxx) | x/x (xxx) |
| Visit 14 (day 85) | IGA score 2+ | n/N* (%) | x/x (xxx) | x/x (xxx) |
| Visit 12 LOCF | IGA score 0 or 1<br>IGA score 2+ | n/N* (%)<br>n/N* (%)<br>Cochran-Mantel-Haenzsel statistic<br>p-value | x/x (xxx)<br>x/x (xxx)<br>xx.xx<br>x.xxx | x/x (xxx)<br>x/x (xxx) |
| Visit 14 LOCF | IGA score 0 or 1<br>IGA score 2+ | n/N* (%)<br>n/N* (%)<br>Cochran-Mantel-Haenzsel statistic<br>p-value | x/x (xxx)<br>x/x (xxx)<br>xx.xx<br>x.xxx | x/x (xxx)<br>x/x (xxx) |

**Footnote:** The Cochran-Mantel-Haenszel test has been stratified by categorical baseline IGA score of (less than 4; or greater or equal to 4). Visit 12/14 LOCF was calculated as the last post baseline measurement prior to or on Visit 12/14. N is the number of subjects in the analysis set; n is the number of subjects meeting the criteria; N\* is the total subjects with IGA measurement; percentages of IGA scores at each visit are calculated using n divided by N\* in each treatment group.

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas Date/time of run: DDMMYYYY HH:MM; Date of data extraction: DDMMYYYY

6-Jul-17

Page X of Y

Analysis Plan: 06Jul2017 Confidential Page X of Y

Programming note: 1) Repeat for visits indicated in the SAP text.

Table 14.3.3.1 Proportion of Subjects who Achieved an EASI 50 Response by Visit Full Analysis Set

| Visit | Parameter | Statistic | GBR 830<br>(N=xx) | Placebo<br>(N=xx) |
|---|---|---|---|---|
| Visit 3 (day 4) | EASI 50 responder | n/N* (%) | x/x (xxx) | x/x (xxx) |
| | EASI 50 non-responder | n/N* (%) | x/x (xxx) | x/x (xxx) |
| Visit 4 (day 8) etc | | | | |
| Visit 12 LOCF | EASI 50 responder | n/N* (%) | x/x (xxx) | x/x (xxx) |
| | EASI 50 non-responder | n/N* (%) | x/x (xxx) | x/x (xxx) |
| Visit 14 LOCF | EASI 50 responder | n/N* (%) | x/x (xxx) | x/x (xxx) |
| | EASI 50 non-responder | n/N* (%) | x/x (xxx) | x/x (xxx) |

**Footnote:** N is the number of subjects in the analysis set; n is the number of subjects meeting the criteria; N\* is the total subjects with EASI measurement; Visit 12/14 LOCF was calculated as the last post baseline measurement prior to or on Visit 12/14. Percentages of EASI 50 responders and non-responders at each visit are calculated using n divided by N\* in each treatment group.

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas

Date/time of run: DDMMYYYY HH:MM; Date of data extraction: DDMMYYYY


Confidential

Programming note: 1) Repeat for visits indicated in the SAP text.

Glenmark Pharmaceutical SA Statistical Analysis Plan – Protocol GBR 830-201

6-Jul-17

Repeat for:

Table 14.3.3.2 Proportion of Subjects who Achieved an EASI 75 Response by Visit Full Analysis Set

Table 14.3.3.3 Analysis of Covariance (ANCOVA) of change from baseline in EASI Score to Visit 12 LOCF Full Analysis Set

| Parameter | Statistic | GBR 830 | Placebo |
|---|---|---|---|
| | | (N=xx) | (N=xx) |
| Baseline (day 1) | n | XX | XX |
| Dascinic (day 1) | Mean | XX.X | XX.X |
| | SD | XX.XX | XX.XX |
| | Median | XX.XX<br>XX.X | XX.XX<br>XX.X |
| | Min. | | |
| | Max. | XX | XX |
| | Max. | XX | XX |
| Visit 12 LOCF | n | XX | xx |
| | Mean | XX.X | XX.X |
| | SD | XX.XX | XX.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | xx | XX |
| Adjusted LS mean [SE] (95% CI) | | xx.x [xx.xx] | xx.x [xx.xx] |
| Adjusted LS mean [SE] (93% CI) | | (xx.xx, xx.xx) | (xx.xx, xx.xx |
| | | (11.11, 11.11) | (АА.АА, АА.АА |
| Treatment difference vs. placebo [1]: | | xx.x [xx.xx] | |
| Adjusted LS mean treatment difference [SE] (95% CI) | | (xx.xx, xx.xx) | |
| p-value | | X.XXX | |

[1] ANCOVA model with treatment group as fixed effect and baseline EASI scoreas covariate. SE: Standard Error. CI: Confidence interval. LS: Least squares.

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Page X of Y

Table 14.3.4.1
Percent Change from Baseline in EASI Clinical Score at Each Visit
Full Analysis Set

| Parameter | Statistic | GBR 830 | Placebo |
|---|---|---|---|
| | | (N=xx) | (N=xx) |
| Baseline (day 1) | n | XX | XX |
| Buseline (day 1) | Mean | XX.X | XX.X |
| | SD | XX.XX | XX.XX |
| | Median | XX.X | XX.XX |
| | Min. | XX | XX |
| | Max. | XX | XX |
| Visit 3 (day 4) | n | XX | XX |
| | Mean | XX.X | XX.X |
| | SD | XX.XX | XX.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |
| Percent change from Baseline to Visit 3 (day 4) | n | XX | XX |
| recent change from Basenne to Visit 3 (day 4) | Mean | XX.X | XX.X |
| | SD | XX.XX | XX.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| etc. | Max. | XX | XX |
| Visit 14 LOCF [1] | n | XX | XX |
| | Mean | XX.X | XX.X |
| | SD | XX.XX | XX.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |
| Percent change from Baseline to Visit 14 LOCF [1] | n | XX | XX |
| 2 street change hom baseline to visit 1 i boot [1] | Mean | XX.X | XX.X |
| | SD | XX.XX | XX.XX |
| | Median | XX.XX | XX.XX |
| | Min. | XX | XX |
| | Max. | XX | Xx |

Footnote: [1] Visit 12/14 LOCF was calculated as the last post baseline measurement prior to or on Visit 12/14.

### Glenmark Pharmaceutical SA Statistical Analysis Plan – Protocol GBR 830-201

6-Jul-17

SOURCE: X:\Numerus\Studies\XXX\XXYYY\Analysis\Prod\Progs\XXXXX.sas

Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY


Page X of Y

Programming note: 1) Repeat for visits indicated in the SAP text.

Repeat for

Table 14.3.4.2

Percent change from Baseline in SCORAD Clinical Score at Each Visit
Full Analysis Set

Table 14.3.2.2
Percent Change from Baseline in IGA Clinical Score at Each Visit
Full Analysis Set

Table 14.3.4.4

Percent change from Baseline in Pruritus NRS Clinical Score at Each Visit
Full Analysis Set

Table 14.3.4.5

Percent change from Baseline in DLQI Clinical Score at Each Visit
Full Analysis Set

 $Table\ 14.3.5$  Changes from Baseline in Transepidermal Water Loss (g/m²/h) by Lesion/Non-Lesion Area Full Analysis Set

| ntistic | GBR 830 | Placebo |
|---------|-----------------------------|------------------------|
| | (N=xx) | (N=xx) |
| | XX | xx |
| an | XX.X | XX.X |
| *** | XX.XX | XX.XX |
| dian | XX.X | XX.X |
| 1. | XX | XX |
| х. | XX | XX |
| | XX | XX |
| an | XX.X | XX.X |
| | XX.XX | XX.XX |
| dian | XX.X | XX.X |
| 1. | XX | XX |
| х. | XX | XX |
| | XX | XX |
| an | XX.X | XX.X |
| | XX.XX | XX.XX |
| | | XX.X |
| | | XX |
| | XX | XX |
| Iin | D<br>Iedian<br>Iin.<br>Iax. | fedian xx.x<br>fin. xx |

**Footnote:** Visit 12/14 LOCF was calculated as the last post baseline measurement prior to or on Visit 12/14.

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas

Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY


Page X of Y

Programming note: 1) Repeat for visits indicated in the SAP text.

Table 14.3.6 Anti-Drug Antibodies to GBR 830 by Visit Full Analysis Set

| Visit Result | | Statistic | GBR 830 | Placebo |
|------------------|----------|-----------|---------|---------|
| | | | (N=xx) | (N=xx) |
| Baseline (day 1) | Positive | n (%) | x (xxx) | x (xxx) |
| | Negative | n (%) | x (xxx) | x (xxx) |
| | Not done | n (%) | x (xxx) | x (xxx) |
| Visit 3 (day 4) | Positive | n (%) | x (xxx) | x (xxx) |
| | Negative | n (%) | x (xxx) | x (xxx) |
| | Not done | n (%) | x (xxx) | x (xxx) |
| etc. | | | | |
| Overall [1] | Positive | n (%) | x (xxx) | x (xxx) |
| | Negative | n (%) | x (xxx) | x (xxx) |
| | Not done | n (%) | x (xxx) | x (xxx) |

#### Footnote:

[1] If any result is positive then a subject will be counted as positive, else if any result is negative (and no result is positive) then a subject will counted as negative, else a subject will be counted as not done.

Percentages of Positive, Negative and Not Done at each visit are based on the total number of Full Analysis Set subjects in each treatment group.

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas

Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY


Page X of Y

Programming note: 1) Repeat for visits indicated in the SAP text.

Table 14.3.8 Changes from Baseline in Leukocytes Sub-Population Cell Counts Full Analysis Set

| Parameter | Statistic | GBR 830 | Placebo |
|-----------------------------------------|-----------|------------|---------|
| Visit | | (N=xx) | (N=xx) |
| Total T | | | |
| Baseline (day 1) | n | XX | XX |
| | Mean | XX.X | XX.X |
| | SD | XX.XX | XX.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |
| Visit 4 (day 8) | n | XX | XX |
| VISIL 4 (day 8) | Mean | XX.X | XX.X |
| | SD | XX.XX | XX.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |
| Change from Baseline to Visit 4 (day 8) | n | XX | Xx |
| Change from Baseline to Visit 4 (day 6) | Mean | XX.X | XX.X |
| | SD | XX.XX | XX.XX |
| | Median | XX.X | XX.XX |
| | Min. | XX.X<br>XX | XX |
| | Max. | XX | Xx |

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas

Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY


Page X of Y

Programming note: Repeat for relevant Parameters and visits.

Repeat for (where appropriate):

#### Table 14.3.9 Changes from Baseline in Cellular Infiltrates Full Analysis Set

**Table 14.3.10** 

Changes from Baseline in Serum Total Immunoglobulin E, Serum Soluble OX40, Serum Soluble OX40 and Circulating Eosinophil Counts
Full Analysis Set

Table 14.3.12 Prohibited Medications Full Analysis Set

| Parameter | Statistic | GBR 830 | Placebo |
|----------------------------------------------|-----------|---------|---------|
| | | (N=xx) | (N=xx) |
| Study day of first prohibited medication [1] | n | VV | VV |
| Study day of first promoticed medication [1] | n<br>Mean | XX | XX |
| | SD | XX.X | XX.X |
| | | XX.XX | XX.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |
| Number of subjects excluded | | | |
| Visit 2 | n (%) | x (xxx) | x (xxx) |
| Visit 3 | n (%) | x (xxx) | x (xxx) |
| Visit 4 | n (%) | x (xxx) | x (xxx) |
| Visit 5 | n (%) | x (xxx) | x (xxx) |
| Visit 6 | n (%) | x (xxx) | x (xxx) |
| Visit 7 | n (%) | x (xxx) | x (xxx) |
| Visit 8 | n (%) | x (xxx) | x (xxx) |
| Visit 9 | n (%) | x (xxx) | x (xxx) |
| Visit 10 | n (%) | x (xxx) | x (xxx) |
| Visit 11 | n (%) | x (xxx) | x (xxx) |
| Visit 12 | n (%) | x (xxx) | x (xxx) |
| Visit 13 | n (%) | x (xxx) | x (xxx) |
| Visit 14 | n (%) | x (xxx) | x (xxx) |

Footnote: [1] Includes only prohibited medication started on or after the first dose of study drug.

Percentages are based on the total number of Full Analysis Set subjects in each treatment group. All visits on and after the first use of prohibited medication will be excluded.

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY


Page X of Y

Table 14.4.1 Overall Treatment Emergent Adverse Events Safety Analysis Set

| | Statistic | GBR 830 | Placebo | Overall |
|---|---|---|---|---|
| | | $(N=xx) \qquad \qquad (N=xx)$ | (N=xx) | (N=xx) |
| Number of subjects experiencing at least one treatment emergent event | | | | |
| AE | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Serious AE | n (%) | x (xxx) | x (xxx) | x (xxx) |
| AE leading to permanent withdrawal of study treatment | n (%) | x (xxx) | x (xxx) | x (xxx) |
| AE leading to withdrawal from study | n (%) | x (xxx) | x (xxx) | x (xxx) |
| AE related to investigational product | n (%) | x (xxx) | x (xxx) | x (xxx) |
| AE leading to death | n (%) | x (xxx) | x (xxx) | x (xxx) |

Footnote: Percentages are based on the total number of Safety Analysis Set subjects in each treatment group. Subjects are counted only once per reason. Only events beginning or worsening after the first dose of study drug are included in this output.

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXXX.sas Date/time of run: DDMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Analysis Plan: 06Jul2017 Confidential Page X of Y

Table 14.4.2.1 Treatment Emergent Adverse Events Safety Analysis Set

| System Organ Class<br>Preferred Term | Statistic | GBR 830<br>(N=xx) | Placebo<br>(N=xx) | Overall (N=xx) |
|---|---|---|---|---|
| Number of subjects with any treatment emergent AE | n (%) | x (xxx) | x (xxx) | x (xxx) |
| System Organ Class 1 | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Preferred Term 1 | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Preferred Term 2 | n (%) | x (xxx) | x (xxx) | x (xxx) |
| System Organ Class 2 | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Preferred Term 1 | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Preferred Term 2 | n (%) | x (xxx) | x (xxx) | x (xxx) |

Footnote: At each level of summarization a subject is counted once if the subject reported one or more events in a given level of summarization.

Percentages are based on the total number of Safety Analysis Set subjects in each treatment group. Preferred terms within the organ classes are sorted in descending order by the overall column. Only events beginning or worsening after the first dose of study drug are included in the summaries. Adverse event terms are coded using MedDRA version 19.0.

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas

Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY


Page X of Y

Repeat for:

Table 14.4.2.2 Serious Treatment Emergent Adverse Events Safety Analysis Set

Table 14.4.2.5
Treatment Emergent Adverse Events Leading to Discontinuation of Study
Safety Analysis Set

6-Jul-17

# Table 14.4.2.6 Treatment Emergent Adverse Events Related to the Investigational Product Safety Analysis Set

Table 14.4.2.7
Treatment Emergent Adverse Events Leading to Death
Safety Analysis Set

Table 14.4.2.8 Treatment Emergent Adverse Events by Severity Safety Analysis Set

| Severity<br>System Organ Class<br>Preferred Term | Statistic | GBR 830<br>(N=xx) | Placebo<br>(N=xx) | Overall<br>(N=xx) |
|---|---|---|---|---|
| Number of subjects with any treatment emergent AE | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Severe | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Moderate | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Mild | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Severe | | | | |
| System Organ Class 1 | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Preferred Term 1 | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Preferred Term 2 | n (%) | x (xxx) | x (xxx) | x (xxx) |
| System Organ Class 2 | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Preferred Term 1 | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Preferred Term 2 | n (%) | x (xxx) | x (xxx) | x (xxx) |

**Footnote**: At each level of summarization a subject is counted once if the subject reported one or more events in a given level of summarization. Subjects with multiple severities will be counted under their most severe category. If severity is missing subject will be considered in the severe category. Preferred terms within the organ classes under severity level are sorted in descending order by the overall column. Only events beginning or worsening after the first dose of study drug are included in the summaries.

Percentages are based on the total number of Safety Analysis Set subjects in each treatment group. Adverse event terms are coded using MedDRA version 19.0.

SOURCE: X:\Numerus\Studies\XXX\XXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Page X of Y

Table 14.4.3 Study Drug Treatment Compliance Safety Analysis Set

| Parameter | Statistic | GBR 830<br>(N=xx) | Placebo<br>(N=xx) | Overall (N=xx) |
|---|---|---|---|---|
| Total % compliance to study treatment [1] | n | XX | XX | XX |
| Total /o compitation to study treatment [1] | Mean | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX |
| | Median | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |
| Number of subjects above 80% compliance | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Visit 2 | | | | |
| Number of subjects who completed 1 hour infusion of study drug | n (%) | x (xxx) | x (xxx) | x (xxx) |
| % compliance to study drug | n | XX | XX | XX |
| , , , | Mean | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX |
| | Median | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX |
| | Max. | XX | XX | XX |
| Visit 7 | | | | |

**Footnote**: [1] Total compliance is calculated as: (Visit 2 actual volume administered + Visit 7 actual volume administered) / (Visit 2 planned volume to be administered + Visit 7 planned volume to be administered) x 100. Percentages are based on the total number of subjects in Safety Analysis Set in each treatment group.

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Page X of Y

Table 14.4.4.1 Concomitant Medications for Atopic Dermatitis and Related Conditions Safety Analysis Set

| ATC Level 1 | Statistic | GBR 830 | Placebo | Overall |
|---|---|---|---|---|
| ATC Level 2 | | (N=xx) | (N=xx) | (N=xx) |
| ATC Level 3 | | | | |
| ATC Level 4 | | | | |
| Preferred Term | | | | |
| ATC Level 1 ATC Level 2 ATC Level 3 ATC Level 4 Preferred term 1 Preferred term 2 Preferred term 3 | n (%)<br>n (%)<br>n (%) | x (xxx)<br>x (xxx)<br>x (xxx) | x (xxx)<br>x (xxx)<br>x (xxx) | x (xxx)<br>x (xxx)<br>x (xxx) |
| Etc | | | | |

**Footnote**: Percentages are based on the total number of subjects in Safety Analysis Set in each treatment group. Preferred terms within the ATC level are sorted in descending order by the overall column Medications were coded using WHO DDE (Sep 2015).

SOURCE: X:\Numerus\Studies\XXX\XXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Page X of Y

Repeat for:

Table 14.4.4.2 Concomitant Non-Drug Treatments Safety Analysis Set

## Glenmark Pharmaceutical SA Statistical Analysis Plan – Protocol GBR 830-201

6-Jul-17

Table 14.4.4.3 Rescue Medications Safety Analysis Set

Programming note: concomitant rescue meds only will be summarized.

Table 14.4.5.1 Change from Baseline in Laboratory Results by Category, Parameter and Visit Safety Analysis Set

**Laboratory Category: Haematology** 

| Parameter<br>Visit | Statistic | GBR 830<br>(N=xx) | Placebo<br>(N=xx) |
|---|---|---|---|
| V 1916 | | | |
| Haemoglobin (unit) | | | |
| Baseline | n | XX | XX |
| | Mean | XX.X | XX.X |
| | SD | XX.XX | XX.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |
| Visit 3 (day 4) | n | XX | XX |
| Visit 5 (day 4) | Mean | XX.X | XX.X |
| | SD | XX.XX | XX.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |
| Change from Baseline to Visit 3 (day 4) | n | XX | XX |
| | Mean | XX.X | XX.X |
| | SD | XX.XX | XX.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |

**Footnote:** Baseline is the last recorded value for each parameter prior to treatment.

SOURCE: X:\Numerus\Studies\XXX\XXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Page X of Y

Programming notes: Repeat for the categories, parameters and relevant visits indicated in the SAP. Also include final assessment visit and change from baseline. Do not present day 1 on the baseline label.

Table 14.4.5.2
Shift Table of Laboratory Results from Baseline to Worst Post Baseline Result by Category and Treatment Group Safety Analysis Set

**Laboratory Category: Haematology** 

**Treatment: GBR 830** 

| Parameter | Worst Post- | Statistic | | | Baseline | | |
|---|---|---|---|---|---|---|---|
| | Baseline Result | | Abnormal, low | Normal | Abnormal, high | Missing | Total |
| Haemoglobin (unit) | | | | | | | |
| 2 ( ) | Abnormal, low | n/N* (%) | x/X(xxx) | x/X(xxx) | x/X (xxx) | x/X(xxx) | x/X(xxx) |
| | Normal | n/N* (%) | x/X (xxx) | x/X (xxx) | x/X (xxx) | x/X (xxx) | x/X (xxx) |
| | Abnormal, high | n/N* (%) | x/X (xxx) | x/X (xxx) | x/X (xxx) | x/X (xxx) | x/X (xxx) |
| | Missing | n/N* (%) | x/X (xxx) | x/X (xxx) | x/X (xxx) | x/X (xxx) | x/X (xxx) |
| | Total | n/N* (%) | x/X (xxx) | x/X (xxx) | x/X (xxx) | x/X (xxx) | x/X (xxx) |

**Footnote**: N\* is the number of subjects with the result at the Baseline visit. Percentages are based on N\* in each treatment group. Baseline is the last recorded value for each parameter prior to treatment. If a subject has both an 'abnormal, low' and an 'abnormal, high' worst post baseline result, both results will be included.

SOURCE: X:\Numerus\Studies\XXX\XXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Page X of Y

Programming notes: Repeat for the categories and parameters indicated in the SAP. If required add 'Abnormal, (low and high)' column and row to the output for all parameters.

Table 14.4.6.1 Change from Baseline in Vital Signs Results by Parameter and Visit Safety Analysis Set

| Parameter | Statistic | GBR 830 | Placebo |
|-----------------------------------------|-----------|---------|---------|
| Visit | | (N=xx) | (N=xx) |
| Systolic blood pressure (mmHg) | | | |
| Baseline | n | XX | XX |
| | Mean | XX.X | XX.X |
| | SD | XX.XX | XX.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |
| Visit 3 (day 4) | n | XX | xx |
| | Mean | XX.X | XX.X |
| | SD | XX.XX | XX.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |
| Change from Baseline to Visit 3 (day 4) | n | XX | XX |
| | Mean | XX.X | XX.X |
| | SD | XX.XX | XX.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |

**Footnote:** Baseline is the last recorded value for each parameter prior to treatment.

SOURCE: X:\Numerus\Studies\XXX\XXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Page X of Y

Programming note: repeat for appropriate visits and parameters- Diastolic blood pressure (mmHg), body temperature ( $^{\circ}$ C), pulse rate (bpm), weight (kg), bmi (kg/m²) Do not present day 1 on the baseline label.

Table 14.4.6.2
Shift Table of Vital Signs from Baseline to Worst Post Baseline Result by Treatment Group Safety Analysis Set

**Treatment: GBR 830** 

| Parameter Worst Post-<br>Visit baseline Result | | Statistic | | Baseline | | | |
|---|---|---|---|---|---|---|---|
| | | Normal | Abnormal<br>(NCS) | Abnormal (CS) | Missing | Total | |
| Systolic blood pressure (mmHg) | | | | | | | |
| (11111115) | Normal | n/N* (%) | x/X (xxx) | x/X (xxx) | x/X (xxx) | x/X (xxx) | x/X (xxx) |
| | Abnormal (NCS) | n/N* (%) | x/X (xxx) | x/X (xxx) | x/X (xxx) | x/X (xxx) | x/X (xxx) |
| | Abnormal (CS) | n/N* (%) | x/X (xxx) | x/X (xxx) | x/X (xxx) | x/X (xxx) | x/X (xxx) |
| | Missing | n/N* (%) | x/X (xxx) | x/X (xxx) | x/X (xxx) | x/X (xxx) | x/X (xxx) |
| | Total | n/N* (%) | x/X (xxx) | x/X(xxx) | x/X (xxx) | x/X (xxx) | x/X (xxx) |
| Diastolic blood pressure (mmHg) | | | | | | | |
| ( | Normal | n/N* (%) | x/X(xxx) | x/X(xxx) | x/X(xxx) | x/X(xxx) | x/X (xxx) |
| | Abnormal (NCS) | n/N* (%) | x/X (xxx) | x/X (xxx) | x/X (xxx) | x/X (xxx) | x/X (xxx) |
| | Abnormal (CS) | n/N* (%) | x/X (xxx) | x/X (xxx) | x/X (xxx) | x/X (xxx) | x/X (xxx) |
| | Missing | n/N* (%) | x/X (xxx) | x/X (xxx) | x/X (xxx) | x/X (xxx) | x/X (xxx) |
| | Total | n/N* (%) | x/X (xxx) | x/X (xxx) | x/X (xxx) | x/X (xxx) | x/X (xxx) |

**Footnote**: N\* is the number of subjects with the result at the Baseline visit. Percentages are based on N\* in each treatment group. NCS: Not Clinically Significant. CS: Clinically significant. Baseline is the last recorded value for each parameter prior to treatment.

SOURCE: X:\Numerus\Studies\XXX\XXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Page X of Y

Programming note: repeat for appropriate visits and parameters- Diastolic blood pressure (mmHg), body temperature (°C), pulse rate (bpm), weight (kg), BMI (kg/m²)

Table 14.4.7
Physical Examination Results
Safety Analysis Set

| Parameter<br>Visit | Statistic | GBR 830<br>(N=xx) | Placebo<br>(N=xx) | Overall (N=xx) |
|---|---|---|---|---|
| VISIT | | | | |
| Thorax/Lungs | | | | |
| Baseline | | | | |
| Done | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Not done | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Worst post-baseline | | | | |
| Not examined | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Normal | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Abnormal, not clinically significant | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Abnormal, clinically significant | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Etc. | . , | , , | . , | |

**Footnote**: Percentages are based on the total number of subjects in Safety Analysis Set in each treatment group. Baseline is the last recorded value for each parameter prior to treatment.

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Page X of Y

Repeat for Parameters: Cardiovascular system, Neurological examination, Other.

Table 14.4.8.1 Change from Baseline in Electrocardiogram Results by Parameter and Visit Safety Analysis Set

| Parameter<br>Visit | Statistic | GBR 830<br>(N=xx) | Placebo<br>(N=xx) |
|---|---|---|---|
| Heart rate (bpm) | | | |
| Baseline | n | XX | XX |
| | Mean | XX.X | XX.X |
| | SD | XX.XX | XX.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |
| Visit 3 (day 4) | n | XX | xx |
| | Mean | XX.X | XX.X |
| | SD | XX.XX | XX,XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |
| Change from Baseline to Visit 3 (day 4) | n | XX | XX |
| | Mean | XX.X | XX.X |
| | SD | XX.XX | XX.XX |
| | Median | XX.X | XX.X |
| | Min. | XX | XX |
| | Max. | XX | XX |

**Footnote**: Baseline is the last recorded value for each parameter prior to treatment.

SOURCE: X:\Numerus\Studies\XXX\XXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Page X of Y

#### Programming Notes:

1. Include all 12-lead ECG data listed in the protocol: PR interval (ms), RR interval (ms), QRS duration (ms), QT interval (ms), QTcF interval (ms), repeat for relevant visits.

Table 14.4.8.2 Overall Interpretations of Electrocardiogram by Visit Safety Analysis Set

| Visit<br>Categorization | Statistic | GBR 830<br>(N=xx) | Placebo<br>(N=xx) | Overall (N=xx) |
|---|---|---|---|---|
| Overall prolongation | | | | |
| QTc interval > 500ms at any visit | n (%) | x (xxx) | x (xxx) | x (xxx) |
| QTc interval > 60ms change at any post baseline visit | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Baseline | | | | |
| Normal | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Abnormal not clinically significant | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Abnormal and clinically significant | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Visit 3 (day 4) | | | | |
| Normal | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Abnormal not clinically significant | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Abnormal and clinically significant | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Visit 4 (day 8) | | | | |
| Normal | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Abnormal not clinically significant | n (%) | x (xxx) | x (xxx) | x (xxx) |
| Abnormal and clinically significant | n (%) | x (xxx) | x (xxx) | x (xxx) |
| etc. | | | | |

**Footnote**: Percentages are based on the total number of subjects in Safety Analysis Set in each treatment group. Baseline is the last recorded value for each parameter prior to treatment.

SOURCE: X:\Numerus\Studies\XXX\XXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Page X of Y

Programming notes: repeat for relevant planned visits.
Table 14.4.9
GBR830 Serum Concentration (ng/mL) Data by Dose Interval
Pharmacokinetic Analysis Set

#### LLOQ=xx.xx ng/mL

| Dose Interval<br>Time Point | n | Mean | SD | CV (%) | Median | Min | Max |
|---|---|---|---|---|---|---|---|
| Dose 1 | | | | | | | |
| pre dose (-0.25 hours) | XX | XX.X | XX.XX | XX.XX | XX.X | XX | XX |
| end of dose (1 hours) | XX | XX.X | XX.XX | XX.XX | XX.X | XX | XX |
| post dose (1.5 hours) | XX | XX.X | XX.XX | XX.XX | XX.X | XX | XX |
| Etc. | | | | | | | |

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

*Programming note: repeat for all time points and dose 2 – see SAP text for dose interval details.* 

Table 14.4.10
Pharmacokinetic Parameters of GBR830 by Dose Interval
Pharmacokinetic Analysis Set

| Dose<br>Interval | Statistic | AUC0-t<br>(μg.h/mL) | AUC0-tau<br>(μg.h/mL) | AUC0-∞<br>(μg.h/mL) | Cmax<br>(µg/mL) | Tmax (h) | λz (1/h) | t1/2 (h) | Vd (L) | CL (L/h) |
|---|---|---|---|---|---|---|---|---|---|---|
| Dose 1 | N | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| 20001 | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | CV (%) | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | Geometric Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Geometric CV<br>(%) | XX.XX | XX.XX | XX.XX | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX | xx.xx |

Footnote: AUC0- $\infty$ =area under the (serum) concentration-time curve to infinity; AUC0-t=area under the (serum) concentration-time curve to the last time point where quantifiable concentration is observed; AUC0-tau=area under the (serum) concentration-time curve to the last observed time point in the interval; CL=clearance; Cmax=maximum concentration; Tmax=Time of Cmax. t1/2=terminal half-life; Vd=volume of distribution.

SOURCE: X:\Numerus\Studies\XXX\XXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Page X of Y

Programming note: repeat for dose 2.

Glenmark Pharmaceutical SA Statistical Analysis Plan – Protocol GBR 830-201

6-Jul-17

# Figure 14.3.1.1 Box plot of biomarker CCL11/hARPby Planned Treatment Group Biological Activity Set

**Footnote:** Source table: 14.3.1.1

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Analysis Plan: 06Jul2017 Confidential Page X of Y

**Repeat for:** Figure 14.3.1.2 to 14.3.1.19 biomarkers as appropriate.

Figure 14.3.3.1 Line Plot of EASI 50 Responders over Time (days) by Planned Treatment Group Full Analysis Set



Footnote: Source table: 14.3.3.1.

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXX.sas
Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Figure 14.3.4.1

Line Plot of Mean ± SE Percentage Change in EASI Score over Time (days) by Planned Treatment Group

Full Analysis Set



**Footnote**: Source table: 14.3.4.1.

Figure 14.3.4.4
Line Plot of Mean ± SE Percentage Change in Pruritus NRS over Time (days) by Planned Treatment Group
Full Analysis Set

Footnote: Source table: 14.3.4.4.

Figure 14.3.6.1 Scatter Plot of Serum Concentration (μg/mL) over Anti Drug Antibody Status by Planned Treatment Group Pharmacokinetic Analysis Set



Figure 14.4.11.1 Mean Serum GBR830 Concentration Data (0 to 2016 hours) Overall Pharmacokinetic Analysis Set



Time since first dose initiation (h)

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

# Figure 14.4.11.2 Individual Subject Profiles of Serum GBR830 Concentration Data (0 to 2016 hours) Pharmacokinetic Analysis Set



SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Page X of Y

Time since first dose initiation (h)

### Listing 16.1.1 Subject Disposition Randomized Subjects

| Planned<br>Treatment | Subject ID | Date of First<br>Treatment | Date of Last<br>Treatment | Date of<br>Withdrawal from<br>Study | Study Day of<br>Withdrawal | Did Subject<br>Complete all<br>Scheduled<br>Visits? | Reason for Withdrawal |
|---|---|---|---|---|---|---|---|
| XXXXXXX | XX-XXXXXX | DDMMMYYYY | DDMMMYYYY | DDMMMYYYY | X | Yes | XXXXXXXXX |
| XXXXXXX | XX-XXXXXX | DDMMMYYYY | DDMMMYYYY | DDMMMYYYY | X | XXX | XXXXXXXXX |
| XXXXXXX | XX-XXXXXX | DDMMMYYYY | DDMMMYYYY | DDMMMYYYY | X | XXX | XXXXXXXXX |
| XXXXXXX | XX-XXXXXX | DDMMMYYYY | DDMMMYYYY | DDMMMYYYY | X | XXX | XXXXXXXXX |
| XXXXXXX | xx-xxxxxx | DDMMMYYYY | DDMMMYYYY | DDMMMYYYY | X | XXX | XXXXXXXXX |
| XXXXXXX | xx-xxxxxx | DDMMMYYYY | DDMMMYYYY | DDMMMYYYY | X | XXX | XXXXXXXXX |
| XXXXXXX | XX-XXXXXX | DDMMMYYYY | DDMMMYYYY | DDMMMYYYY | X | XXX | XXXXXXXXX |

Footnote: If status is 'Lost to Follow up' Reason for withdrawal will include the date of last contact with subject. If Subject status is 'Death', date of death will be included.

SOURCE: X:\Numerus\Studies\XXX\XXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Listing 16.1.2 Analysis Populations Screened Subjects

| Subject ID | Screened | Randomized | Full Analysis Set | Safety Analysis Set | Pharmacokinetic<br>Analysis Set | <b>Biological Activity Set</b> |
|---|---|---|---|---|---|---|
| xx-xxxxxx | Yes | Yes | Yes | Yes | Yes | Yes |
| XX-XXXXXX | XXX | XXX | XXX | XXX | XXX | XXX |
| XX-XXXXXX | XXX | XXX | XXX | XXX | XXX | XXX |

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Listing 16.1.3
Subject Inclusion/Exclusion Criteria
Screened Subjects

| Planned<br>Treatment | Subject ID | Visit | Inclusion<br>Criteria<br>met? | Reason Inclusion<br>Criteria not met | Exclusion criteria met? | Reason Exclusion criteria not met | Randomization status |
|---|---|---|---|---|---|---|---|
| | XX-XXXXXX | Screening | No | xxxxxxxxxxxxx | Yes | | Screen Failed |
| | xx-xxxxxx | Screening | Yes | | Yes | | |
| | | Baseline | Yes | | No | XXXXXXXXXXXXXXX | Screen Failed |
| | xx-xxxxxx | Screening | Yes | | Yes | | |
| XXX | xx-xxxxxx | Baseline | Yes | | Yes | | Randomized |

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

### Listing 16.1.4 Screen Failure Subjects Screened Subjects

| Subject ID | Reason for Screen Failure | Rescreened | Replaced | Previous Screening Number |
|---|---|---|---|---|
| XX-XXXXXX | Xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | Yes | No | XX-XXXXX |
| XX-XXXXXX | Xxxxxxxxxxxxxxxxxxxxxxx | Yes | No | XX-XXXXXX |
| XX-XXXXXX | Xxxxxxxxxxxxxxxxxxxxxxx | No | Yes | |

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Listing 16.1.5
Subject Randomization Information
Randomized Subjects

| Planned<br>Treatment | Subject ID | <b>Date of Consent</b> | Date of<br>Randomization | Randomization number | Blind<br>Broken? | Date Blind Broken | Reason for Blind<br>Broken |
|---|---|---|---|---|---|---|---|
| GBR 830 | xx-xxxxxx | DDMMMYYYY | DDMMMYYYY | XXXX | Yes | DDMMMYYYY | XXXXXXXXXXXXXX |
| Placebo | xx-xxxxxx | DDMMMYYYY | DDMMMYYYY | XXXX | No | | |
| xxxxxxx | xx-xxxxxx | DDMMMYYYY | DDMMMYYYY | XXXX | XXX | | |
| ΑΛΛΑΛΑ | AA AAAAAA | | | AAAA | AAA | | |

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Analysis Plan: 06Jul2017 Confidential Page X of Y

Listing 16.2.1.1.1
Subject Demographic and Baseline Characteristics – Part 1
Randomized Subjects

| Planned<br>Treatment | Subject ID | Date of Birth (Age) | Sex | Race | Weight<br>(kg) | Height (cm) | Body Mass<br>Index (kg/m²) | Body Surface<br>Area (m²) |
|---|---|---|---|---|---|---|---|---|
| xxxxxxx | xx-xxxxx | DDMMMYYYY<br>(xx) | Male | Asian | XX.X | XX.X | xxx | Xxx |
| xxxxxxx | xx-xxxxxx | DDMMMYYYY<br>(xx) | Female | xxxxxxx | XX.X | XX.X | XXX | Xxx |
| xxxxxxx | xx-xxxxxx | DDMMMYYYY<br>(xx) | xxxx | xxxxxxx | XX.X | XX.X | XXX | Xxx |
| xxxxxxx | xx-xxxxxx | DDMMMYYYY<br>(xx) | xxxx | xxxxxxx | XX.X | XX.X | XXX | Xxx |
| xxxxxxx | xx-xxxxxx | DDMMMYYYY<br>(xx) | xxxx | xxxxxxx | XX.X | XX.X | XXX | Xxx |
| XXXXXXX | xx-xxxxxx | DDMMMYYYY<br>(xx) | XXXX | xxxxxxx | XX.X | XX.X | xxx | Xxx |

SOURCE: X:\Numerus\Studies\XXX\XXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Page X of Y

Repeat for:

Listing 16.2.1.1.2
Subject Demographic and Baseline Characteristics – Part 1
Screen Failure Subjects

# Listing 16.2.1.2.1 Subject Demographic and Baseline Characteristics – Part 2 Randomized Subjects

| Planned<br>Treatment | Subject ID | Age at AD diagnosis | Ethnicity | Country | Child Bearing Potential, Specify | Duration of Non Child<br>Bearing Potential |
|---|---|---|---|---|---|---|
| xxxxxxx | xx-xxxxxx | xx | Hispanic or Latino | Canada | N/A | |
| XXXXXXX | XX-XXXXXX | XX | Not Hispanic or Latino | XXXXXXX | No, Post menopausal | > 1 year |
| XXXXXXX | XX-XXXXXX | XX | XXXX | XXXXXXX | | |
| XXXXXXXX | XX-XXXXXX | XX | XXXX | XXXXXXXX | | |
| XXXXXXXX | XX-XXXXXX | XX | XXXX | XXXXXXX | | |
| XXXXXXXX | XX-XXXXXX | XX | XXXX | XXXXXXX | | |

Page X of Y

Repeat for:

Listing 16.2.1.2.2
Subject Demographic and Baseline Characteristics – Part 2
Screen Failure Subjects

### Listing 16.2.2 Atopic Dermatitis History Randomized Subjects

| Planned<br>Treatment | Subject<br>ID | Years<br>since AD<br>diagnosis | Type of AD | Any<br>History of<br>Allergy? | Was Patch<br>Test<br>Performed? | Any<br>Known<br>Allergen<br>identified? | Concomitant<br>Atopic Illness | Remarks | Result of Skin<br>Biopsy<br>performed in<br>Past? | Any treatment administered for AD or associated conditions? |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxxx | XXX-<br>XXXXX | XX | Intrinsic | Yes | Yes | XXXXXXXXXX<br>XX | Asthma | | Eosinophilic | Yes |
| xxxxxxx | xxx-<br>xxxxx | XX | Extrinsic | No | No | | Asthma, Skin<br>Conditions | | Non-eosinophilic | No |
| xxxxxxx | xxx-<br>xxxxx | XX | Intrinsic | No | No | | Asthma, Other , xxxxxx | xxxxxxxx | Other, xxxxxx | |
| | | | | | | | None | | Not done | |

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Listing 16.2.3 Medical/Surgical History Randomized Subjects

| Planned<br>Treatment | Subject ID | Start Date | End date | Ongoing? | Body System | Condition/Procedure | Severity grade |
|---|---|---|---|---|---|---|---|
| xxxxxxx | xx-xxxxxx | DDMMMYYYY | | Yes | HEENT | xxxxxxxxxxx | Mild |
| xxxxxxx | xx-xxxxxx | DDMMMYYYY | DDMMMYYYY | No | XXXXXXX | XXXXXXXXXXX | Moderate |
| XXXXXXX | XX-XXXXXX | <b>DDMMMYYYY</b> | DDMMMYYYY | XXX | XXXXXXXX | xxxxxxxxxxx | Severe |
| XXXXXXX | XX-XXXXXX | DDMMMYYYY | DDMMMYYYY | XXX | XXXXXXXX | xxxxxxxxxxx | Not Known |

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMYYYY HH:MM; Date of data extraction: DDMMYYYY

### Listing 16.2.4.1 Smoking, Alcohol and Drug Abuse History – Part 1 Randomized Subjects

| Planned<br>Treatment | Subject ID | Alcohol<br>User? | Alcohol Stop<br>Date | Alcohol<br>Consumption<br>(ml/Week) | Is There<br>History of<br>Alcohol<br>Abuse? | Drug<br>Abuse? | Drug Abuse Stop<br>Date | Form of<br>Drug | Clinically<br>Significant? |
|---|---|---|---|---|---|---|---|---|---|
| xxxxxxx<br>xxxxxxx<br>xxxxxxx | xxx-xxxx<br>xxx-xxxx<br>xxx-xxxx | Former<br>Current<br>N/A | DDMMMYYYY | xxxx.xx<br>xxxx.xx<br>N/A | Yes<br>No<br>No | Former<br>Current<br>N/A | DDMMMYYYY | xxxxxxx | Yes<br>No |

Footnote: Clinical significance of drug use is determined by the opinion of the investigator or if the subject meets the DSM-V criteria for abuse.

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas Date/time of run: DDMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Analysis Plan: 06Jul2017 Confidential Page X of Y

Listing 16.2.4.2 Smoking, Alcohol and Drug Abuse History – Part 2 Randomized Subjects

| Planned<br>Treatment | Subject ID | Smoker? | Smoking Stop<br>Date | Number of<br>Cigarettes<br>per day | Smokeless<br>Tobacco User? | Tobacco<br>Consumption<br>Stop Date | Form of Tobacco |
|---|---|---|---|---|---|---|---|
| xxxxxxx | XXX-XXXXX | Former | DDMMMYYYY | XXX | Former | DDMMMYYYY | xxxxxxxxxx |
| XXXXXXX | XXX-XXXXX | Current | | XXX | Current | | |
| | XXX-XXXXX | N/A | | N/A | N/A | | |

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Listing 16.2.5.1
Atopic Dermatitis and Related Conditions Baseline Prior Medications
Randomized Subjects

| Planned<br>Treatment | Subject ID | ATC Level/<br>Preferred Term/<br>Verbatim Term | Start Date | Stop Date | Ongoing<br>at<br>Baseline | Dose (Unit) | Route/Frequency | Indication |
|---|---|---|---|---|---|---|---|---|
| xxxxxxx | xxx-xxxxx | Xxxxxxxxxxxxxx/<br>Xxxxxxxxxxxxxx/<br>xxxxxxxx | DDMMMYYYY | | Yes | xxx (xxx) | PO/OD | xxxxxxx |
| | | Xxxxxxxxxxxxxx/<br>Xxxxxxxxxxxxxx/<br>xxxxxxxx | DDMMMYYYY | DDMMMYYYY | xxx | xxx (xxx) | XXX | xxxxxxx |
| | | Xxxxxxxxxxxxxx/<br>Xxxxxxxxxxxxxx/<br>xxxxxxxx | DDMMMYYYY | DDMMMYYYY | xxx | xxx (xxx) | XXX | xxxxxxx |
| | | Xxxxxxxxxxxxx/<br>Xxxxxxxxxxxxxx/<br>xxxxxxxxx | DDMMMYYYY | DDMMMYYYY | XXX | xxx (xxx) | XXX | xxxxxx |
| xxxxx | XXX-XXXXXX | Xxxxxxxxxxxxx/<br>Xxxxxxxxxxxxxx/<br>xxxxxxxxx | | | | | | |

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Page X of Y

Repeat for:

Listing 16.2.5.2
Other Baseline Prior Medications
Randomized Subjects

# Listing 16.2.6 Baseline Physical Examination Randomized Subjects

| Planned<br>Treatment | Subject ID | Physical<br>Examination<br>Performed? | Body System | Results | Comments |
|---|---|---|---|---|---|
| xxxxx | xxx-xxxxxx | Done | Neck<br>HEENT<br>Skin | Normal<br>Abnormal CS<br>Not Examined | XXXX<br>XXXX |
| xxxxx | xxx-xxxxxx | Not Done | | | |

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Listing 16.3.1
Active AD mRNA Expression Signature and Pathologic Epidermal Phenotype Measures
Full Analysis Set

| Planned<br>Treatment | Subject ID | Parameter | Visit (Study Day)* | Visit Date | Measurement | Measurement Change<br>From Baseline |
|---|---|---|---|---|---|---|
| xxxxxxx | xx-xxxxxx | hARP | 2 ( 1)* | DDMMMYYYY | XXX.XX | N/A |
| | | | 7 (29) | DDMMMYYYY | XXX.XX | XXX.XX |
| | | | Unscheduled (31) | DDMMMYYYY | XXX.XX | XXX.XX |
| | | | 13 (71) | DDMMMYYYY | XXX.XX | XXX.XX |
| | | K16 | 2(1)* | DDMMMYYYY | XXX.XX | N/A |
| | | | 7 (29) | DDMMMYYYY | XXX.XX | xxx.xx |
| | | | 13 (71) | DDMMMYYYY | XXX.XX | xxx.xx |
| | etc. | | | | | |
| XXXXXXX | XX-XXXXXX | hARP | 2(1)* | DDMMMYYYY | XXX.XX | N/A |
| | | | 7 (29) | DDMMMYYYY | XXX.XX | XXX.XX |
| | | | 13 (71) | DDMMMYYYY | XXX.XX | XXX.XX |
| | | K16 | 2(1)* | DDMMMYYYY | XXX.XX | N/A |
| | | | 7 (29) | DDMMMYYYY | XXX.XX | XXX.XX |
| | | | 13 (71) | DDMMMYYYY | XXX.XX | xxx.xx |

**Footnote:** \* indicates the baseline record.

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Page X of Y

Programming notes: 1) Repeat for parameters mRNA in primary analysis table

Listing 16.3.2 IGA Scores Full Analysis Set

| Planned<br>Treatment | Subject ID | Visit (Study Day)* | Visit Date | IGA Score# | Score Category |
|---|---|---|---|---|---|
| XXXXXXX | xx-xxxxxx | 2 (1)* | DDMMMYYYY | 0 | 0 or 1 |
| | | 3 (4) | DDMMMYYYY | 3 | 2 + |
| | | 4(8) | <b>DDMMMYYYY</b> | 3 | 2 + |
| | | 5 (15) | <b>DDMMMYYYY</b> | 3 | 2 + |
| | | 6 (22) | <b>DDMMMYYYY</b> | | 2 + |
| | | 7 (29) | <b>DDMMMYYYY</b> | 4 | 2 + |
| | | 8 (32) | <b>DDMMMYYYY</b> | XX | XX |
| | | 9 (36) | DDMMMYYYY | XX | XX |
| | | 10 (43) | <b>DDMMMYYYY</b> | XX | XX |
| | | 11 (50) | DDMMMYYYY | XX | XX |
| | | 12 (57) | DDMMMYYYY | XX | XX |
| | | 13 (71) | DDMMMYYYY | xx# | XX |
| | | 14 (85) | DDMMMYYYY | xx# | XX |

**Footnote:** \* indicates the baseline record. # indicates measures that were excluded following a prohibited medication.

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Listing 16.3.3 EASI Scores Randomized Subjects

| Planned<br>Treatment | Subject ID | Visit (Study Day)* | Visit Date | EASI score # | EASI 50 responder? | EASI 75 responder? | Percent change from Baseline |
|---|---|---|---|---|---|---|---|
| xxxxxxx | xx-xxxxxx | 2 (1)* | DDMMMYYYY | 60 | N/A | N/A | N/A |
| | | 3 (4) | DDMMMYYYY | 15 | Yes | Yes | XX |
| | | 4 (8) | DDMMMYYYY | | No | No | XX |
| | | 5 (15) | DDMMMYYYY | XXX | XXX | Xxx | XX |
| | | 6 (22) | DDMMMYYYY | XXX | XXX | Xxx | XX |
| | | 7 (29) | DDMMMYYYY | XXX | XXX | Xxx | XX |
| | | 8 (32) | DDMMMYYYY | XXX | XXX | Xxx | XX |
| | | 9 (36) | DDMMMYYYY | XXX | XXX | Xxx | XX |
| | | 10 (43) | DDMMMYYYY | XXX | XXX | Xxx | XX |
| | | 11 (50) | DDMMMYYYY | XXX | XXX | Xxx | XX |
| | | 12 (57) | DDMMMYYYY | XXX | XXX | Xxx | XX |
| | | 13 (71) | DDMMMYYYY | XXX | XXX | Xxx | XX |
| | | 14 (85) | DDMMMYYYY | XXX | XXX | Xxx | XX |

**Footnote:** \* indicates the baseline record. # indicates measures that were excluded following a prohibited medication.

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

### Listing 16.3.4.1 SCORAD Clinical Scores Full Analysis Set

| Planned<br>Treatment | Subject ID | Visit (Study Day)* | Visit Date | Measurement# | Measurement Change from Baseline | Percent change fron<br>Baseline |
|---|---|---|---|---|---|---|
| xxxxxxx | xx-xxxxxx | 2 (1)* | DDMMMYYYY | XX | N/A | N/A |
| | | 3 (4) | DDMMMYYYY | XX | XX | XX |
| | | 4(8) | DDMMMYYYY | XX | XX | XX |
| | | 5 (15) | DDMMMYYYY | XX | XX | XX |
| | | 6 (22) | DDMMMYYYY | XX | XX | XX |
| | | 7 (29) | <b>DDMMMYYYY</b> | XX | XX | XX |
| | | 8 (32) | <b>DDMMMYYYY</b> | XX | XX | XX |
| | | 9 (36) | DDMMMYYYY | XX | XX | XX |
| | | 10 (43) | <b>DDMMMYYYY</b> | XX | XX | XX |
| | | 11 (50) | DDMMMYYYY | XX | XX | XX |
| | | 12 (57) | DDMMMYYYY | XX | XX | XX |
| | | 13 (71) | DDMMMYYYY | XX | XX | XX |
| | | 14 (85) | DDMMMYYYY | XX | XX | XX |

**Footnote:** \* indicates the baseline record. # indicates measures that were excluded following a prohibited medication.

SOURCE: X:\Numerus\Studies\XXX\XXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Page X of Y

Repeat for:

Listing 16.3.4.4
Pruritus NRS Clinical Scores
Full Analysis Set

Listing 16.3.4.5 DLQI Clinical Scores Full Analysis Set

Listing 16.3.5
Transepidermal Water Loss Readings
Full Analysis Set

| Planned<br>Treatment | Subject ID | Area | Visit (Study Day)* | Visit Date | Measurement# | Measurement change<br>from baseline |
|---|---|---|---|---|---|---|
| xxxxxxx | xx-xxxxxx | Lesion | 2 (1)* | DDMMMYYYY | xxx.xx | N/A |
| | | | 3 (4) | DDMMMYYYY | XXX.XX | XXX.XX |
| | | | 4 (8) | DDMMMYYYY | XXX.XX | XXX.XX |
| | | | 5 (15) | DDMMMYYYY | XXX.XX | XXX.XX |
| | | | 6 (22) | DDMMMYYYY | XXX.XX | XXX.XX |
| | | | 7 (29) | DDMMMYYYY | XXX.XX | XXX.XX |
| | | | 8 (32) | DDMMMYYYY | XXX.XX | XXX.XX |
| | | | 9 (36) | DDMMMYYYY | XXX.XX | XXX.XX |
| | | | 10 (43) | DDMMMYYYY | XXX.XX | XXX.XX |
| | | | 11 (50) | DDMMMYYYY | XXX.XX | XXX.XX |
| | | | 12 (57) | DDMMMYYYY | XXX.XX | XXX.XX |
| | | | 13 (71) | DDMMMYYYY | XXX.XX | XXX.XX |
| | | | 14 (85) | DDMMMYYYY | XXX,XX | XXX.XX |
| | | Non-Lesion | 2(1)* | DDMMMYYYY | XXX.XX | N/A |
| | etc. | | . , | | | |

**Footnote:** \* indicates the baseline record. # indicates measures that were excluded following a prohibited medication.

SOURCE: X:\Numerus\Studies\XXX\XXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMYYYY HH:MM; Date of data extraction: DDMMYYYY

### Listing 16.3.6 Anti-Drug Antibodies (ADA) Safety Analysis Set

| Actual<br>Treatment | Subject ID | Visit (Study Day)* | Visit Date | Titration# | Antibody | Neutralizing<br>Antibody |
|---|---|---|---|---|---|---|
| xxxxxxx | XX-XXXXXX | 2 (1)* | DDMMMYYYY | XXX | Negative | |
| | | 5 (15) | DDMMMYYYY | XXX | Negative | |
| | | 7 (29) | DDMMMYYYY | XXX | Positive | |
| | | 12 (57) | DDMMMYYYY | | Negative | |
| | | 14 (85) | DDMMMYYYY | XXX | Negative | |

Footnote: \* indicates the baseline record. # indicates measures that were excluded following a prohibited medication.

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

### Listing 16.3.8 Leukocytes Sub-Population Cell Counts Full Analysis Set

| Planned<br>Treatment | Subject ID | Parameter | Visit (Study Day)* | Visit Date | Measurement# | Measurement Change from Baseline | Percent change from<br>Baseline |
|---|---|---|---|---|---|---|---|
| xxxxxxx | xx-xxxxxx | XXX | 2 (1)* | DDMMMYYYY | XX | N/A | N/A |
| | | | 7 (29)<br>13 (71) | DDMMMYYYY<br>DDMMMYYYY | XX<br>XX# | XX<br>XX | XX<br>XX |

Footnote: \* indicates the baseline record. # indicates measures that were excluded following a prohibited medication.

Date/time of run: DDMMMYYYY HH:MM

Analysis Plan: 06Jul2017 Confidential Page X of Y

Repeat for:

Listing 16.3.9 Cellular Infiltrates Full Analysis Set

Listing 16.3.10 Serum Total Immunoglobulin E, Serum Soluble OX40, Serum Soluble OX40 and Circulating Eosinophil Counts Full Analysis Set

### Listing 16.3.12 Prohibited Medications Full Analysis Set

| Actual<br>Treatment | Subject ID | Prohibited Medication | Date of Prohibited<br>Medication | Study Day |
|---|---|---|---|---|
| VVVVVV | VV VVVVVV | VVVVVVVV | DDMMMYYYY | VV |
| XXXXXXX | XX-XXXXXX | XXXXXXXX | | XX |
| | | XXXXXXXX | DDMMMYYYY | XX |
| | | XXXXXXXX | DDMMMYYYY | XX |

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Listing 16.4.1.1.1 Adverse Events – Part 1 Safety Analysis Set

| Actual<br>Treatment | Subject<br>ID | AE<br>No. | Age | Sex | System Organ Class<br>(Preferred Term)<br>[Verbatim Term] | Start Date/Time<br>(Study Day) | Stop Date/Time<br>(Study Day) | Time on<br>Treatment<br>at Onset of<br>Event<br>(Days) | Duration<br>of AE<br>(days) | SAE |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxxx | xx-<br>xxxxxx | 1 | xx | XX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/<br>HH:MM (xxx) | DDMMMYYYY/<br>HH:MM (xxx) | xx | xx | Y |
| | | 2 | XX | XX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/<br>HH:MM (xxx) | DDMMMYYYY/<br>HH:MM (xxx) | XX | xx | |
| | | 3 | xxxx | XXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/<br>HH:MM (xxx) | DDMMMYYYY/<br>HH:MM (xxx) | XX | XX | |

Footnote: SAE: Serious Adverse Event.

SOURCE: X:\Numerus\Studies\XXX\XXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Page X of Y

Repeat for:

Listing 16.4.1.2.1 Serious Adverse Events – Part 1 Safety Analysis Set

### Glenmark Pharmaceutical SA Statistical Analysis Plan – Protocol GBR 830-201

6-Jul-17

Listing 16.4.1.5.1

Adverse Events Leading to Discontinuation of Study – Part 1

Safety Analysis Set

Listing 16.4.1.7.1

Adverse Events Leading to Death – Part 1

Safety Analysis Set

### Listing 16.4.1.1.2 Adverse Events – Part 2 Safety Analysis Set

| Actual<br>Treatment | Subject ID | AE No. | Severity | Relationship<br>to Study<br>Treatment | Action Taken with<br>Study Treatment | Other Action<br>Taken | Outcome | Treatment<br>Emergent<br>Flag |
|---|---|---|---|---|---|---|---|---|
| xxxxxxx | xx-xxxxxx | 1 | Mild | Related | Permanently withdrawn | Concomitant Medication given | Improved | Y |
| | | 2 3 | Moderate<br>Xxxx | Not Related xxxx | XX<br>XX | xx<br>xx | XX<br>XX | N |

SOURCE: X:\Numerus\Studies\XXX\XXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Page X of Y

Repeat for:

Listing 16.4.1.2.2 Serious Adverse Events – Part 2 Safety Analysis Set Include SAE criteria detail

Listing 16.4.1.5.2

Adverse Events Leading to Discontinuation of Study – Part 2

Safety Analysis Set

Listing 16.4.1.7.2

Adverse Events Leading to Death – Part 2

Safety Analysis Set

Listing 16.4.2 Study Drug Administration Safety Analysis Set

| Actual<br>Treatment | Subject ID | Visit (Study<br>Day) | Dosing Date | Start time | End time | Total<br>Volume<br>Prepared<br>(mL) | Planned<br>Volume to be<br>Administered<br>(mL) | Actual<br>Volume<br>Administered<br>(mL) | Compliance (%) |
|---|---|---|---|---|---|---|---|---|---|
| | | 2 (1) | | 1111.343.4 | IIII.MM | | | | |
| XXXXXXX | XX-XXXXXX | 2 (1) | DDMMMYYYY | HH:MM | HH:MM | XX.XX | XX.XX | XX.XX | XX.XX |
| | | 7 (29) | DDMMMYYYY | HH:MM | HH:MM | XX.XX | XX.XX | XX.XX | XX.XX |
| | | Overall | | | | XX.XX | XX.XX | XX.XX | XX.XX |
| xxxxxxx | xx-xxxxxx | 2 (1) | DDMMMYYYY | НН:ММ | НН:ММ | XX.XX | XX.XX | XX.XX | xx.xx |
| | | 7 (29) | DDMMMYYYY | HH:MM | НН:ММ | XX.XX | XX.XX | xx.xx | XX.XX |
| | | Overall | | | | XX.XX | XX.XX | XX.XX | xx.xx |

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

### Listing 16.4.3.1 Concomitant Medications Safety Analysis Set

| Actual<br>Treatment | Subject ID | ATC Level/<br>Preferred Term/<br>Verbatim Term | Start Date (Study<br>Day)[1] | Stop Date | Ongoing? | Dose (Unit) | Route/Frequency | Indication |
|---|---|---|---|---|---|---|---|---|
| xxxxxxx | xxx-xxxxx | Xxxxxxxxxxxxx/<br>Xxxxxxxxxxxxx/<br>xxxxxxxxxx | DDMMMYYYY<br>(xx) | | Yes | xxx (xxx) | PO/OD | xxxxxx |
| | | Xxxxxxxxxxxxxx/<br>Xxxxxxxxxxxxxx/<br>xxxxxxxx | DDMMMYYYY<br>(xx) | DDMMMYYYY | xxx | xxx (xxx) | XXX | XXXXXXX |
| | | Xxxxxxxxxxxxxx/<br>Xxxxxxxxxxxxxx/<br>xxxxxxxx | DDMMMYYYY<br>(xx) | DDMMMYYYY | XXX | xxx (xxx) | xxx | XXXXXX |
| | | Xxxxxxxxxxxx/<br>Xxxxxxxxxxxxxx/<br>xxxxxxxxxx | DDMMMYYYY<br>(xx) | DDMMMYYYY | XXX | xxx (xxx) | XXX | XXXXXX |
| xxxxx | XXX-XXXXXX | Xxxxxxxxxxxxx/<br>Xxxxxxxxxxxxx/<br>xxxxxxxxxx | | | | | | |

<sup>1.</sup> Footnote: [1] medications that started prior to Baseline will have 'NA' as the study day. Medications have been coded using WHO DDE (Sep 2015).

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Page X of Y

Repeat for:

Listing 16.4.3.3 Rescue Medications Safety Analysis Set
### Listing 16.4.3.2 Concomitant Non-Drug Therapies Safety Analysis Set

| Actual<br>Treatment | Subject ID | Non-Drug Treatment | Start Date (Study<br>Day) | Stop Date | Ongoing? | Reason |
|---|---|---|---|---|---|---|
| xxxxxxx | xxx-xxxxx | xxxxxxxx | DDMMMYYYY<br>(xx) | | Yes | xxxxxxxxxxx |
| | | xxxxxxxxx | DDMMMYYYY<br>(xx) | DDMMMYYYY | XXX | xxxxxxxxxxx |
| | | xxxxxxxxxx | DDMMMYYYY<br>(xx) | DDMMMYYYY | xxx | xxxxxxxxxx |
| | | xxxxxxxxxxx | DDMMMYYYYY<br>(xx) | DDMMMYYYY | XXX | xxxxxxxxxxx |
| xxxxx | xxx-xxxxxx | xxxxxxxxx | | | | |

<sup>1.</sup> Footnote: Medications that started prior to Baseline will have 'NA' as the study day. Medications have been coded using WHO DDE (Sep 2015).

SOURCE: X:\Numerus\Studies\XXX\XXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

### Listing 16.4.4.1.1 Heamatology Results Safety Analysis Set

| Actual<br>Treatment | Subject ID | Age/Sex | Laboratory<br>Parameter (unit) | Visit<br>(Study<br>Day) | Date/Time of collection | Result | Normal Range | Comment |
|---|---|---|---|---|---|---|---|---|
| xxxxxxx | xxx-xxxxx | xx/Male | xxxxxxxxx (xx) | 2 (1) | DDMMMYYYY/<br>MM:HH | xxx (H) | xx - xx | xxxxxxxx |
| | | | | 3 (4) | DDMMMYYYY/<br>MM:HH | xxx (L) | xx - xx | XXXXXXXX |
| | | | | 4 (8) | DDMMMYYYY/<br>MM:HH | XXX | xx - xx | XXXXXXXX |
| | | | | U (26) | | | | |
| | etc. | | | | | | | |

Footnote: H = result above normal range; L = result below normal range; U = unscheduled visit.

SOURCE: X:\Numerus\Studies\XXX\XXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Repeat for:

Page X of Y

### Listing 16.4.4.1.2 Subjects with Abnormal Hematology Results Safety Analysis Set

Listing 16.4.4.2.1 Serum Biochemistry Results Safety Analysis Set

Listing 16.4.4.2.2
Subjects with Abnormal Serum Biochemistry Results
Safety Analysis Set

6-Jul-17

Listing 16.4.4.3 Urinalysis Results Safety Analysis Set

Listing 16.4.4.4 Serology Results Safety Analysis Set

Listing 16.4.4.5 Other Laboratory Test Results Safety Analysis Set

Listing 16.4.5 Vital Signs Results Safety Analysis Set

| Actual<br>Treatment | Subject ID | Visit<br>(Study<br>Day) | Date | Scheduled<br>Time | Weight<br>(kg) | Systolic<br>Blood<br>Pressure<br>(mmHg) | Diastolic<br>Blood<br>Pressure<br>(mmHg) | Pulse<br>(beats/min) | Body<br>Temperature<br>(°C) | BMI (kg/m²) |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxxx | xxx-xxxxx | 2(1) | DDMMMYYYY | Pre-dose | XX.X | Xxx | XX | XX | XX.X | XX |
| | | . , | | X | XX.X | Xxx | XX | xx* | XX.X | XX |
| | | | | XX | XX.X | Xxx | XX | XX | XX.X | XX |
| | | | | XX | XX.X | Xxx | XX | XX | XX.X | XX |
| | | | | XX | XX.X | Xxx | XX | XX | XX.X | XX |
| | | 3 (4)<br>U (25) | DDMMMYYYY | | | | | | | |

**Footnote**: Clinically significant findings are signified by a \*. U = unscheduled visit.

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

# Listing 16.4.6 Brief Physical Examination Safety Analysis Set

| Actual<br>Treatment | Subject ID | Physical<br>Examination<br>Performed? | Body System | Results | Comments |
|---|---|---|---|---|---|
| xxxxx | xxx-xxxxxx | Done | Thorax/Lungs<br>Cardiovascular System<br>Neurological Examination | Normal<br>Abnormal CS<br>Not Examined | XXXX<br>XXXX |
| xxxxx | xxx-xxxxxx | Not Done | | | |

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Listing 16.4.7 Electrocardiogram (ECG) Results Safety Analysis Set

| Actual<br>Treatment | Subject ID | Visit<br>(Study<br>Day) | Date/Time of<br>Assessment | Heart<br>Rate<br>(Bpm) | PR Interval<br>(ms) | RR<br>Interval<br>(ms) | QRS<br>Interval<br>(ms) | QT Interval<br>(ms) | QTcF<br>Interval<br>(ms) | Finding |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxxx | xxx-xxxxx | 2(1) | DDMMYYYY/<br>HH:MM | xxx | XXX | xxx | xxx | XXX | xxx | Normal |
| | | XXX | | XXX | XXX | XXX | XXX | XXX | XXX | Abnormal, NCS |
| | | XXX | | XXX | XXX | XXX | XXX | XXX | XXX | |
| | | XXX | | XXX | XXX | XXX | XXX | XXX | XXX | |
| | | U (25) | | XXX | XXX | XXX | XXX | XXX | XXX | |

Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Analysis Plan: 06Jul2017 Confidential Page X of Y

Programming notes: Triplicate measures will be recorded in the visit description. I.e. 2 (1) – triplicate 1, 2 (1) – triplicate 2 etc.

# Listing 16.4.8 Individual GBR830 Serum Concentration (ng/mL) Data Pharmacokinetic Analysis Set

LLOQ=xx.xx ng/mL

| Subject ID | Study Day | | | Time Deviation | Reported | Comment |
|---|---|---|---|---|---|---|
| | | Scheduled | Actual | | (mins) | Concentration (ng/mL) |
| xxx-xxxxxx | | | | | | XXX.X |
| | | | | | | XXX.X |
| | | | | | | XXX.X |
| | | | | | | XXX.X |
| | | | | | | XXX.X |
| | | | | | | XXX.X |
| | | | | | | XXX.X |
| xxx-xxxxxx | | | | | | |
| | | | | Etc. | | |

SOURCE: X:\Numerus\Studies\XXX\XXXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Page X of Y

*Programming note: repeat for all time points and dose 2 – see SAP text for dose interval details.* 

6-Jul-17

Listing 14.4.9

#### Individual Pharmacokinetic Parameters of GBR830 Pharmacokinetic Analysis Set

| Subject ID | Dose<br>Interval | AUC0-t<br>(μg.h/mL) | AUC0-tau<br>(μg.h/mL) | AUC∞<br>(μg.h/mL) | Cmax<br>(μg/mL) | Tmax (h) | λz (1/h) | t1/2 (h) | Vd (L) | CL (L/h) |
|---|---|---|---|---|---|---|---|---|---|---|
| XX-XXXXXX | Dose 1 | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | NA | NA | XXX.X | XXX.X |
| | Dose 2 | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| xx-xxxxxx | Dose 1 | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | NA | NA | XXX.X | XXX.X |
| | Dose 2 | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| xx-xxxxxx<br>Etc. | Dose 1 | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | NA | NA | XXX.X | XXX.X |

**Footnote**: AUC0-∞=area under the (serum) concentration-time curve to infinity; AUC0-t=area under the (serum) concentration-time curve to the last time point where quantifiable concentration is observed; AUC0-tau=area under the (serum) concentration-time curve to the last observed time point in the interval; CL=clearance; Cmax=maximum concentration; Tmax=Time of Cmax. t1/2=terminal half-life; Vd=volume of distribution.

Listing~16.4.10 Time Points used to Calculate the GBR830 Elimination Rate Constant (\$\lambda z\$) Pharmacokinetic Analysis Set

| Subject ID | Lower Time (h) | Upper Time (h) | Number of Points | Adjusted R-Square | λz (1/h) | t½ (h) |
|---|---|---|---|---|---|---|
| XX-XXXXXX | XXX | XXX | XX | X.XXXX | XX.XXXX | XXX |

SOURCE: X:\Numerus\Studies\XXX\XXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMYYYY HH:MM; Date of data extraction: DDMMYYYY

Listing 16.4.11
Reasons Pharmacokinetic Parameters Could Not be Determined
Pharmacokinetic Analysis Set

| Subject ID | Pharmacokinetic<br>Parameter (Unit) | Original Value | Comment |
|---|---|---|---|
| xx-xxxxxx | xxxxxxx (xx) | XXX.X | xxxxxxxxxxxxxxxxxxxxxx |
| | xxxxxxx (xx) | XXX.X | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | xxxxxxx (xx) | XXX.X | xxxxxxxxxxxx |
| xx-xxxxxx | xxxxxxx (xx) | XXX.X | xxxxxxxxxxxxxxxxxxxxxx |

# Listing 16.5.2 Protocol Deviations Randomized Subjects

| Planned<br>Treatment | Subject | Protocol<br>Deviation<br>Number | Date reported<br>(Visit) | Deviation coding | Deviation Description, verbatim | Description of the actions taken | Reported to Ethics? |
|---|---|---|---|---|---|---|---|
| xxxxxxxxx | xx-xxxxxx | XX | DDMMMYYYY<br>(x) | Subject non-compliance with study procedures | XXX | List the description of the actions taken | Yes |
| | | XX | DDMMMYYYY<br>(x) | Randomization error | XXX | List the description of the actions taken | No |

SOURCE: X:\Numerus\Studies\XXX\XXYYY\Analysis\Prod\Progs\XXXXX.sas
Date/time of run: DDMMMYYYY HH:MM; Date of data extraction: DDMMYYYY

# 12. REFERENCES

- 1. Du Bois D, Du Bois EF. A formula to estimate the approximate surface area if height and weight be known. Archives of Internal Medicine. 17 (6): 863–71.Basra et al. The Dermatology Life Quality Index 1994–2007: a comprehensive review of validation data and clinical results. Br J Dermatol. 2008; 159: 997-1035.
- 2. Finlay et al. A simple practical measure for routine clinical use. Clin Exp Dermatol.1994;19:210-16
- 3. Hanifin et al. Diagnostic features of atopic dermatitis. Acta Derm Venereol Suppl (Stockh). 1980;92:44-7.
- 4. Hanifin et al. The eczema area and severity index (EASI): assessment of reliability in atopic dermatitis. Exp Dermatol, 2001, 10: 11-18.
- 5. Kunz B et al. Clinical validation and guidelines for the SCORAD index: consensus report of the European task for on atopic dermatitis. Dermatology. 1997:195:10-19.
- 6. No authors listed. (1993). Severity scoring of atopic dermatitis: the SCORAD index. Dermatology, 1993, 186: 23-31.